Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM) – Dihydropyridine CCBs vs Hydrochlorothiazide

NCT05125224

November 23, 2021

# 1. Comparison Details

# a. Intended aim(s)

To evaluate the comparative risk of dementia onset between patients treated with <u>dihydropyridine CCBs versus hydrochlorothiazide</u> for hypertension.

# b. Primary endpoint

Incident dementia (i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere).

# 2. Person responsible for implementation of replication in Aetion

Mufaddal Mahesri

# 3. Data Source(s)

Medicare, 2008-2018

# 4. Study Design Diagrams





#### 5. Cohort Identification

## a. Cohort Summary

This study will employ a new user, active comparator, observational cohort study design comparing dihydropyridine CCBs to hydrochlorothiazide. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of dihydropyridine CCBs or hydrochlorothiazide (index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).

### b. Key details regarding cohort creation

#### Index date:

• Day of initiation of new dihydropyridine CCBs or hydrochlorothiazide use

## Inclusion criteria for analyses 1, 3, 4:

- Aged ≥ 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage
- No use of dihydropyridine CCBs, hydrochlorothiazide, or other antihypertensives, listed in section c, any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least two claims with hypertension diagnosis recorded in 365 days prior to index date

### Inclusion criteria for analysis 2:

- Aged > 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage
- No use of dihydropyridine CCBs, hydrochlorothiazide, or other antihypertensives, listed in section c, any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- At least two claims with hypertension diagnosis recorded in 365 days prior to index date
- 180-day continuous use of dihydropyridine CCBs or hydrochlorothiazide starting on the index date

# c. Antihypertensive drugs

| ACE inhibitors | |
|----------------|--------------|
| Benazepril | Moexipril |
| Captopril | Perindopril |
| Enalapril | Quinapril |
| Fosinopril | Ramipril |
| Lisinopril | Trandolapril |

| Beta-blockers | |
|---------------|--------------|
| Acebutolol | Levobunolol |
| Atenolol | Metipranolol |
| Betaxolol | Metoprolol |
| Bisprolol | Nadolol |
| Bucindolol | Penbutolol |
| Carteolol | Pindolol |
| Esmolol | Propranolol |
| Labetalol | Timolol |
| Landiolol | Nebivolol |

| Dihydropyridine CCBs | |
|----------------------|-------------|
| Amlodipine | Nifedipine |
| Felodipine | Nimodipine |
| Isradipine | Nisoldipine |
| Nicardipine | |

| Non-dihydropyridine CCBs | |
|--------------------------|------------|
| Bepridil | Mibefradil |
| Diltiazem | Verapamil |

| Diuretics | |
|---------------------|--------------------|
| Bendroflumethiazide | Quinethazone |
| Benzthiazide | Trichlormethiazide |
| Chlorothiazide | Bumetanide |
| Chlorthalidone | Torsemide |
| Cyclothiazide | Ethacrynic acid |
| Hydrochlorothiazide | Ethacrynate sodium |
| Hydroflumethiazide | Furosemide |
| Indapamide | Triamterene |
| Methyclothiazide | Amiloride |
| Metolazone | Spironolactone |
| Polythiazide | Eplerenone |

# d. Flowchart of the study cohort assembly

| | Less Excluded Patients | Remaining Patients |
|---|---|---|
| All patients | | 23,466,175 |
| Did not meet cohort entry criteria | -13,612,351 | 9,853,824 |
| Excluded due to insufficient enrollment | -3,966,812 | 5,887,012 |
| Excluded due to prior use of referent | -5,374,387 | 512,625 |
| Excluded based on Dementia Exclusion | -73,305 | 439,320 |
| Excluded based on Hypertension Diagnosis | -36,628 | 402,692 |
| Excluded based on Nursing Home Admission | -56,906 | 345,786 |
| Excluded based on prior use of Any Antihypertensive | -180,058 | 165,728 |
| Excluded because patient qualified in >1 exposure category | -410 | 165,318 |
| Excluded because patient did not begin follow-up | -1,598 | 163,720 |
| Patients in dihydropyridine CCB group | | 77,152 |
| Patients in hydrochlorothiazide group | | 86,568 |
| Final cohort | | 163,720 |

# 6. Variables

# a. Exposure-related variables:

# Study drug:

The study exposure of interest is initiation of dihydropyridine CCBs

# Comparator:

Initiators of dihydropyridine CCBs will be compared to initiators of hydrochlorothiazide

# b. Covariates:

| Demographics | |
|--------------|-----------------------------|
| Age | Region |
| Gender | Calendar year of index date |
| Race | Low income subsidy |

| Dementia risk factors | |
|-------------------------|------------------|
| Diabetes | Anxiety |
| Obesity | Bipolar disorder |
| Coronary artery disease | Schizophrenia |
| Depression | |

| Markers for healthy behavior, frailty, healthcare use | |
|---|---|
| Smoking | Number of hospitalizations |
| Mammography | Number of physician office visits |
| Colonoscopy | Number of serum creatinine tests ordered |
| Fecal occult blood test | Composite frailty score |
| Influenza vaccination | Number of C-reactive protein tests ordered |
| Pneumococcal vaccination | Osteoporosis |
| Herpes zoster vaccination | Fractures |

| Bone mineral density test | Falls |
|-----------------------------------|----------------------------|
| Number of distinct generic agents | Use of supplemental oxygen |
| Number of emergency room visits | Combined comorbidity score |
| Number of outpatient visits | |

| Comedication use | |
|---|---|
| Lithium | Nitrates |
| Anti-epileptic mood stabilizers | Lipid lowering drugs |
| Anti-epileptics (other than mood stabilizers) | Non-insulin diabetes medications |
| Atypical antipsychotics | Insulin |
| Benzodiazepines | Antidepressants |
| Serotonin-norepinephrine reuptake Inhibitors | Typical antipsychotics |
| Selective serotonin reuptake inhibitors | Anticoagulants |
| Tricyclic antidepressants (TCAs) | Antiplatelet agents |

| Comorbid conditions | |
|---|---|
| Atrial fibrillation | Chronic liver disease |
| Coronary artery disease | Asthma |
| Heart failure | Ischemic heart disease |
| Stroke or transient ischemic attack | Chronic obstructive pulmonary disease |
| Peripheral vascular disease | Malignancy |
| Hyperlipidemia | Drug or alcohol abuse or dependence |
| Renal dysfunction | Venous thromboembolism |

ICD-9, ICD-10, HCPCS, and NDC codes used to define the covariates listed above are available in Appendix A.

- c. Outcome variables and study follow-up:
- <u>Primary outcome</u>: incident dementia, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Outcome will be defined by 1 inpatient claim or 2 outpatient claims in analysis 1, 2, 3. In analysis 4, the outcome will be defined by 1 inpatient or 1 outpatient claims and 1 prescription claim for a symptomatic treatment [donepezil, galantamine, rivastigmine, and memantine] within 6 months of each other with outcome date assigned to second event in the sequence.
- Secondary outcomes: Individual component:

#### Alzheimer's disease

| Condition | ICD-9 and ICD-10 codes |
|---|---|
| Alzheimer's disease | 331.0*, F00*, G30* |
| Vascular dementia | 290.4*, F01* |
| Senile, presenile, or unspecified dementia | 290.0*, 290.1*. 290.3*, 797*, F03* |
| Dementia in other diseases classified elsewhere | 331.1*, 331.2*, 331.7*, 294.1*, F02* |

For analysis 1,3, and 4 the follow-up will start the day after initiation of dihydropyridine CCBs and hydrochlorothiazide and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (dihydropyridine CCBs and hydrochlorothiazide) plus a defined grace period (i.e., 90 days after the end of the last prescription's days' supply in main analyses).

For analysis 2, the follow-up will start 180 days after initiation of dihydropyridine CCBs and hydrochlorothiazide and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Maximum allowed follow-up time (1095 days) reached

# 7. Feasibility counts

| Analysis scheme | Total Dihydropyridine<br>CCB/HCTZ initiators | N outcome | Dementia Rate per<br>1,000 person-years<br>(95% CI) | Follow-up time in<br>days; Median [IQR] |
|---|---|---|---|---|
| 1: As treated | 77,152 (47.1%) | 2.611 | 16 10 (15 66 16 72) | 220 [70 604] |
| | 86,568 (52.9%) | 3,611 | 16.19 (15.66, 16.72) | 238 [79, 684] |
| 2: 6 mo induction period, 'as started' | 43,252 (46.6%) | 2 905 | 20.02 (20.26.21.57) | 926 [410, 1,005] |
| | 49,514 (53.4%) | 3,895 | 20.92 (20.26, 21.57) | 836 [410, 1,095] |
| 3: exclude 6 mo follow-up | 42,768 (46.5%) | 2.516 | 45 30 (14 70 45 00) | 424 [457 005] |
| (symptoms to claims period) | 49,150 (53.5%) | 2,516 | 15.38 (14.78, 15.99) | 434 [157, 885] |
| 4: Outcome Dx + Rx | 77,152 (47.1%) | 1 214 | E 40 (E 00 E 70) | 241 [01 601] |
| | 86,568 (52.9%) | 1,214 | 5.40 (5.09, 5.70) | 241 [81, 691] |

## 8. Propensity score analysis

We will use a propensity-score (PS)¹-based approach to account for measured confounding in this study. The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., the repurposing candidate) versus the reference drug conditional on baseline covariates using multivariable logistic regression constructed separately in each data source. On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. Therefore, analyses conditioned on the PS provide effect estimates that are free from measured confounding. For all our analyses, initiators of each exposure of interest will be matched with initiators of the reference exposure based on their PS within each data source.² Pair matching will be conducted using a nearest-neighbor algorithm, which seeks to minimize the distance between propensity scores in each pair of treated and reference patients,³ and a caliper of 0.025 on the natural scale of the PS will be used to ensure similarity between the matched patients.⁴

We report multiple diagnostics for PS analysis in this protocol. First, the PS distributional overlap is provided between two groups before and after matching to ensure comparability of these groups.<sup>5</sup> Next, balance in each individual covariate between two treatment groups is reported using standardized differences.<sup>6</sup>

# a. PS distributions stratified by treatment group

# Pre-matching propensity score overlap:



# Post-matching propensity score overlap:



# b. Table for covariate balance

| | Uni | matched | | | PS-Matched | |
|---|---|---|---|---|---|---|
| Variable | Dihydropyridine<br>CCBs<br>(N = 84,102) | Hydrochlorothiazide<br>(N = 92,119) | St. Diff | Dihydropyridine<br>CCBs<br>(N = 64,254) | Hydrochlorothiazide<br>(N = 64,254) | St. Diff |
| Demographics | | | | | | |
| Age, mean (SD) | 73.97 (7.17) | 72.80 (6.64) | 0.17 | 73.44 (6.85) | 73.48 (6.93) | -0.01 |
| Gender, n (%) | | | | | | |
| Male | 40,877 (48.6%) | 38,709 (42.0%) | 0.13 | 29,244 (45.5%) | 29,337 (45.7%) | 0.00 |
| Female | 43,225 (51.4%) | 53,410 (58.0%) | -0.13 | 35,010 (54.5%) | 34,917 (54.3%) | 0.00 |
| Race, n (%) | | | | | | |
| White | 60,095 (71.5%) | 70,611 (76.7%) | -0.12 | 47,346 (73.7%) | 47,312 (73.6%) | 0.00 |
| Black | 11,436 (13.6%) | 10,523 (11.4%) | 0.07 | 8,092 (12.6%) | 8,107 (12.6%) | 0.00 |
| Asian | 5,260 (6.3%) | 3,544 (3.8%) | 0.11 | 3,295 (5.1%) | 3,280 (5.1%) | 0.00 |
| Hispanic | 3,089 (3.7%) | 3,604 (3.9%) | -0.01 | 2,463 (3.8%) | 2,466 (3.8%) | 0.00 |
| Native American | 668 (0.8%) | 681 (0.7%) | 0.01 | 471 (0.7%) | 472 (0.7%) | 0.00 |
| Unknown | 856 (1.0%) | 811 (0.9%) | 0.01 | 646 (1.0%) | 655 (1.0%) | 0.00 |
| Region, n (%) | | | | | | |
| Northeast; n (%) | 18,248 (21.7%) | 17,640 (19.1%) | 0.06 | 13,566 (21.1%) | 13,590 (21.2%) | 0.00 |
| South; n (%) | 34,062 (40.5%) | 39,651 (43.0%) | -0.05 | 26,587 (41.4%) | 26,540 (41.3%) | 0.00 |
| Midwest; n (%) | 14,789 (17.6%) | 17,959 (19.5%) | -0.05 | 11,556 (18.0%) | 11,569 (18.0%) | 0.00 |
| West; n (%) | 17,003 (20.2%) | 16,869 (18.3%) | 0.05 | 12,545 (19.5%) | 12,555 (19.5%) | 0.00 |
| Calendar year of index date, n (%) | | | | | | |
| 2008 | 7,577 (9.0%) | 12,853 (14.0%) | -0.16 | 6,730 (10.5%) | 6,532 (10.2%) | 0.01 |
| 2009 | 4,626 (5.5%) | 7,329 (8.0%) | -0.10 | 4,054 (6.3%) | 3,965 (6.2%) | 0.00 |
| 2010 | 3,323 (4.0%) | 5,367 (5.8%) | -0.08 | 2,867 (4.5%) | 2,891 (4.5%) | 0.00 |
| 2011 | 2,617 (3.1%) | 3,933 (4.3%) | -0.06 | 2,241 (3.5%) | 2,194 (3.4%) | 0.01 |

| 2012 | 1,939 (2.3%) | 2,505 (2.7%) | -0.03 | 1,604 (2.5%) | 1,607 (2.5%) | 0.00 |
|---|---|---|---|---|---|---|
| 2013 | 18,406 (21.9%) | 19,616 (21.3%) | 0.01 | 14,158 (22.0%) | 14,176 (22.1%) | 0.00 |
| 2014 | 14,482 (17.2%) | 14,256 (15.5%) | 0.05 | 10,810 (16.8%) | 10,852 (16.9%) | 0.00 |
| 2015 | 12,149 (14.4%) | 10,439 (11.3%) | 0.09 | 8,471 (13.2%) | 8,569 (13.3%) | 0.00 |
| 2016 | 6,121 (7.3%) | 5,395 (5.9%) | 0.06 | 4,409 (6.9%) | 4,510 (7.0%) | 0.00 |
| 2017 | 5,933 (7.1%) | 4,897 (5.3%) | 0.07 | 4,125 (6.4%) | 4,147 (6.5%) | 0.00 |
| 2018 | 6,929 (8.2%) | 5,529 (6.0%) | 0.09 | 4,785 (7.4%) | 4,811 (7.5%) | 0.00 |
| Low income subsidy, n (%) | 22,550 (26.8%) | 21,688 (23.5%) | 0.08 | 16,102 (25.1%) | 16,071 (25.0%) | 0.00 |
| Dementia risk factors, n (%) | | | | | | |
| Diabetes | 57,634 (68.5%) | 66,738 (72.4%) | -0.09 | 45,146 (70.3%) | 45,024 (70.1%) | 0.00 |
| Obesity | 12,536 (14.9%) | 14,948 (16.2%) | -0.04 | 9,833 (15.3%) | 9,872 (15.4%) | 0.00 |
| Coronary artery disease | 23,415 (27.8%) | 18,050 (19.6%) | 0.19 | 15,043 (23.4%) | 15,080 (23.5%) | 0.00 |
| Depression | 11,217 (13.3%) | 10,868 (11.8%) | 0.05 | 7,885 (12.3%) | 7,906 (12.3%) | 0.00 |
| Anxiety | 10,337 (12.3%) | 9,587 (10.4%) | 0.06 | 7,268 (11.3%) | 7,252 (11.3%) | 0.00 |
| Bipolar disorder | 1,154 (1.4%) | 967 (1.0%) | 0.04 | 747 (1.2%) | 763 (1.2%) | 0.00 |
| Schizophrenia | 718 (0.9%) | 603 (0.7%) | 0.02 | 468 (0.7%) | 465 (0.7%) | 0.00 |
| Markers for healthy behavior, frailty, healthcare use | | | | | | |
| Smoking, n (%) | 19,064 (22.7%) | 13,987 (15.2%) | 0.19 | 11,693 (18.2%) | 11,694 (18.2%) | 0.00 |
| Mammography, n (%) | 13,593 (16.2%) | 18,485 (20.1%) | -0.10 | 11,762 (18.3%) | 11,659 (18.1%) | 0.01 |
| Colonoscopy, n (%) | 8,820 (10.5%) | 9,946 (10.8%) | -0.01 | 6,772 (10.5%) | 6,720 (10.5%) | 0.00 |
| Fecal occult blood test, n (%) | 6,726 (8.0%) | 7,984 (8.7%) | -0.03 | 5,380 (8.4%) | 5,327 (8.3%) | 0.00 |
| Influenza vaccination, n (%) | 46,348 (55.1%) | 50,992 (55.4%) | -0.01 | 35,620 (55.4%) | 35,580 (55.4%) | 0.00 |
| Pneumococcal vaccination, n (%) | 19,455 (23.1%) | 17,866 (19.4%) | 0.09 | 13,934 (21.7%) | 14,028 (21.8%) | 0.00 |
| Bone mineral density test, n (%) | 38 (0.0%) | 50 (0.1%) | -0.04 | 33 (0.1%) | 33 (0.1%) | 0.00 |
| Number of distinct prescriptions, mean (SD) | 9.06 (5.42) | 8.53 (5.16) | 0.10 | 8.75 (5.20) | 8.73 (5.32) | 0.00 |
| Number of emergency room visits, mean (SD) | 0.75 (1.42) | 0.47 (1.05) | 0.22 | 0.57 (1.13) | 0.56 (1.16) | 0.01 |
| Number of outpatient visits, mean (SD) | 12.17 (17.93) | 11.46 (15.93) | 0.04 | 11.95 (17.95) | 11.94 (16.28) | 0.00 |

| Number of hospitalizations, mean (SD) | 0.50 (0.89) | 0.23 (0.59) | 0.36 | 0.31 (0.64) | 0.30 (0.68) | 0.02 |
|---|---|---|---|---|---|---|
| Number of physician office visits, mean (SD) | 4.89 (11.60) | 4.86 (10.44) | 0.00 | 4.95 (11.86) | 4.94 (10.65) | 0.00 |
| Number of C-reactive protein tests ordered, mean (SD) | 0.20 (0.80) | 0.19 (0.74) | 0.01 | 0.20 (0.76) | 0.20 (0.75) | 0.00 |
| Number of serum creatinine tests ordered, mean (SD) | 3.12 (3.26) | 2.78 (2.48) | 0.12 | 2.92 (2.79) | 2.90 (2.65) | 0.01 |
| Composite frailty score, mean (SD) | 0.18 (0.06) | 0.17 (0.05) | 0.18 | 0.18 (0.05) | 0.18 (0.05) | 0.00 |
| Osteoporosis, n (%) | 10,688 (12.7%) | 10,862 (11.8%) | 0.03 | 7,973 (12.4%) | 7,938 (12.4%) | 0.00 |
| Fractures, n (%) | 5,444 (6.5%) | 4,941 (5.4%) | 0.05 | 3,707 (5.8%) | 3,719 (5.8%) | 0.00 |
| Falls, n (%) | 3,458 (4.1%) | 2,864 (3.1%) | 0.05 | 2,200 (3.4%) | 2,185 (3.4%) | 0.00 |
| Use of supplemental oxygen, n (%) | 1,341 (1.6%) | 713 (0.8%) | 0.07 | 674 (1.0%) | 646 (1.0%) | 0.00 |
| Combined comorbidity score, mean (SD) | 3.77 (2.55) | 2.82 (1.96) | 0.42 | 3.17 (2.11) | 3.17 (2.12) | 0.00 |
| Comedication use, n (%) | | | | | | |
| Lithium | 214 (0.3%) | 125 (0.1%) | 0.04 | 105 (0.2%) | 115 (0.2%) | 0.00 |
| Anti-epileptic mood stabilizers | 1,194 (1.4%) | 1,039 (1.1%) | 0.03 | 786 (1.2%) | 817 (1.3%) | -0.01 |
| Anti-epileptics (other than mood stabilizers) | 10,125 (12.0%) | 10,191 (11.1%) | 0.03 | 7,319 (11.4%) | 7,241 (11.3%) | 0.00 |
| Atypical antipsychotics | 1,789 (2.1%) | 1,585 (1.7%) | 0.03 | 1,187 (1.8%) | 1,208 (1.9%) | -0.01 |
| Benzodiazepines | 8,850 (10.5%) | 8,105 (8.8%) | 0.06 | 6,385 (9.9%) | 6,414 (10.0%) | 0.00 |
| Serotonin-norepinephrine reuptake inhibitors | 3,030 (3.6%) | 3,370 (3.7%) | -0.01 | 2,327 (3.6%) | 2,331 (3.6%) | 0.00 |
| Selective serotonin reuptake inhibitors | 10,010 (11.9%) | 10,833 (11.8%) | 0.00 | 7,512 (11.7%) | 7,472 (11.6%) | 0.00 |
| Tricyclic antidepressants (TCAs) | 2,429 (2.9%) | 2,813 (3.1%) | -0.01 | 1,875 (2.9%) | 1,780 (2.8%) | 0.01 |
| Typical antipsychotics | 385 (0.5%) | 364 (0.4%) | 0.01 | 256 (0.4%) | 259 (0.4%) | 0.00 |
| Anticoagulants | 5,110 (6.1%) | 4,654 (5.1%) | 0.04 | 3,562 (5.5%) | 3,501 (5.4%) | 0.00 |
| Antiplatelet agents | 9,820 (11.7%) | 6,533 (7.1%) | 0.16 | 5,674 (8.8%) | 5,690 (8.9%) | 0.00 |
| Nitrates | 5,497 (6.5%) | 3,329 (3.6%) | 0.13 | 3,040 (4.7%) | 3,028 (4.7%) | 0.00 |
| Lipid lowering drugs | 46,937 (55.8%) | 51,602 (56.0%) | 0.00 | 35,627 (55.4%) | 35,605 (55.4%) | 0.00 |
| Non-insulin diabetes medications | 31,333 (37.3%) | 41,954 (45.5%) | -0.17 | 26,022 (40.5%) | 25,941 (40.4%) | 0.00 |

| Insulin | 9,749 (11.6%) | 9,237 (10.0%) | 0.05 | 6,812 (10.6%) | 6,766 (10.5%) | 0.00 |
|---|---|---|---|---|---|---|
| Antidepressants | 16,567 (19.7%) | 17,906 (19.4%) | 0.01 | 12,432 (19.3%) | 12,306 (19.2%) | 0.00 |
| Comorbid conditions, n (%) | | | | | | |
| Atrial fibrillation | 7,462 (8.9%) | 5,612 (6.1%) | 0.11 | 4,678 (7.3%) | 4,664 (7.3%) | 0.00 |
| Heart failure | 11,641 (13.8%) | 8,192 (8.9%) | 0.15 | 6,833 (10.6%) | 6,906 (10.7%) | 0.00 |
| Stroke or transient ischemic attack | 11,828 (14.1%) | 6,556 (7.1%) | 0.23 | 6,107 (9.5%) | 6,119 (9.5%) | 0.00 |
| Peripheral vascular disease | 12,670 (15.1%) | 10,411 (11.3%) | 0.11 | 8,413 (13.1%) | 8,318 (12.9%) | 0.01 |
| Hyperlipidemia | 67,245 (80.0%) | 75,032 (81.5%) | -0.04 | 51,808 (80.6%) | 51,804 (80.6%) | 0.00 |
| Renal dysfunction | 20,650 (24.6%) | 10,046 (10.9%) | 0.36 | 9,729 (15.1%) | 9,670 (15.0%) | 0.00 |
| Chronic liver disease | 6,381 (7.6%) | 5,492 (6.0%) | 0.06 | 4,301 (6.7%) | 4,322 (6.7%) | 0.00 |
| Asthma | 10,723 (12.7%) | 10,329 (11.2%) | 0.05 | 7,691 (12.0%) | 7,736 (12.0%) | 0.00 |
| Ischemic heart disease | 25,168 (29.9%) | 20,034 (21.7%) | 0.19 | 16,486 (25.7%) | 16,579 (25.8%) | 0.00 |
| Chronic obstructive pulmonary disease | 17,814 (21.2%) | 15,798 (17.1%) | 0.10 | 12,232 (19.0%) | 12,133 (18.9%) | 0.00 |
| Malignancy | 22,389 (26.6%) | 21,557 (23.4%) | 0.07 | 16,078 (25.0%) | 16,184 (25.2%) | 0.00 |
| Drug or alcohol abuse or dependence | 9,725 (11.6%) | 7,347 (8.0%) | 0.12 | 6,048 (9.4%) | 6,009 (9.4%) | 0.00 |
| Venous thromboembolism | 3,415 (4.1%) | 2,835 (3.1%) | 0.05 | 2,169 (3.4%) | 2,127 (3.3%) | 0.01 |

## 9. Statistical analysis plans

Incidence rates for the outcome will be estimated for the treatment and reference groups before and after PS matching. The competing risk of death could be of concern for the current set of analyses if mortality is frequent among patients included in the cohort and if differences in the risk of mortality between treatment and reference groups are substantial. In the PS-matched sample, we will use cause-specific hazard models<sup>7</sup> to provide hazard ratios averaged over the entire follow-up period as well as interval specific hazard ratios (1, 2, and 3 years) for the association between the treatment of interest and risk of ADRD after considering all-cause mortality as a competing event. Pre-specified subgroup analyses will be conducted based on age, sex, and baseline cardiovascular disease. In addition to the Medicare dataset, we will pursue a similar analysis within Clinical Practice Research Datalink (CPRD), a UK population health dataset, to validate our results.

### 10. References

- 1. Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.
- 2. Rassen JA, Avorn J, Schneeweiss S. Multivariate-adjusted pharmacoepidemiologic analyses of confidential information pooled from multiple health care utilization databases. *Pharmacoepidemiology and drug safety.* 2010;19(8):848-857.
- **3.** Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. *Pharmacoepidemiol Drug Saf.* May 2012;21 Suppl 2:69-80.
- **4.** Austin PC. Some Methods of Propensity-Score Matching had Superior Performance to Others: Results of an Empirical Investigation and Monte Carlo simulations. *Biometrical Journal*. 2009;51(1):171-184.
- 5. AM Walker AM, Patrick A, Lauer M, et al. Tool for Assessing the Feasibility of Comparative Effectiveness Research. Comp Effect Res 2013;3:11-20.
- **6.** Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Statistics in medicine*. May 10 2014;33(10):1685-1699.
- 7. Austin PC, Lee DS, Fine JP. Introduction to the analysis of survival data in the presence of competing risks. *Circulation*. 2016;133(6):601-609.

| | EXPOSURE vs. COMPARISON |
|---|---|
| Dihydropyridine CCBs vs Hydrochlorothiazide | |
| | INCLUSION CRITERIA |
| | on the index date |
| Hypertension diagnosis Measured 365 d | ays prior to drug initiation for at least two claims in any diagnosis position and inpatient or outpatient outpatient setting – |
| 2 Issaultanasia | |
| - | 401.1, 401.9, 402.10, 402.90, 404.10, 404.90, 405.11, 405.19, 405.99 |
| | – 110-115.x, N26.2 |
| 3 Sufficient enrollment Medicare Part A | B, and D enrollment with no HMO coverage for 365 days prior to and on the cohort entry date |
| The state of the s | EXCLUSION CRITERIA |
| Prior history of dementia Measured any | time prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| ICD9 disanceis | - 046.1x, 290.xx (excluding 290.8), 291.2, 292.82, 294.1x, 294.2x, 331.0-331.2, 331.7, 331.82, 331.83, 333.4, 780.93, 797 |
| _ | s = F01.xx-F03.xx, G30.xx-G31.85, F41.xx |
| 1 | |
| NDC brand nam | ie – ""ARICEPT", "ARICEPT ODT", "EXELON", "NAMENDA", "NAMENDA XR", "NAMZARIC", "RAZADYNE", "RAZADYNE ER", or "REMINYL" |
| | me – "DONEPEZIL HCL", "GALANTAMINE HBR", "MEMANTINE HCL", "MEMANTINE HCL/DONEPEZIL HCL", "RIVASTIGMINE", or "RIVASTIGMINE |
| TARTRATE" | |
| No prior use of antihypertensive medications NDC generic name | ne – "AMLODIPINE BESYLATE/BENAZEPRIL HCL", "BENAZEPRIL HCL", "BENAZEPRIL HCL/HYDROCHLOROTHIAZIDE", "CAPTOPRIL", "CAPTOPRIL'HYDROCHLOROTHIAZIDE", |
| | LEATE", "ENALAPRIL MALEATE/DILTIAZEM MALATE", "ENALAPRIL MALEATE/FELODIPINE", "ENALAPRIL MALEATE/HYDROCHLOROTHIAZIDE", "ENALAPRILAT DIHYDRATE", |
| "FOSINOPRIL SO | DDIUM", "FOSINOPRIL SODIUM/HYDROCHLOROTHIAZIDE", "LISINOPRIL", "LISINOPRIL/DIETARY SUPPLEMENT,COMB.10", "LISINOPRIL/HYDROCHLOROTHIAZIDE", "MOEXIPRIL |
| HCL", "MOEXIPF | RIL HCL/HYDROCHLOROTHIAZIDE", "PERINDOPRIL ARGININE/AMLODIPINE BESYLATE", "PERINDOPRIL ERBUMINE", "QUINAPRIL HCL", "QUINAPRIL |
| HCL/HYDROCHL | DROTHIAZIDE", "RAMIPRIL", "TRANDOLAPRIL", "TRANDOLAPRIL/VERAPAMIL HCL", "ACEBUTOLOL HCL", "ATENOLOL", "ATENOLOL/CHLORTHALIDONE", "BETAXOLOL HCL", |
| "BISOPROLOL F | JMARATE", "BISOPROLOL FUMARATE/HYDROCHLOROTHIAZIDE", "BRIMONIDINE TARTRATE/TIMOLOL MALEATE", "CARTEOLOL HCL", "DORZOLAMIDE HCL/TIMOLOL |
| MALEATE", "DO | RZOLAMIDE HCL/TIMOLOL MALEATE/PF", "ESMOLOL HCL", "ESMOLOL HCL IN SODIUM CHLORIDE, ISO-OSMOTIC", "ESMOLOL HCL IN STERILE WATER", "LABETALOL HCL", |
| | DEXTROSE 5 % IN WATER", "LEVOBUNOLOL HCL", "METIPRANOLOL", "METOPROLOL SUCCINATE", "METOPROLOL SUCCINATE/HYDROCHLOROTHIAZIDE", "METOPROLOL |
| TARTRATE", "M | ETOPROLOL TARTRATE/DIETARY SUPPLEMENT,COMB.10", "METOPROLOL TARTRATE/HYDROCHLOROTHIAZIDE", "NADOLOL", "NADOLOL/BENDROFLUMETHIAZIDE", |
| | L", "NEBIVOLOL HCL/VALSARTAN", "PENBUTOLOL SULFATE", "PINDOLOL", "PROPRANOLOL HCL", "PROPRANOLOL HCL/HYDROCHLOROTHIAZIDE", "TIMOLOL", "TIMOLOL" |
| | NIDINE TAR/DORZOLAMIDE HCL/LATANOPROST/PF", "TIMOLOL MALEATE", "TIMOLOL MALEATE/BRIMONIDINE TARTRATE/DORZOLAMIDE HCL/PF", "TIMOLOL |
| | COLAMIDE HCL/LATANOPROST/PF", "TIMOLOL MALEATE/HYDROCHLOROTHIAZIDE", "TIMOLOL MALEATE/LATANOPROST/PRESERVATIVE FREE", "TIMOLOL MALEATE/PF", |
| | IIFUMARATE/AMLODIPINE BESYLATE", "ALISKIREN HEMIFUMARATE/AMLODIPINE/HYDROCHLOROTHIAZIDE", "AMLODIPINE BESYLATE", "AMLODIPINE |
| | RVASTATIN CALCIUM", "AMLODIPINE BESYLATE/BENAZEPRIL HCL", "AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL", "AMLODIPINE BESYLATE/VALSARTAN", |
| | ESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE", "BEPRIDIL HCL", "DILTIAZEM HCL", "DILTIAZEM HCL IN 0.9 % SODIUM CHLORIDE", "DILTIAZEM HCL/DEXTROSE 5 % IN |
| | AZEM MALATE", "ENALAPRIL MALEATE/DILTIAZEM MALATE", "ENALAPRIL MALEATE/FELODIPINE", "FELODIPINE", "ISRADIPINE", "MIBARRIL DI-HCL", "NICARDIPINE HCL", |
| | CL IN 0.9 % SODIUM CHLORIDE", "NICARDIPINE IN 5 % DEXTROSE IN WATER", "NICARDIPINE IN DEXTROSE, ISO-OSMOTIC", "NICARDIPINE IN SODIUM CHLORIDE, ISO-<br>EDIPINE", "NIFEDIPINE, MICRONIZED", "NIMODIPINE", "NISOLDIPINE", "OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZIDE", "PERINDOPRIL |
| | ODIPINE BESYLATE", "TELMISARTAN/AMLODIPINE BESYLATE", "TRANDOLAPRIL/VERAPAMIL HCL", "VERAPAMIL HCL", "ALISKIREN |
| | E/AMLODIPINE/HYDROCHLOROTHIAZIDE", "ALISKIREN HEMIFUMARATE/HYDROCHLOROTHIAZIDE", "AMILORIDE HCL", "AMILORIDE HCL," HYDROCHLOROTHIAZIDE", |
| | ESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE", "ATENOLOL/CHLORTHALIDONE", "AZILSARTAN MEDOXOMIL/CHLORTHALIDONE", "BENAZEPRIL |
| | DROTHIAZIDE", "BENDROFLUMETHIAZIDE", "BISOPROLOL FUMARATE/HYDROCHLOROTHIAZIDE", "BUMETANIDE", "CANDESARTAN CILEXETIL/HYDROCHLOROTHIAZIDE", " |
| | DROCHLOROTHIAZIDE", "CHLOROTHIAZIDE", "CHLOROTHIAZIDE SODIUM", "CHLORTHALIDONE", "CLONIDINE HCL/CHLORTHALIDONE", |
| | HYDROCHLOROTHIAZIDE", "DESERPIDINE/METHYCLOTHIAZIDE", "ENALAPRIL MALEATE/HYDROCHLOROTHIAZIDE", "EPLERENONE", "EPROSARTAN |
| | ROCHLOROTHIAZIDE", "ETHACRYNATE SODIUM", "ETHACRYNIC ACID", "FOSINOPRIL SODIUM/HYDROCHLOROTHIAZIDE", "FUROSEMIDE", "FUROSEMIDE IN 0.9 % SODIUM |
| | ROSEMIDE/DEXTROSE 5 % IN WATER", "GUANETHIDINE SULFATE/HYDROCHLOROTHIAZIDE", "HYDRALAZINE HCL/HYDROCHLOROTHIAZIDE", "HYDRALAZINE |
| II I | /HYDROCHLOROTHIAZIDE", "HYDROCHLOROTHIAZIDE", "HYDROFLUMETHIAZIDE", "INDAPAMIDE", "IRBESARTAN/HYDROCHLOROTHIAZIDE", |
| 1 1 | DROCHLOROTHIAZIDE", "LOSARTAN POTASSIUM/HYDROCHLOROTHIAZIDE", "METHYCLOTHIAZIDE", "METHYLDOPA/CHLOROTHIAZIDE", |
| | 'HYDROCHLOROTHIAZIDE", "METOLAZONE", "METOPROLOL SUCCINATE/HYDROCHLOROTHIAZIDE", "METOPROLOL TARTRATE/HYDROCHLOROTHIAZIDE", "MOEXIPRIL |
| HCL/HYDROCHL | DROTHIAZIDE", "NADOLOL/BENDROFLUMETHIAZIDE", "OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZIDE", "OLMESARTAN |
| MEDOXOMIL/H | YDROCHLOROTHIAZIDE", "POLYTHIAZIDE", "PRAZOSIN HCL/POLYTHIAZIDE", "PROPRANOLOL HCL/HYDROCHLOROTHIAZIDE", "QUINAPRIL HCL/HYDROCHLOROTHIAZIDE", |
| "RAUWOLFIA SI | RPENTINA/BENDROFLUMETHIAZIDE", "RESERPINE/CHLOROTHIAZIDE", "RESERPINE/HYDROCHLOROTHIAZIDE", "RESERPINE/HYDROFLUMETHIAZIDE", |
| | THYCLOTHIAZIDE", "RESERPINE/POLYTHIAZIDE", "SPIRONOLACTONE", "SPIRONOLACTONE, MICRONIZED", "SPIRONOLACTONE/HYDROCHLOROTHIAZIDE", |
| "TELMISARTAN | /HYDROCHLOROTHIAZIDE", "TIMOLOL MALEATE/HYDROCHLOROTHIAZIDE", "TORSEMIDE", "TRIAMTERENE", "TRIAMTERENE/HYDROCHLOROTHIAZIDE", |
| "TRICHLORMET | HIAZIDE", "VALSARTAN/HYDROCHLOROTHIAZIDE" |

| Covariate list | |
|---|---|
| Catagony | Potential confounders |
| Category | ICD-9 |
| | Age |
| | Gender |
| Demographics | Race |
| 20mograpmos | Region |
| | Calendar year of index date |
| | Low income subsidy |
| | Diabetes |
| | Obesity |
| | Coronary artery disease |
| Dementia risk factors | Depression |
| | Anxiety |
| | Bipolar disorder |
| | Schizophrenia |
| | Smoking |
| | Mammography |
| | Colonoscopy |
| Lifestyle factors and markers for healthy behavior | Fecal occult blood test |
| • | Influenza vaccination |
| | Pneumococcal vaccination |
| | Herpes zoster vaccination |
| | BMD test |
| | Number of distinct generic agents |
| | Number of emergency room visits |
| Hardelland Planta and a second | Number of outpatient visits |
| Healthcare utilization measures | Number of hospitalizations |
| | Number of physician office visits |
| | Number of CRP tests ordered |
| | Number of serum creatinine tests ordered |
| | Commonite firstly |
| | Composite frailty score |
| | Osteoporosis |
| Frailty markers | Fractures |
| | Falls |
| | Use of supplemental oxygen |
| | A combined comorbidity score |
| | Lithium |
| | Lithium |
| | Anti-epileptic mood stabilizers Anti-epileptics (other than mood stabilizers) |
| | Atypical antipsychotics |
| | Benzodiazepines |

| | SNRIs |
|---------------------|-------------------------------------|
| | SSRIs |
| Comedications | TCAs |
| Comedications | Typical antipsychotics |
| | Anticoagulants |
| | Antiplatelet agents |
| | Nitrates |
| | Lipid lowering drugs |
| | Non-insulin diabetes medications |
| | Insulin |
| | Antidepressants |
| | Atrial fibrillation |
| | Coronary artery disease |
| | Heart failure |
| | Stroke or TIA |
| | Peripheral vascular disease |
| | Diabetes |
| | Hyperlipidemia |
| Comorbid conditions | Renal dysfunction |
| | Chronic liver disease |
| | Asthma |
| | Ischemic heart disease |
| | COPD |
| | Malignancy |
| | Drug or alcohol abuse or dependence |
| | VTE |

# Appendix A Demographics

| Calendar year of index date |
|-----------------------------|
| Year |
| 2008 |
| 2009 |
| 2010 |
| 2011 |
| 2012 |
| 2013 |
| 2014 |
| 2015 |
| 2016 |
| 2017 |
| 2018 |

### Low income subsidy

https://www.cms.gov/Medicare/Eligibility-and-Enrollment/LowIncSubMedicarePresCov/Downloads/StateLISGuidance021009.pdf

#### Diabetes


| E133519 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, right eye E133522 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, right eye E133523 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye E133523 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment involving the macula, bilateral E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment involving the macula, unspecified eye E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with macular edema, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye |
|---|---|
| E133521 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, right eye E133522 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye E133523 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment on involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified diabetes mellitus with proliferative diabetic retinopathy E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy | Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye |
| retinopathy with traction retinal detachment involving the macula, right eye E133522 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye E133523 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, left eye E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye | retinopathy with traction retinal detachment involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye |
| E133522 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with craction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment and detachment and rhegmatogenous retinal detachment and detachment and rhegmatogenous retinal detachment and detachment and rhegmatogenous retinal detachment and detachment and detachment and detachment and detachment and detachm |
| E133522 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye E133523 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with cardinor retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with crombined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment and detachment and rhegmatogenous retinal detachment and detachment and rhegmatogenous retinal detachment and detachment and rhegmatogenous retinal detachment and detachment and detachment and detachment and detachment and detachment and detachment and detachm |
| retinopathy with traction retinal detachment involving the macula, left eye 133523 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral 13529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye 13531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye 13532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye 13533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye 13533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral 1513539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye 1513541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment and rhegmatogenous retinal detachment, right eye 1513542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with traction retinal detachment involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye |
| E133523 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment involving the macula, bilateral E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye E133542 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye |
| retinopathy with traction retinal detachment involving the macula, bilateral E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment involving the macula, unspecified eye E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with traction retinal detachment involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Proliferative diabetic retinopathy Proliferative diabetic retinopathy |
| E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment involving the macula, unspecified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye | macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Proliferative diabetic retinopathy Proliferative diabetic retinopathy |
| E133529 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment involving the macula, unspecified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye | macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Proliferative diabetic retinopathy Proliferative diabetic retinopathy |
| retinopathy with traction retinal detachment involving the macula, unspecified eye E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with traction retinal detachment involving the macula, unspecified eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy 36203 Proliferative diabetic retinopathy 36204 Proliferative diabetic retinopathy 36205 Proliferative diabetic retinopathy 36206 Proliferative diabetic retinopathy |
| E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | macula, unspecified eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy 36203 Proliferative diabetic retinopathy 36204 Proliferative diabetic retinopathy 36205 Proliferative diabetic retinopathy 36206 Proliferative diabetic retinopathy 36207 Proliferative diabetic retinopathy |
| E133531 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy Proliferative diabetic retinopathy |
| retinopathy with traction retinal detachment not involving the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with reaction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with traction retinal detachment not involving the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Proliferative diabetic retinopathy Proliferative diabetic retinopathy Proliferative diabetic retinopathy |
| the macula, right eye E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye E133542 136202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | the macula, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified deye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy Proliferative diabetic retinopathy |
| E133532 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 Nother specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and retinopathy with combined traction retinal detachment and retinopathy with combined traction retinal detachment and retinopathy with combined traction retinal detachment and retinopathy with combined traction retinal detachment and |
| retinopathy with traction retinal detachment not involving the macula, left eye E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye Proliferative diabetic retinopathy Proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with traction retinal detachment not involving the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy Other specified diabetes mellitus with proliferative diabetic retinopathy Proliferative diabetic retinopathy Proliferative diabetic retinopathy |
| E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye E133542 Proliferative diabetic retinopathy | the macula, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| E133533 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye Proliferative diabetic retinopathy | Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with traction retinal detachment not involving the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and retinopathy with combined traction retinal detachment and |
| the macula, bilateral E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | the macula, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| E133539 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye Proliferative diabetic retinopathy | Other specified diabetes mellitus with proliferative diabetic retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and retinopathy with combined traction retinal detachment and |
| retinopathy with traction retinal detachment not involving the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with traction retinal detachment not involving the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| the macula, unspecified eye E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | the macula, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| E133541 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye E133542 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye Proliferative diabetic retinopathy | retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| rhegmatogenous retinal detachment, right eye E133542 Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| E133542 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with combined traction retinal detachment and |
| retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, left eye | retinopathy with combined traction retinal detachment and |
| rhegmatogenous retinal detachment, left eye | |
| | rhegmatogenous retinal detachment, left eye |
| E1225/2 26202 Other specified diphotes mollitus with proliferative diphote Dialiferative diphote retinantity. | • |
| TEACHER TO A DECLE SOLUTION OF THE SOLUTION OF | 36202 Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy |
| | n ecinopachy with compined traction retinal detachment and I |
| E133549 36202 Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy | retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, bilateral |
| | rhegmatogenous retinal detachment, bilateral |
| reunopatny with combined traction retinal detachment and | rhegmatogenous retinal detachment, bilateral |
| retinopatny with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative Proliferative diabetic retinopathy |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy Other specified diabetes mellitus with stable proliferative diabetic retinopathy |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye E133553 diabetic retinopathy, bilateral | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy Other specified diabetes mellitus with stable proliferative diabetic retinopathy Proliferative diabetic retinopathy |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye Proliferative diabetic retinopathy Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 Yellow Proliferative diabetic retinopathy retinopathy without macular edema, right eye | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy diabetic retinopathy unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, right eye E133592 36202 Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy |
| E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133592 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, right eye E133592 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye |
| E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy mithout macular edema, right eye E133592 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye E133593 36202 Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy retinopathy without macular edema, left eye E133593 Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, right eye E133592 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye E133593 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye E133593 York Proliferative diabetic retinopathy retinopathy without macular edema, bilateral | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, bilateral |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133592 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, right eye E133593 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye E133599 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, bilateral E133599 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy Proliferative diabetic retinopathy retinopathy without macular edema, bilateral E133599 7016 Proliferative diabetic retinopathy Proliferative diabetic retinopathy | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy |
| rhegmatogenous retinal detachment, unspecified eye E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, right eye E133592 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye E133593 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye E133593 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye E133593 York Specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, bilateral | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy |
| E133551 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, right eye E133552 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, left eye E133553 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, bilateral E133559 36202 Other specified diabetes mellitus with stable proliferative diabetic retinopathy diabetic retinopathy, unspecified eye E133591 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye E133592 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, left eye E133593 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, bilateral E133599 36202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, bilateral E133599 76202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, unspecified eye E133599 76202 Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, unspecified eye | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, right eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, left eye Other specified diabetes mellitus with stable proliferative diabetic retinopathy, bilateral Other specified diabetes mellitus with stable proliferative diabetic retinopathy, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, right eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, left eye Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, unspecified eye Other specified diabetes mellitus with proliferative diabetic retinopathy retinopathy without macular edema, unspecified eye |
| retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, bilateral E133549 36202 Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy | |
| | Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy |
| E122542 26202 Other specified dishetes mollitus with preliferative dishetic Preliferative dishetic retinantity. | |
| rhegmatogenous retinal detachment, left eye | |
| rhegmatogenous retinal detachment, left eye | |
| | rhegmatogenous retinal detachment, left eye |
| rhegmatogenous retinal detachment, left eye | |
| | rhegmatogenous retinal detachment, left eye |
| | rhegmatogenous retinal detachment, left eye |
| | rhegmatogenous retinal detachment, left eye |
| | integriatogenous retinal detaciment, rett eye |
| E1225/2 26202 Other specified dishetes multiple with evaliforative dishetic Dreliferative dishetic retires the | |
| E1225/2 26202 Other specified dispetes mollitus with proliferative dispeties dispeties dispeties retinantity. | |
| E1325/2 26202 Other specified diphotos mollifus with proliferative diphotos diphotos retires attached | |
| E1225/2 26202 Other specified dishetes multiple with proliferative dishetic Proliferative dishetic retires the | |
| E1225/2 26202 Other energified dishetes mollitus with proliferative dishetic Proliferative dishetic retinanting | |
| | 00000 Obber and effect dishere and like a with and if and it. Deslife and it and it and it and it. |
| ELECTION I DESCRIPTION AND THE SUBMITTED INTO THE PROPERTY OF | 36202 Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy |
| | 00000 Other specified dishetes mollitus with multi-matical dishets. Desliferant and the street was the |
| E1325/2 26202 Other specified dispetes mallitus with proliferative dispeties dispeties dispeties attached | |
| | rnegmatogenous retinai detacnment, ieπ eye |
| | rhegmatogenous retinal detachment, left eye |
| | rhegmatogenous retinal detachment, left eye |
| rhegmatogenous retinal detachment, left eye | |
| | rhegmatogenous retinal detachment, left eye |
| | rhegmatogenous retinal detachment, left eye |
| | inegnatogenous retinal detadiment, leit eye |
| | The grid to get hour retained detailment, left eye |
| E1325/2 26303 Other specified displates multiple with availforation displate a displate retires the | |
| E1325/2 26202 Other specified dishetes multiple with preliferative dishetic dishetic retinanthy. | |
| E1225/2 26202 Other specified dispetes mollitus with preliferative dispeties dispeties dispeties attended to | |
| E122E42 26202 Other specified dispetes multips with preliferative dispeties dispeties dispeties dispeties at the control of th | |
| E122E42 26202 Other specified dispetes multips with preliferative dispeties dispeties dispeties dispeties at the control of th | I I |
| E122542 26202 Other specified dishetes mollitus with preliferative dishetic Dreliferative dishetic retinantity. | |
| E122542 26202 Other specified dishetes mollitus with preliferative dishetic Breliferative dishetic retinantity. | |
| E1225/2 26202 Other specified dishetes multiply with preliferative dishetic Decliferative dishetic retirements. | 1 |
| E1225/2 26202 Other specified dishetes mollitus with proliferative dishetic Proliferative dishetic retinantity | |
| E1225/2 26202 Other specified dishetes mollitus with proliferative dishetic Proliferative dishetic retinantial | |
| E1225/2 26202 Other specified disheter muliture with preliferative dishetic section of the secti | 1 |
| E1225/12 26202 Other specified dishetes mollitus with preliferative dishetic Preliferative dishetic retinantial | į l |
| E1225/12 26202 Other specified dishetes mollitus with preliferative dishetic Decliferative dishetic retires the | |
| | rnegmatogenous retinai detachment, ieπ eye |
| | rhegmatogenous retinal detachment, left eye |
| rhegmatogenous retinal detachment, left eye | |
| | rhegmatogenous retinal detachment, left eye |
| | rhegmatogenous retinal detachment, left eye |
| | rhegmatogenous retinal detachment, left eye |
| | rnegmatogenous retinai detachment, ieπ eye |
| E1225/2 26202 Other specified dispetes mollitus with preliferative dispeties dispeties dispeties at the control of the control | |
| E1225/2 26202 Other specified dispetes mellitus with preliferative dispeties dispeties dispeties at the control of the control | į |
| E1225/12 26202 Other specified dishetes mallitus with preliferative dishetic Preliferative dishetic retinantial | |
| ELECTION 1 SOCIAL TOTALE SPECIAL DISTRICT MEDITAL WITH DEGINERATIVE DISTRETATIVE DI | 36202 Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy |
| rhegmatogenous retinal detachment, bilateral | retinopathy with combined traction retinal detachment and |
| E133549 36202 Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy | |
| rationalthy with combined traction ratioal datachment and | rhegmatogenous retinal detachment, bilateral |
| retinopatny with combined traction retinal detachment and | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic Proliferative diabetic retinopathy |
| | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and |
| rhegmatogenous retinal detachment, unspecified eye | rhegmatogenous retinal detachment, bilateral Other specified diabetes mellitus with proliferative diabetic retinopathy with combined traction retinal detachment and rhegmatogenous retinal detachment, unspecified eye |


## Obesity


## Appendix A Dementia risk factors


Orlistat
Sibutramine
Phentermine
Benzphetamine
Phendimetrazine
Diethylpropion

Hypertension

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| 110 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
| 110 | 4011 | Essential (primary) hypertension | Benign essential hypertension |
| 110 | 4019 | Essential (primary) hypertension | Unspecified essential hypertension |
| 1160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| l161 | 4019 | Hypertensive emergency | Unspecified essential hypertension |
| 1169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| l119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| l110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| l119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| l110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart failure |
| l110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| 1129 | 40300 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, malignant, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| l120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, malignant, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| l129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney disease | kidney disease stage I through stage IV, or unspecified |
| l120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| l129 | 40390 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, unspecified, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| I120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40401 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |

| l1311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
|---|---|---|---|
| 11311 | 40402 | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| 1132 | 40403 | failure and with stage 5 chronic kidney disease, or end | with heart failure and with chronic kidney disease stage V |
| | | - ' | · |
| l1310 | 40410 | stage renal disease Hypertensive heart and chronic kidney disease without | or end stage renal disease Hypertensive heart and chronic kidney disease, benign, |
| 11510 | 40410 | | |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| 1120 | 40411 | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I |
| 11011 | 10110 | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and with stage 5 chronic kidney disease, or end | heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| l1310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| 1130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| I1311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| 1132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| I150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| I158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| I150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| I151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| l152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| l158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| 1159 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |

onary artery disease


| 33519 |
|----------|
| 33520 |
| 33521 |
| 33522 |
| 33523 |
| 33524 |
| 33525 |
| 33526 |
| 33527 |
| 33528 |
| 33529 |
| 33530 |
| 33531 |
| 33532 |
| 33533 |
| 33534 |
| 33535 |
| 33536 |
| 33545 |
| 33572 |
| CPT |
| 92973 |
| 92982 |
| 92984 |
| 92995 |
| 92996 |
| 92920 |
| 92921 |
| 92924 |
| 92925 |
| 92937 |
| 92938 |
| 92941 |
| 92943 |
| 92944 |
| ICD10 Dx |
| 1208 |


| Insertion of non-drug-eluting coronary artery stent(s) insertion of non-drug-elut |
|---|
| Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sitent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, anondrug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, situation of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, situation of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Art |
| 02720DZ 3606 with Intraluminal Device, Open Approach stent(s) |
| Dilation of Coronary Artery, Three Arteries, self-self-self-self-self-self-self-self- |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries on Ondrug-eluting or Open Approach Dilation of Coronary Artery, Three Arteries on Ondrug-eluting or Open Approach Dilation of Coronary Artery, Three Arteries on Ondrug-eluting or Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Intraluminal Devices, Open Open Approach Dilation of Coronary Artery, Three Arteries or Open Approach Dilation of Coronary Artery, Three Arteries or Open Approach Dilation of Coronary Artery, Three Arteries or Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal Devices, Open Open Open Approach Dilation of Coronary Artery, Three Arteries or Open |
| Bifurcation, with Two Intraluminal Devices, Coronary artery Stent(s) Insertion of |
| 02720E6 3606 Open Approach Insertion of Dilation of Coronary Artery, Three Arteries with Two Intraluminal Devices, Open coronary artery stent(s) 02720EZ 3606 Approach stent(s) 02720EZ 3606 Approach stent(s) 02720EA 3606 Approach stent(s) 02720F6 3606 Open Approach stent(s) 02720F6 3606 Open Approach stent(s) 02720F2 3606 Open Approach stent(s) 02720F2 3606 Approach stent(s) 02720F2 3606 Approach stent(s) 02720F2 3606 Approach stent(s) 02720F2 3606 Approach stent(s) 02720F2 3606 Approach stent(s) 02720F3 3606 Devices, Open Approach stent(s) 02720F3 3606 Devices, Open Approach stent(s) 02720F3 3606 Device, Open Approach stent(s) 02720F3 3606 Approach stent(s) 02720F3 3606 Approach stent(s) 02720F3 3606 Approach stent(s) 02720F3 3606 Approach stent(s) 02720F3 3606 Approach stent(s) 02720F4 3606 Approach stent(s) 02720F5 Sentent Stent(s) 02720F6 Sentent Stent(s) 02720F6 Sentent Stent(s) 02720F7 Sentent Stent(s) |
| Dilation of Coronary Artery, Three Arteries with Two Insertion of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinon-drug-eluting coronary artery stent(s) |
| Dilation of Coronary Artery, Three Arteries with Two Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, selfurcation, with Three Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery artery artery artery stent(s) Dilation of Coronary Artery, Three Arteries coronary artery arte |
| with Two Intraluminal Devices, Open stent(s) Approach Insertion of On-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch on-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch on-drug-eluting coronary artery stent(s) |
| 02720EZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stent(s) 02720F6 3606 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Three Intraluminal Devices, open coronary artery stent(s) 02720FZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries with Three Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, political for non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, political for non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sinch-drug-eluting coronary artery stent(s) |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith Three Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith Three Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith Four or More Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith Four or More Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith Four or More Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith(s) Dilation of Coronary Artery, Three Arteries send-rug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith Radioactive Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries swith Radioactive Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Open coronary artery stent(s) |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Intraluminal Devices, Open Dilation of Coronary Artery, Three Arteries with Three Intraluminal Devices, Open Oz720FZ 3606 Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal Oz720G6 Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Devices, Open Oz720GZ 3606 Approach Dilation of Coronary Artery, Three Arteries, with Four or More Intraluminal Devices, Open Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal Device, Open Approach Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Ozonary artery Stent(s) |
| Bifurcation, with Three Intraluminal Devices, stent(s) Open Approach Insertion of |
| 02720F6 3606 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries ocoronary artery stent(s) 02720FZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal coronary artery stent(s) 02720G6 3606 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries onon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries onon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries onon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries onon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries onon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries onon-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Coronary artery stent(s) |
| Dilation of Coronary Artery, Three Arteries with Three Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal coronary artery stent(s) Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Insertion of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Sentence of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, coronary artery coronary artery stent(s) |
| Dilation of Coronary Artery, Three Arteries with Three Intraluminal Devices, Open 02720FZ 3606 Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal Devices, Open Dilation of Coronary Artery, Three Arteries Bifurcation of Coronary Artery, Three Arteries Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Devices, Open Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Devices, Open Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal Device, Open Approach Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open O2720TZ 3606 Approach Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open O2720TZ 3606 Approach Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open O2720TZ 3606 Dilation of Coronary Artery, Three Arteries, Sifurcation, with Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Coronary Artery Coronary Corona |
| with Three Intraluminal Devices, Open Approach Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal O2720G6 Dilation of Coronary Artery, Three Arteries Bifurcation, with Four or More Intraluminal O2720G6 Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Devices, Open O2720GZ Approach Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Devices, Open O2720GZ Bifurcation, with Radioactive Intraluminal O2720T6 Dilation of Coronary Artery, Three Arteries Bifurcation, with Radioactive Intraluminal Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open O2720TZ Approach Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open O2720TZ Bifurcation, with Intraluminal Device, Bifurcation, with Intraluminal Device, Coronary artery |
| 02720FZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery 02720G6 3606 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery 02720GZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery 02720GZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting sifurcation, with Radioactive Intraluminal coronary artery 02720TG 3606 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, poen stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal coronary artery 02720G6 3606 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting with Four or More Intraluminal Devices, Open coronary artery 02720GZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal Device, Open stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal coronary artery 02720TZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery 02720TZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting stent(s) Insertion of non-drug-eluting coronary artery 02720TZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting non-drug-eluting coronary artery Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Intraluminal Coronary artery Stent(s) Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Devices, Open O2720GZ 3606 Approach Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Devices, Open O2720GZ 3606 Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal Coronary artery O2720T6 Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open O2720TZ 3606 Approach Dilation of Coronary Artery, Three Arteries with Radioactive Intraluminal Device, Open O2720TZ 3606 Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Coronary artery O2720TZ Coronary Artery, Three Arteries, Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Coronary artery |
| Bifurcation, with Four or More Intraluminal coronary artery stent(s) Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, significant of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, significant of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, significant of non-drug-eluting coronary artery stent(s) |
| Bifurcation, with Four or More Intraluminal coronary artery stent(s) Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, sifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, significant of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, significant of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, significant of non-drug-eluting coronary artery stent(s) |
| 02720G6 3606 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) 02720GZ 3606 Approach Insertion of non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stent(s) Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery |
| Dilation of Coronary Artery, Three Arteries with Four or More Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, shifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, shifurcation, with Radioactive Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries shifurcation of stent(s) Dilation of Coronary Artery, Three Arteries shifurcation of stent(s) Dilation of Coronary Artery, Three Arteries stent(s) Dilation of Coronary Artery, Three Arteries, shifurcation of stent(s) Dilation of Coronary Artery, Three Arteries, shifurcation, with Intraluminal Device, coronary artery stenty |
| with Four or More Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting |
| with Four or More Intraluminal Devices, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting |
| 02720GZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stent(s) 02720T6 3606 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery stent(s) 02720TZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting non-drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting coronary artery stifunction, with Intraluminal Device, coronary artery |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal coronary artery 02720T6 3606 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery 02720TZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, Coronary artery 02720TZ Society Stent(s) Insertion of non-drug-eluting coronary artery |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Radioactive Intraluminal coronary artery 02720T6 3606 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery 02720TZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, Dilation of Coronary Artery, Three Arteries, Bifurcation, with Intraluminal Device, coronary artery 02720TZ September 1 |
| Bifurcation, with Radioactive Intraluminal coronary artery 3606 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting sifurcation, with Intraluminal Device, coronary artery |
| 02720T6 3606 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery 02720TZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting non-drug-eluting coronary artery Bifurcation, with Intraluminal Device, coronary artery |
| Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting Bifurcation, with Intraluminal Device, coronary artery |
| Dilation of Coronary Artery, Three Arteries non-drug-eluting with Radioactive Intraluminal Device, Open coronary artery 3606 Approach stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, non-drug-eluting Bifurcation, with Intraluminal Device, coronary artery |
| with Radioactive Intraluminal Device, Open coronary artery stent(s) 102720TZ 3606 Approach stent(s) 102720TZ Insertion of Insertion o |
| 02720TZ 3606 Approach stent(s) Dilation of Coronary Artery, Three Arteries, non-drug-eluting Bifurcation, with Intraluminal Device, coronary artery |
| Dilation of Coronary Artery, Three Arteries, non-drug-eluting Bifurcation, with Intraluminal Device, coronary artery |
| Dilation of Coronary Artery, Three Arteries, non-drug-eluting Bifurcation, with Intraluminal Device, coronary artery |
| Bifurcation, with Intraluminal Device, coronary artery |
| 02/2500 5000 Percutations Approach (Stenit's) |
| Insertion of |
| Dilation of Coronary Artery, Three Arteries non-drug-eluting with Intraluminal Device, Percutaneous coronary artery |
| 02723DZ 3606 Approach stent(s) |
| Insertion of |
| Dilation of Coronary Artery, Three Arteries, non-drug-eluting |
| Bifurcation, with Two Intraluminal Devices, coronary artery |
| 02723E6 3606 Percutaneous Approach stent(s) |
| Insertion of |
| Dilation of Coronary Artery, Three Arteries non-drug-eluting |
| with Two Intraluminal Devices, Percutaneous coronary artery |
| 02723EZ 3606 Approach stent(s) |
| Insertion of |
| Dilation of Coronary Artery, Three Arteries, non-drug-eluting |
| Bifurcation, with Three Intraluminal Devices, coronary artery |
| 02723F6 3606 Percutaneous Approach stent(s) |
| Insertion of |
| Dilation of Coronary Artery, Three Arteries non-drug-eluting |
| with Three Intraluminal Devices, coronary artery |
| 02723FZ 3606 Percutaneous Approach stent(s) |


| Dilation of Coronary Artery, One Artery, Sthraction, with Drug-eluting intraluminal Coronary artery Stentis Dilation of Coronary Artery, One Artery with Drug-eluting intraluminal bevice, Open Dilation of Coronary Artery, One Artery Dilation of Coronary Artery, One Artery Silveration, with Two Drug-eluting Dilation of Coronary Artery, One Artery Dilation of Coronary Artery, One Artery Dilation of Coronary Artery, One Artery Dilation of Coronary Artery, One Artery Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Open Dilation of Coronary Artery, One Artery Dilation | I | | | linear of |
|---|---|---|---|---|
| Bituration, with Drug-eluting Intraluminal coronary artery sterifs | | | | Insertion of |
| Dilation of Coronary Artery, One Artery with coronary artery stentigl or section of drug-eluting stentigl or section of drug-eluting coronary artery stentigl or section of drug-eluting section of drug-eluting section o | | | | |
| Dilation of Coronary Artery, One Artery with Drug-eluting intraluminal Device, Open (appearance) Dilation of Coronary Artery, One Artery (appearance) Dilation of Coronary Artery, One Artery (appearance) Dilation of Coronary Artery, One Artery (appearance) Dilation of Coronary Artery, One Artery (appearance) Dilation of Coronary Artery, One Artery with Coronary artery (appearance) Dilation of Coronary Artery, One Artery (appearance) Dilation of Coronary Artery, One Arte | | | | · · · |
| Dilation of Coronary Artery, One Artery with coronary artery stent(s) Dilation of Coronary Artery, One Artery stent(s) Dilation of Coronary Artery, One Artery stent(s) Dilation of Coronary Artery, One Artery stent(s) Dilation of Coronary Artery, One Artery with cross stent(s) Dilation of Coronary Artery, One Artery with cross stent(s) Dilation of Coronary Artery, One Artery with cross stent(s) Dilation of Coronary Artery, One Artery with free Drug-eluting stental minal Devices, Open Approach Dilation of Coronary Artery, One Artery stent(s) Dilation of Coronary Artery, One Artery with cross stent(s) Dilation of Coronary Artery, One Artery with free Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with free Drug-eluting strail minal Devices, Device, Percutaneous Approach Dilation of Coronary Artery, One Artery with free Drug-eluting strail minal Devices, Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery with free Drug-eluting strail minal Devices, Device, Drug-eluting strail minal Devices, Device, Drug-eluting strail min | 0270046 | 3607 | Device, Open Approach | `` |
| Duge duting intraluminal Device, Open (coronary artery tents) Approach (sents) Dilation of Coronary Artery, One Artery, or Coronary artery stents) Dilation of Coronary Artery, One Artery with (coronary artery) Dilation of Coronary Artery, One Artery, (coronary artery) Dilation of Coronary Artery, One Artery, (coronary artery) Dilation of Coronary Artery, One Artery, (coronary artery) Dilation of Coronary Artery, One Artery with (coronary artery) Dilation of Coronary Artery, One Artery, (coronary) Dilation of Coronary Artery, One Artery, (c | | | | Insertion of |
| Dilation of Coronary Artery, One Artery with coronary artery strents) Dilation of Coronary Artery, One Artery with Three Drug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Three Drug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Three Drug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Three Drug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Coronary artery strents) Dilation of Coronary Artery, One Artery with Coronary artery strents) Dilation of Coronary Artery, One Artery with Coronary artery strents) Dilation of Coronary Artery, One Artery with Grug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Grug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Grug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Grug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Drug-eluting intraluminal Device, One Artery, Grug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Drug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Grug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Grug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Grug-eluting coronary artery strents) Dilation of Coronary Artery, One Artery with Grug-eluting coronary artery strents) Dilation of Coronar | | | Dilation of Coronary Artery, One Artery with | drug-eluting |
| Dilation of Coronary Artery, One Artery, Bfurcation, with Two Drug-eluting Dilation of Coronary Artery, One Artery with Dilation of Coronary Artery, One Artery with Two Drug-eluting intraluminal Devices, Open Agroach Dilation of Coronary Artery, One Artery with Dilation of Coronary Artery, One Artery, Bfurcation, with Two Drug-eluting Dilation of Coronary Artery, One Artery, Bfurcation, with Drug-eluting intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting intraluminal Dilation of Coronary Artery, One Artery with Four or More Drug-eluting intraluminal Dilation of Coronary Artery, One Artery with Four or More Drug-eluting intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery with Drug-eluting intraluminal Device, Dilation of Coronary Artery, One Artery with Drug-eluting intraluminal Device, Dilation of Coronary Artery, One Artery with Drug-eluting intraluminal Device, Dilation of Coronary Artery, One Artery with Drug-eluting intraluminal Device, Dilation of Coronary Artery, One Artery, Bfurcation, with Two Drug-eluting Dilation of Coronary Artery, One Artery with Two Drug-eluting intraluminal Devices, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bfurcation, with Two Drug-eluting intraluminal Device, Percutaneous Approach Dilation of Coronary Artery, One Artery, Bfurcation, with Two D | | | Drug-eluting Intraluminal Device, Open | coronary artery |
| Dilation of Coronary Artery, One Artery 0270056 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting prosphere 0270052 3607 Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting intraluminal Devices, Open 0270052 3607 Approach Dilation of Coronary Artery, One Artery Sifurcation, with Two Drug-eluting 0270066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery Sifurcation, with Four or More Drug-eluting 0270066 3607 Open Approach Dilation of Coronary Artery, One Artery Sifurcation, with Four or More Drug-eluting 0270076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with four or More Drug-eluting intraluminal 0270072 3600 Devices, Open Approach Dilation of Coronary Artery, One Artery, Sifurcation, With Drug-eluting Intraluminal 0270072 3600 Devices, Open Approach Dilation of Coronary Artery, One Artery, Sifurcation, With Drug-eluting Intraluminal 0270074 3607 Device, Open Approach Dilation of Coronary Artery, One Artery, Sifurcation, With Drug-eluting Intraluminal 0270078 Coronary Artery, One Artery, Sifurcation, With Drug-eluting Intraluminal 0270079 Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, Open Approach Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, Open Approach Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, Open Approach Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with True Drug-eluting Intraluminal Devices, Open Approach D | 027004Z | 3607 | Approach | stent(s) |
| Sifurcation, with Two Drug-eluting coronary artery coronary | | | | Insertion of |
| 0270056 3607 Intraluminal Devices, Open Approach Insertion of drug-eluting formation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Open Approach Insertion of drug-eluting formation of Coronary Artery, One Artery, One Artery, One Artery of Grug-eluting Oz70052 3607 Approach Intraluminal Devices, Open Approach Intraluminal Devices, Open Approach Intraluminal Devices, Open Approach Intraluminal Devices, Open Approach Intraluminal Devices, Open Approach Insertion of drug-eluting Oz70062 3607 Open Approach Intraluminal Devices, Open Approach Insertion of Oz70062 Intraluminal Devices, Open Approach Intraluminal Devices, Open Approach Insertion of Oz70063 Intraluminal Devices, Open Approach Insertion of Oz70064 Intraluminal Devices, Open Approach Insertion of Oz70074 Intraluminal Devices, Open Approach Insertion of Oz70075 Intraluminal Oz70075 In | | | Dilation of Coronary Artery, One Artery, | drug-eluting |
| Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, with Insertion of drug-eluting patients with Three Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting patients with Three Drug-eluting pati | | | Bifurcation, with Two Drug-eluting | coronary artery |
| Dilation of Coronary Artery, One Artery with coronary artery stent(s) Dilation of Coronary Artery, One Artery of drug eluting or Onary artery or Onary artery or Onary artery or Onary artery or Onary artery, One Artery with or Onary Artery, One Artery with or Onary artery or Onary artery, One Artery, One Artery, One Artery, One Artery or Onary artery or Onary artery, One Artery or Onary or Onary or Onary artery or Onary artery or Onary artery or Onary or Onary or Onary artery, One Artery with Onary or Onary Onary or Onary artery or Onary artery or Onary | 0270056 | 3607 | Intraluminal Devices, Open Approach | stent(s) |
| Two Druge pluting Intraluminal Devices, Open and Coronary artery stent(s) Dilation of Coronary Artery, One Artery, druge-luting Bifurcation, with Three Druge-luting coronary artery stent(s) Dilation of Coronary Artery, One Artery with coronary artery stent(s) | | | | Insertion of |
| Two Druge pluting Intraluminal Devices, Open and Coronary artery stent(s) Dilation of Coronary Artery, One Artery, druge-luting Bifurcation, with Three Druge-luting coronary artery stent(s) Dilation of Coronary Artery, One Artery with coronary artery stent(s) | | | Dilation of Coronary Artery, One Artery with | drug-eluting |
| 027005Z 3607 Approach Insertion of drug-eluting coronary artery Bifurcation, with Three Drug-eluting coronary artery Insertion of drug-eluting coronary artery Insertion of drug-eluting coronary artery Insertion of drug-eluting coronary artery Insertion of drug-eluting Insertion of Dilation of Coronary Artery, One Artery with Insertion of Dilation of Coronary Artery, One Artery with Insertion of Dilation of Coronary Artery, One Artery with Insertion of Dilation of Coronary Artery, One Artery with Insertion of Dilation of Coronary Artery, One Artery with Insertion of Dilation of Coronary Artery, One Artery, One Artery with Insertion of Dilation of Coronary Artery, One Artery, | | | | |
| Dilation of Coronary Artery, One Artery, stent(s) 0270066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting intraluminal Devices, Open Approach stent(s) 0270062 3607 Open Approach insertion of drug-eluting coronary artery stent(s) 0270063 3607 Open Approach insertion of drug-eluting coronary artery open Approach insertion of drug-eluting eluting coronary artery open Approach insertion of drug-eluting eluting elutin | 0270057 | 3607 | | |
| Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, O27006Z 3607 Open Approach Dilation of Coronary Artery, One Artery O27006Z 3607 Open Approach Dilation of Coronary Artery, One Artery, O27006Z 3607 Open Approach Dilation of Coronary Artery, One Artery, O27006Z 3607 Open Approach Dilation of Coronary Artery, One Artery, O27007Z 3607 Open Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal O27007Z 3607 Open Approach Dilation of Coronary Artery, One Artery with Four or More Drug-eluting Intraluminal O27007Z 3607 Open Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Drug-eluting Intraluminal O27007Z 3607 Open Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Drug-eluting Intraluminal O27034G 3607 Open Approach Dilation of Coronary Artery, One Artery with Orug-eluting Intraluminal Device, O27034Z 3607 Open Approach Dilation of Coronary Artery, One Artery with Orug-eluting Intraluminal Device, O27034Z 3607 Open Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting O27034C 3607 Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting O27035Z 3607 Approach Dilation of Coronary Artery, One Artery Bifurcation, with Two Drug-eluting O27036G 3607 Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting O27036C 3607 Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting O27036C 3607 Approach Dilation of Coronary Artery, One Artery Dilatio | 0270002 | 3007 | 7.56.000. | `` |
| Bifurcation, with Three Drug-eluting coronary artery stent(s) | | | Dilation of Coronary Artery One Artery | |
| 0270066 3607 Intraluminal Devices, Open Approach Insertion of drug-eluting coronary artery, One Artery with Three Drug-eluting Intraluminal Devices, stent(s) 0270062 3607 Open Approach Insertion of drug-eluting coronary artery stent(s) 0270076 3607 Intraluminal Devices, Open Approach Insertion of drug-eluting coronary artery stent(s) 0270076 3607 Intraluminal Devices, Open Approach Intraluminal Devices, Open Approach Insertion of drug-eluting coronary artery stent(s) 0270072 3607 Devices, Open Approach Insertion of drug-eluting coronary artery stent(s) 0270072 3607 Devices, Open Approach Insertion of drug-eluting coronary artery stent(s) 0270073 3607 Devices, Open Approach Insertion of drug-eluting ocronary artery stent(s) 0270346 3607 Device, Percutaneous Approach Insertion of drug-eluting ocronary artery stent(s) 0270347 3607 Device, Percutaneous Approach Insertion of drug-eluting ocronary artery stent(s) 0270348 3607 Device, Percutaneous Approach Insertion of drug-eluting ocronary artery stent(s) 0270349 3607 Device, Percutaneous Approach Insertion of drug-eluting ocronary artery stent(s) 0270340 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270350 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270351 3607 Percutaneous Approach Insertion of drug-eluting ocronary artery stent(s) 0270352 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270360 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270361 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270362 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270362 3607 Percutaneous Approach Insertion of drug-eluting ocronary artery stent(s) 0270362 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270363 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270364 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270365 3607 Approach Insertion of drug-eluting ocronary artery stent(s) 0270367 3607 | | | | |
| Dilation of Coronary Artery, One Artery with three Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispensive drug-eluting drug-eluting intraluminal Device, percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, dispensive drug-eluting drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting intraluminal Devices, percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispensive drug-eluting coronary artery stent(s) Dilation of Co | 0270066 | 2607 | | |
| Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with four of More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent | 02/0000 | 3007 | пистанинная Бечнез, Орен Арриовин | |
| Three Drug-eluting Intraluminal Devices, stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with for or More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery with for or More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting intraluminal Device, coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting intraluminal Devices, percutaneous stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary art | | | Dilation of Caranary Artary, One Artary, with | |
| 027006Z 3607 Open Approach Insertion of drug-eluting coronary artery drug-eluting coronary artery stent(s) 0270076 3607 Intraluminal Devices, Open Approach stent(s) 0270076 3607 Intraluminal Devices, Open Approach stent(s) 0270077 3607 Devices, Open Approach stent(s) 0270078 3607 Devices, Open Approach stent(s) 0270079 3607 Devices, Open Approach stent(s) 0270070 3607 Devices, Open Approach stent(s) 0270346 3607 Device, Open Approach stent(s) 0270347 Devices, Open Approach stent(s) 0270348 3607 Device, Percutaneous Approach stent(s) 0270349 Device, Percutaneous Approach stent(s) 0270340 September S | | | | |
| Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) 10270076 3607 intraluminal Devices, Open Approach stent(s) 10270072 3607 Devices, Open Approach stent(s) 10270072 3607 Devices, Open Approach stent(s) 10270072 3607 Devices, Open Approach stent(s) 10270073 3607 Devices, Open Approach stent(s) 10270074 3607 Devices, Open Approach stent(s) 10270075 September 1 | | | | |
| Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with coronary artery stent(s) Dilation of Coronary Artery, One Artery with coronary artery stent(s) Dilation of Coronary Artery, One Artery with coronary artery stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting Drug-eluting intraluminal Device, coronary artery stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Dilation of Coronary Artery, One Artery with Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, One Artery, Dilation of Coronary Artery, One Artery with Dilation of Coronary Artery, One Artery with Dilation of Coronary Artery, One Artery with Dilation of Coronary Artery, One Artery with Dilation of Coronary Artery, One Artery with Dilation of Coronary Artery, One Artery, Dilation of Coronary Artery, One Artery Dilation of Coronary Artery, One Artery Dilation of Coronary Artery | 0270062 | 3607 | Open Approach | `` |
| Dilation of Coronary Artery, One Artery with foruge-luting coronary artery stent(s) Dilation of Coronary Artery, One Artery with four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, One Artery with foruge-luting coronary artery stent(s) Devices, Open Approach Dilation of Coronary Artery, One Artery, drug-eluting Interaluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, insertion of stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, percutaneous stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting intraluminal Devices, percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery with prove or More Drug-eluting intraluminal Devices, coronary artery stent(s) | | | | |
| Oz70076 3607 Intraluminal Devices, Open Approach Insertion of Insertion of | | | | |
| Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, one Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with coronary artery stent(s) Dilation of Coronary Artery, One Artery with Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispetition of drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispetition of drug-eluting drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispetition of drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispetition of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting intraluminal Devices, Percutaneous stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispetition of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispetition of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispetition of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, dispetition of drug-eluting coronary artery stent(s) | | | | coronary artery |
| Dilation of Coronary Artery, One Artery with four or More Drug-eluting Intraluminal coronary artery stent(s) Devices, Open Approach stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting coronary artery stent(s) Device, Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with Drug-eluting intraluminal Device, coronary artery stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting intraluminal Devices, Percutaneous stent(s) Dilation of Coronary Artery, One Artery with drug-eluting intraluminal Devices, Devices, Devices, Devices, Stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, De | 0270076 | 3607 | Intraluminal Devices, Open Approach | stent(s) |
| Four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting drug-eluting coronary artery Dilation of Coronary Artery, One Artery, drug-eluting coronary artery Dilation of Coronary Artery, One Artery with drug-eluting drug-eluting coronary artery Dilation of Coronary Artery, One Artery with drug-eluting coronary artery Dilation of Coronary Artery, One Artery with drug-eluting drug-eluting coronary artery Dilation of Coronary Artery, One Artery, linsertion of drug-eluting intraluminal Device, Percutaneous Approach Dilation of Coronary Artery, One Artery, linsertion of drug-eluting intraluminal Devices, Percutaneous coronary artery Dilation of Coronary Artery, One Artery with drug-eluting intraluminal Devices, percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, linsertion of drug-eluting coronary artery Dilation of Coronary Artery, One Artery, linsertion of drug-eluting intraluminal Devices, percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery, linsertion of drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery stent(s) Dilation of Coronary Artery, One Artery, linsertion of drug-eluting intraluminal Devices, percutaneous coronary artery stent(s) | | | | Insertion of |
| Devices, Open Approach Stent(s) Insertion of Insertion of drug-eluting Gronary Artery, One Artery, drug-eluting Gronary artery Oz70346 3607 Device, Percutaneous Approach Stent(s) Insertion of Insertion o | | | Dilation of Coronary Artery, One Artery with | drug-eluting |
| Dilation of Coronary Artery, One Artery, Bifurcation, with Drug-eluting Intraluminal O270346 3607 Device, Percutaneous Approach Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, O270342 3607 Device, Percutaneous Approach Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, O270342 O270343 Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous O270356 O270356 Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, O270357 Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, O270358 Dilation of Coronary Artery, One Artery, Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Dilation of Coronary Artery, One Artery, Dilation of Coronary Artery, Dilation of Corona | | | Four or More Drug-eluting Intraluminal | coronary artery |
| Dilation of Coronary Artery, One Artery, Bifurcation, with Drug-eluting Intraluminal Dilation of Coronary Artery, One Artery with Stent(s) Dilation of Coronary Artery, One Artery with Drug-eluting Oronary artery Dilation of Coronary Artery, One Artery with Drug-eluting Oronary artery Dilation of Coronary Artery, One Artery, Insertion of Oronary artery Bifurcation, with Two Drug-eluting Intraluminal Devices, Oronary artery Dilation of Coronary Artery, One Artery, Insertion of Oronary artery Dilation of Coronary Artery, One Artery with Orug-eluting Intraluminal Devices, Percutaneous Oronary artery Dilation of Coronary Artery, One Artery with Orug-eluting Intraluminal Devices, Oronary artery Dilation of Coronary Artery, One Artery with Orug-eluting Oronary artery Dilation of Coronary Artery, One Artery, Insertion of Orug-eluting Intraluminal Devices, Oronary artery Dilation of Coronary Artery, One Artery, Insertion of Orug-eluting Intraluminal Devices, Percutaneous Oronary artery Dilation of Coronary Artery, One Artery with Orug-eluting Oronary artery Dilation of Coronary Artery, One Artery with Orug-eluting Oronary artery Dilation of Coronary Artery, One Artery with Orug-eluting Oronary artery Dilation of Coronary Artery, One Artery with Orug-eluting Oronary artery Dilation of Coronary Artery, One Artery with Orug-eluting Oronary artery Dilation of Coronary Artery, One Artery, Insertion of Orug-eluting Oronary Artery Dilation of Coronary Artery, One Artery, Insertion of Orug-eluting Or | 027007Z | 3607 | Devices, Open Approach | stent(s) |
| Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting oronary artery 27034Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting drug-eluting oronary artery 270356 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting (Intraluminal Devices, Percutaneous oronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting (Insertion of Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, One Artery with drug-eluting (Insertion of Dilation of Coronary Artery, One Artery, Insertion of drug-eluting (Insertion of Dilation of Coronary Artery, One Artery, Insertion of Dilation of Coronary Artery, One Artery, Insertion of Dilation of Coronary Artery, One Artery, Insertion of Dilation of Coronary Artery, One Artery with Three Drug-eluting (Insertion of Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting drug-eluting (Insertion of Bifurcation, with Four or More Drug-eluting (Insertion of | | | | Insertion of |
| 0270346 3607 Device, Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, coronary artery stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting Intraluminal Device, Insertion of drug-eluting Intraluminal Devices, Percutaneous Insertion of drug-eluting Intraluminal Devices, Percutaneous Insertion of drug-eluting Intraluminal Devices, Percutaneous Insertion of drug-eluting Insertion of Insertion Insertion of Insertion of Insertion of Insertion of | | | Dilation of Coronary Artery, One Artery, | drug-eluting |
| Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, coronary artery stent(s) 27034Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) 270356 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting intraluminal Devices, stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, One Artery with Approach stent(s) Dilation of Coronary Artery, One Artery with Approach stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, sercutaneous coronary artery stent(s) | | | Bifurcation, with Drug-eluting Intraluminal | coronary artery |
| Dilation of Coronary Artery, One Artery with Drug-eluting Intraluminal Device, coronary artery stent(s) Dilation of Coronary Artery, One Artery, Insertion of Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting Intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, One Artery, Insertion of Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, Percutaneous stent(s) Dilation of Coronary Artery, One Artery with Grug-eluting Coronary artery stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Insertion of Grug-eluting Intraluminal Devices, Percutaneous coronary artery stent(s) | 0270346 | 3607 | Device, Percutaneous Approach | stent(s) |
| Drug-eluting Intraluminal Device, coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, one Artery, insertion of drug-eluting insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting insertion of drug-eluting coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) | | | | Insertion of |
| Drug-eluting Intraluminal Device, coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, drug-eluting drug-eluting coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, one Artery, insertion of drug-eluting insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting insertion of drug-eluting coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, One Artery, insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery stent(s) | | | Dilation of Coronary Artery, One Artery with | drug-eluting |
| 027034Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting drug-eluting (oronary artery) 0270356 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, Percutaneous (oronary artery) Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, (oronary artery) 027035Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting Intraluminal Devices, Percutaneous (oronary artery) 0270366 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting Insertion of drug-eluting (oronary artery) Dilation of Coronary Artery, One Artery with Insertion of drug-eluting (oronary artery) Dilation of Coronary Artery, One Artery with Insertion of drug-eluting (oronary artery) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting (oronary artery) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting (oronary artery) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting (oronary artery) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting (oronary artery) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting (oronary artery) | | | 1 | |
| Dilation of Coronary Artery, One Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous 3607 Approach Dilation of Coronary Artery, One Artery with Two Drug-eluting Insertion of Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, O27035Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous O27036G 3607 Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, O27036Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, O27036Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, O27036Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Coronary artery Insertion of drug-eluting Insertion of drug-eluting coronary artery Insertion of drug-eluting coronary artery | 027034Z | 3607 | | |
| Bifurcation, with Two Drug-eluting drug-eluting coronary artery 0270356 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 7 Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 8 Dilation of Coronary Artery, One Artery, coronary artery 9 Dilation of Coronary Artery, One Artery, coronary artery 9 Dilation of Coronary Artery, One Artery, coronary artery 9 Dilation of Coronary Artery, One Artery, coronary artery 9 Dilation of Coronary Artery, One Artery, coronary artery 9 Dilation of Coronary Artery, One Artery with coronary artery 9 Dilation of Coronary Artery, One Artery with coronary artery 9 Dilation of Coronary Artery, One Artery with coronary artery 9 Dilation of Coronary Artery, One Artery, coronary artery 1 Dilation of Coronary Artery, One Artery, coronary artery 1 Dilation of Coronary Artery, One Artery, coronary artery 1 Dilation of Coronary Artery, One Artery, coronary artery 1 Dilation of Coronary Artery, One Artery, coronary artery 1 Dilation of Coronary Artery, coronary artery 1 Dilation of Coronary Artery, one Artery, coronary artery 1 Dilation of Coronary Artery, one Artery, coronary artery 1 Dilation of Coronary Artery, one Artery, coronary artery | | | | i |
| Intraluminal Devices, Percutaneous coronary artery 3607 Approach stent(s) Insertion of drug-eluting Two Drug-eluting Intraluminal Devices, coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting intraluminal Devices, coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting insertion of drug-eluting coronary artery 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery | | | | |
| 0270356 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, coronary artery 027035Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting drug-eluting intraluminal Devices, Percutaneous coronary artery 0270366 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with Three Drug-eluting drug-eluting insertion of drug-eluting insertion of drug-eluting coronary artery 0270366 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting coronary artery 027036Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting insertion of drug-eluting insertion of drug-eluting coronary artery Dilation of Coronary Artery, One Artery, Insertion of drug-eluting insertion of drug-eluting coronary artery Dilation of Coronary Artery, One Artery, Insertion of drug-eluting intraluminal Devices, Percutaneous coronary artery | | | | |
| Dilation of Coronary Artery, One Artery with drug-eluting Two Drug-eluting Intraluminal Devices, coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting Intraluminal Devices, Percutaneous coronary artery 0270366 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting Intraluminal Devices, Percutaneous coronary artery Insertion of drug-eluting Intraluminal Devices, Percutaneous coronary artery | 0270356 | 3607 | • | |
| Dilation of Coronary Artery, One Artery with Two Drug-eluting Intraluminal Devices, 27035Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous O270366 3607 Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, O27036Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, O27036Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous O27036Z Gruph Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous O27036Z Gruph Percutaneous O27036 | 02/0330 | 3007 | Proposition | |
| Two Drug-eluting Intraluminal Devices, coronary artery 27035Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting drug-eluting coronary artery Dilation of Coronary Artery, One Artery with drug-eluting Insertion of Dilation of Coronary Artery, One Artery with drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery Dilation of Coronary Artery, One Artery with drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery Dilation of Coronary Artery, One Artery, Insertion of drug-eluting Intraluminal Devices, Percutaneous Coronary artery Dilation of Coronary Artery, One Artery, Insertion of drug-eluting Intraluminal Devices, Percutaneous coronary artery | | | Dilation of Coronary Artery, One Artery with | |
| 027035Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Insertion of drug-eluting drug-eluting coronary artery 0270366 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery 027036Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, stent(s) Dilation of Coronary Artery, One Artery, coronary artery Stent(s) Dilation of Coronary Artery, One Artery, coronary artery Stent(s) Dilation of Coronary Artery, One Artery, stent(s) Dilation of Coronary Artery, One Artery, stent(s) Dilation of Coronary Artery, One Artery, stent(s) Dilation of Coronary Artery, One Artery, stent(s) Dilation of Coronary Artery, One Artery, stent(s) Dilation of Coronary Artery, one Artery, stent(s) | | | | |
| Dilation of Coronary Artery, One Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous O270366 3607 Approach Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, O27036Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery O27036Z Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Dilation of Coronary Artery, One Artery with Order-One Artery | 0270257 | 2607 | | |
| Bifurcation, with Three Drug-eluting drug-eluting coronary artery 0270366 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery 027036Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, one A | 02/0352 | 3607 | | , , |
| Intraluminal Devices, Percutaneous coronary artery 0270366 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery 027036Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous coronary artery | | | | |
| 0270366 3607 Approach stent(s) Dilation of Coronary Artery, One Artery with drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery 027036Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous coronary artery | | | | |
| Insertion of Dilation of Coronary Artery, One Artery with Three Drug-eluting Intraluminal Devices, 027036Z 3607 Percutaneous Approach Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Insertion of drug-eluting drug-eluting coronary artery | | | • | |
| Dilation of Coronary Artery, One Artery with drug-eluting Three Drug-eluting Intraluminal Devices, coronary artery 27036Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous coronary artery | 0270366 | 3607 | Approach | `` |
| Three Drug-eluting Intraluminal Devices, coronary artery 027036Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous coronary artery | | | | |
| 027036Z 3607 Percutaneous Approach stent(s) Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting drug-eluting Intraluminal Devices, Percutaneous coronary artery | | | Dilation of Coronary Artery, One Artery with | drug-eluting |
| Dilation of Coronary Artery, One Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Insertion of drug-eluting coronary artery | | | Three Drug-eluting Intraluminal Devices, | coronary artery |
| Bifurcation, with Four or More Drug-eluting drug-eluting Intraluminal Devices, Percutaneous coronary artery | 027036Z | 3607 | Percutaneous Approach | stent(s) |
| Intraluminal Devices, Percutaneous coronary artery | | | Dilation of Coronary Artery, One Artery, | Insertion of |
| Intraluminal Devices, Percutaneous coronary artery | | | Bifurcation, with Four or More Drug-eluting | drug-eluting |
| 0270376 3607 Approach stent(s) | 0270376 | 3607 | | |


| Dilation of Coronary Artery, Two Arteries with cronary artery stent(s) Dilation of Coronary Artery, Two Arteries, coronary artery stent(s) Dilation of Coronary Artery, Two Arteries, direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of four or More Drug eluting intraluminal direction of direction of direction of direction of direction of direction of direction of Dilation of Coronary Artery, Three Arteries, direction of Dilation of Coronary Artery, Three Arteries, direction of direction of direction of Dilation of Coronary Artery, Three Arteries direction of | luccution of | | 1 | |
|---|---|---|---|---|
| Three Drug-eluting Intraluminal Devices, coronary artery | Insertion of | Dilation of Caranagu Artagu Two Artarias with | | |
| Dilation of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries, and Forestina of Grown of Coronary Artery, Two Arteries with a forum of Grown of Grown of Coronary Artery, Two Arteries with forum of Grown of More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal of Grown or More Drug-eluting Intraluminal or Grown or Approach stent(s) Dilation of Coronary Artery, Three Arteries, and Grown or G | = = | · | | |
| Dilation of Coronary Artery, Two Arteries, dinsertion of Bifurcation, with Four or More Drug-eluting drug-eluting drug-eluting coronary artery stent(s) 3607 Endoscopic Approach stent(s) Dilation of Coronary Artery, Two Arteries with Insertion of Grug-eluting Devices, Percutaneous Endoscopic coronary artery stent(s) 0271472 3607 Approach Significant of Coronary Artery, Two Arteries with Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) 0272046 3607 Device, Open Approach stent(s) 0272047 3607 Approach Significant of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) 0272048 3607 Approach Significant of Coronary Artery, Three Arteries drug-eluting Sifurcation, with Two Drug-eluting Coronary artery stent(s) 0272049 Significant of Coronary Artery, Three Arteries, drug-eluting Sifurcation, with Two Drug-eluting Coronary artery Stent(s) 0272050 Significant of Coronary Artery, Three Arteries drug-eluting Sifurcation, with Two Drug-eluting Coronary artery Stent(s) 0272051 Significant of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach Stent(s) 0272052 3607 Open Approach Significant of Coronary Artery, Three Arteries Sifurcation, with Twee Drug-eluting Coronary artery Stent(s) 0272066 Significant of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) 0272067 Significant Signific | | , | 2607 | 0274467 |
| Bifurcation, with Four or More Drug-eluting coronary artery stent(s) 0271476 3607 Endoscopic Approach stent(s) Dilation of Coronary Artery, Two Arteries with four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) 0271472 3607 Approach stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting moronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Fo | ` ' | | 3607 | 02/1462 |
| Intraluminal Devices, Percutaneous coronary artery stent(s) Dilation of Coronary Artery, Two Arteries with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) | | · | | |
| Dilation of Coronary Artery, Three Arteries with Insertion of Grug-eluting Intraluminal Devices, Open Approach | 0 0 | , | | |
| Dilation of Coronary Artery, Two Arteries with Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary arte | | - | 2607 | 0274476 |
| Four or More Drug-eluting Intraluminal Devices, Percutaneous Endoscopic coronary artery stent(s) Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting mornary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) | | | 3607 | 02/14/6 |
| Devices, Percutaneous Endoscopic coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, direction of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, direction of drug-eluting coronary artery stent(s) Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | | · | | |
| 027147Z 3607 Approach Stent(s) Insertion of drug-eluting coronary artery stent(s) O272046 3607 Device, Open Approach O272046 O272047 O272047 O272047 O272048 O | ŭ ŭ | | | |
| Dilation of Coronary Artery, Three Arteries, setults and setulting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, with Drug-eluting Intraluminal pevice, Open Approach Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, setults insertion of drug-eluting coronary artery stent(s) | | - | 2607 | 0274 477 |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Device, Open Approach Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, T | ` ' | Approacn | 3607 | 02/14/2 |
| Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, or | | Dilation of Common Adam Thomas Adams | | |
| 0272046 3607 Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting linsertion of drug-eluting with Two Drug-eluting linsertion of drug-eluting with Two Drug-eluting linsertion of drug-eluting sention of Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting linsertion of drug-eluting with Three Drug-eluting linsertion of drug-eluting linsertion of drug-eluting with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries, and proach stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting linsertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting linsertion of drug-eluting coronary artery stent(s) | = = | · | | |
| Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | | | | |
| Dilation of Coronary Artery, Three Arteries with Drug-eluting Intraluminal Device, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting gradient stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, oronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) | ` ' | Device, Open Approach | 3607 | 0272046 |
| with Drug-eluting Intraluminal Device, Open coronary artery stent(s) Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) 0272052 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting sifurcation, with Four or More Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) | | | | |
| 0272042 3607 Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting 0272056 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, with Two Drug-eluting Intraluminal Devices, oronary artery 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 027206B 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, with Three Drug-eluting Coronary artery 027206C 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Coronary artery stent(s) Insertion of drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Open Approach Dilation of Coronary Artery Open | = = | | | |
| Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, coronary artery 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 10272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 027207G 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 1 Insertion of drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 1 Insertion of drug-eluting coronary artery 2 Stent(s) Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery 2 Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | ' ' | | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Two Drug-eluting 0272056 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, 027205Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 0272066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, 027206Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, 027206Z 3607 Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting coronary artery stent(s) Insertion of drug-eluting with Four or More Drug-eluting Intraluminal coronary artery stent(s) Insertion of Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery | | Approach | 3607 | 027204Z |
| Bifurcation, with Two Drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries with Two Drug-eluting loronary Artery, Three Arteries with Two Drug-eluting loronary Artery, Three Arteries, and Dilation of Coronary Artery, Three Arteries and Dilation of Coronary Artery, Three Arteries and Dilation of Coronary Artery, Three Arteries and Dilation of Coronary Artery, Three Arteries, and Dilation of Coronary Artery, Three Arteries and Dilation of Coronary Artery, Three Arteries, and Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery coronary artery stent(s) | | | | |
| 0272056 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, coronary artery stent(s) O27205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, shifurcation, with Three Drug-eluting coronary artery stent(s) O272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) O27206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Approach stent(s) Dilation of Coronary Approach stent(s) Dilation of Coronary Approach stent(s) Dilation of Coronary Approach stent(s) Insertion of drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Two Drug-eluting Intraluminal Devices, ocronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, ocronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting drug-eluting coronary artery 3607 Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Devices, Open Approach stent(s) 3607 Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | | | | |
| Dilation of Coronary Artery, Three Arteries with Two Drug-eluting Intraluminal Devices, stent(s) Open Approach Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting coronary artery stent(s) Oz72066 3607 Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Insertion of Dilation of Coronary Artery, Three Arteries, drug-eluting Gronary Artery, Three Arteries, Dilation of Coronary Artery, Three Arteries, drug-eluting Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries Gronary Artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Sifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Stent(s) Insertion of Gronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Gronary Artery Gronary Artery Stent(s) Insertion Of Gronary Artery Stent Stent(s) Insertion Of Gronary Artery Stent | ` ' | Intraluminal Devices, Open Approach | 3607 | 0272056 |
| with Two Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, With Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Sifurcation, with Four or More Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Coronary artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Coronary artery Stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery Stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery | | | | |
| 027205Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery with Four or More Drug-eluting Intraluminal coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Insertion of drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery | | · | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 0272066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Dilation of Coronary Artery, Three Arteries O272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal O27207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery O27207Z O27 | , coronary artery | with Two Drug-eluting Intraluminal Devices, | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Three Drug-eluting 0272066 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting O272076 3607 Dilation of Coronary Artery, Three Arteries Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting O272072 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Coronary artery Stent(s) Insertion of drug-eluting coronary artery stent(s) Insertion of drug-eluting Coronary artery Stent(s) Insertion of drug-eluting Coronary Artery Stent(s) Insertion of drug-eluting Coronary artery Stent(s) Insertion of drug-eluting Coronary artery O272072 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery | stent(s) | Open Approach | 3607 | 027205Z |
| Bifurcation, with Three Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, sifurcation, with Four or More Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 3607 Devices, Open Approach stent(s) | Insertion of | | | |
| 0272066 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery 0272072 3607 Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 0272072 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, stent(s) Dilation of Coronary Artery, Three Arteries, grid drug-eluting drug-eluting coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, grid drug-eluting coronary artery 027207Z Grid drug-eluting drug-eluting coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries, | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) O27206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Bifurcation, with Four or More Drug-eluting coronary artery stent(s) O272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) O27207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting stent(s) Bifurcation, with Drug-eluting Intraluminal coronary artery | coronary artery | Bifurcation, with Three Drug-eluting | | |
| Dilation of Coronary Artery, Three Arteries with Three Drug-eluting Intraluminal Devices, coronary artery 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting coronary artery Bifurcation, with Four or More Drug-eluting coronary artery 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, green of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Insertion of drug-eluting Dilation of Coronary Artery, Three Arteries, green artery Bifurcation, with Drug-eluting Intraluminal coronary artery | | Intraluminal Devices, Open Approach | 3607 | 0272066 |
| with Three Drug-eluting Intraluminal Devices, coronary artery stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting | Insertion of | | | |
| 027206Z 3607 Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting coronary artery stent(s) Insertion of drug-eluting coronary artery stent(s) Insertion of drug-eluting coronary artery stent(s) Insertion of drug-eluting insertion of drug-eluting coronary artery coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting Coronary artery O272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal O27207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery O27207Z Graph Grap | es, coronary artery | with Three Drug-eluting Intraluminal Devices, | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Four or More Drug-eluting 0272076 3607 Intraluminal Devices, Open Approach Dilation of Coronary Artery, Three Arteries with Four or More Drug-eluting Intraluminal 027207Z 3607 Devices, Open Approach Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary Artery Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal Coronary artery drug-eluting drug-eluting coronary artery | stent(s) | Open Approach | 3607 | 027206Z |
| Bifurcation, with Four or More Drug-eluting coronary artery 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery Insertion of drug-eluting coronary artery | Insertion of | | | |
| 0272076 3607 Intraluminal Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery Coronary artery | drug-eluting | Dilation of Coronary Artery, Three Arteries, | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery | coronary artery | Bifurcation, with Four or More Drug-eluting | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting with Four or More Drug-eluting Intraluminal coronary artery Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | stent(s) | Intraluminal Devices, Open Approach | 3607 | 0272076 |
| with Four or More Drug-eluting Intraluminal coronary artery 3607 Devices, Open Approach stent(s) Insertion of Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | Insertion of | | | |
| 027207Z 3607 Devices, Open Approach stent(s) Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | 0 0 | | | |
| Dilation of Coronary Artery, Three Arteries, drug-eluting Bifurcation, with Drug-eluting Intraluminal coronary artery | l coronary artery | with Four or More Drug-eluting Intraluminal | | |
| Dilation of Coronary Artery, Three Arteries, Bifurcation, with Drug-eluting Intraluminal coronary artery | | Devices, Open Approach | 3607 | 027207Z |
| Bifurcation, with Drug-eluting Intraluminal coronary artery | Insertion of | | | |
| | drug-eluting | | | |
| 0272346 3607 Device, Percutaneous Approach | coronary artery | Bifurcation, with Drug-eluting Intraluminal | | |
| Jeney | stent(s) | Device, Percutaneous Approach | 3607 | 0272346 |
| Insertion of | Insertion of | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| with Drug-eluting Intraluminal Device, coronary artery | coronary artery | with Drug-eluting Intraluminal Device, | | |
| 027234Z 3607 Percutaneous Approach stent(s) | stent(s) | Percutaneous Approach | 3607 | 027234Z |
| Dilation of Coronary Artery, Three Arteries, Insertion of | Insertion of | Dilation of Coronary Artery, Three Arteries, | | |
| Bifurcation, with Two Drug-eluting drug-eluting | drug-eluting | Bifurcation, with Two Drug-eluting | | |
| Intraluminal Devices, Percutaneous coronary artery | coronary artery | Intraluminal Devices, Percutaneous | | |
| 0272356 3607 Approach stent(s) | stent(s) | Approach | 3607 | 0272356 |
| Insertion of | Insertion of | | | |
| Dilation of Coronary Artery, Three Arteries drug-eluting | drug-eluting | Dilation of Coronary Artery, Three Arteries | | |
| with Two Drug-eluting Intraluminal Devices, coronary artery | | | | |
| 027235Z 3607 Percutaneous Approach stent(s) | | | 3607 | 027235Z |


| | | Dilation of Coronary Artery, Four or More | Insertion of |
|---|---|---|---|
| | | Arteries, Bifurcation, with Two Drug-eluting | drug-eluting |
| | | Intraluminal Devices, Percutaneous | coronary artery |
| 0273456 | 3607 | Endoscopic Approach | stent(s) |
| 0275430 | 3007 | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Two Drug-eluting Intraluminal | drug-eluting |
| | | Devices, Percutaneous Endoscopic | coronary artery |
| 027345Z | 3607 | Approach | stent(s) |
| 0273432 | 3007 | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries, Bifurcation, with Three Drug-eluting | drug-eluting |
| | | Intraluminal Devices, Percutaneous | coronary artery |
| 0273466 | 3607 | Endoscopic Approach | stent(s) |
| 0275400 | 3007 | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Three Drug-eluting Intraluminal | drug-eluting |
| | | Devices, Percutaneous Endoscopic | coronary artery |
| 027346Z | 3607 | Approach | stent(s) |
| 0275402 | 3007 | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries, Bifurcation, with Four or More | drug-eluting |
| | | Drug-eluting Intraluminal Devices, | coronary artery |
| 0273476 | 3607 | Percutaneous Endoscopic Approach | stent(s) |
| 0275470 | 3007 | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Four or More Drug-eluting | drug-eluting |
| | | Intraluminal Devices, Percutaneous | coronary artery |
| 027347Z | 3607 | Endoscopic Approach | |
| 02/34/2 | 3007 | Endoscopic Appi dacii | stent(s) Insertion of |
| | | | drug-eluting |
| NaDCC | 2607 | | coronary artery |
| NoPCS | 3607 | | stent(s) |
| СРТ | | | |
| 92980 | | | |
| 92980<br>92981 | | | |
| 92981 | | | |
| 92981<br>92928 | | | |
| 92981 | | | |
| 92981<br>92928 | | | |
| 92981<br>92928<br>92929 | | | |
| 92981<br>92928<br>92929<br>92933<br>92934 | ICD9 Dx | Long DesiCD10 | Long DesiCD9 |
| 92981<br>92928<br>92929<br>92933 | ICD9 Dx | LongDesICD10 | LongDesICD9 Postmyocardial |
| 92981<br>92928<br>92929<br>92933<br>92934 | ICD9 Dx<br>4110 | | Postmyocardial |
| 92981<br>92928<br>92929<br>92933<br>92934<br>ICD10 Dx | | LongDesICD10 Dressler's syndrome | Postmyocardial infarction syndrome |
| 92981<br>92928<br>92929<br>92933<br>92934<br>ICD10 Dx | 4110 | Dressler's syndrome | Postmyocardial infarction syndrome Intermediate |
| 92981<br>92928<br>92929<br>92933<br>92934<br>ICD10 Dx | | Dressler's syndrome Unstable angina | Postmyocardial infarction syndrome |
| 92981<br>92928<br>92929<br>92933<br>92934<br>ICD10 Dx | 4110 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of | Postmyocardial infarction syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 | 4110 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of native coronary artery with | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate |
| 92981<br>92928<br>92929<br>92933<br>92934<br>ICD10 Dx | 4110 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 | 4110 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 | 4110<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 | 4110 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 | 4110<br>4111<br>4111 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 | 4110<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 I25710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 I25710 | 4110<br>4111<br>4111<br>4111<br>4111 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 I25710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx I241 I200 I25710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of native coronary | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome |

## Appendix A Dementia risk factors


## Depression


Anxiety


Bipolar disorder


Schizophrenia


# Appendix A Dementia risk factors


#### **Smoking**


CPT codes
99406
99407
G0436
G0437
G9016
S9453
S4995
G9276
G9458
1034F
4001F
4004F

OR dispensing of: At least one nicotine or varenicline prescription

#### Mammography


Colonoscopy


Appendix A Lifestyle factors and markers for healthy behavior

| 45380 |
|-------|
| 45381 |
| 45382 |
| 45383 |
| 45384 |
| 45385 |
| 45386 |
| 45387 |
| 45388 |
| 45389 |
| 45390 |
| 45391 |
| 45392 |
| HCPCS |
| G0105 |
| G0121 |

#### Fecal occult blood test


#### Influenza vaccination


#### Pneumococcal vaccination


## Appendix A Lifestyle factors and markers for healthy behavior

| 90670 |
|-------|
| 90732 |

### Herpes zoster vaccination


#### BMD test

| CPT |
|-------|
| 76070 |
| 76075 |
| 76076 |
| 76977 |
| 77080 |
| 77085 |

### Appendix A Healthcare utilization measures

#### Number of generic medications

NDC generic drug name has any value

If multiple events on a single day, the value is measured as combined values.

#### Number of ED visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99281 | 99282 | 99283 | 99284 | 99285 | 99288 |

#### Number of outpatient visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99450 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99455 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99456 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99499 |
| 99213 | 99271 | 99357 | 99391 | 99402 | |

#### Number of hospitalizations

The occurrence of MEDPAR with the following attributes:

Inpatient admission type code exists

The occurrence of carrier claims with the following attributes:

20 = Non swing bed SNF claim

30 = Swing bed SNF claim

50 = Hospice claim

60 = Inpatient claim

61 = Inpatient 'full-encounter' claim

#### Number of PCP visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

01 = General practice

08 = Family practice

11 = Internal medicine

84 = Preventive medicine (eff 5/92)

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99429 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99450 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99455 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99456 |
| 99213 | 99271 | 99357 | 99391 | 99402 | 99499 |

#### Number of CRP tests

| CPT | |
|-------|-------|
| 86140 | 86141 |

#### Number of serum creatinine tests


## Appendix A Frailty markers

#### Frailty Score for Claims Data

Kim DH. Schneeweiss S. Glynn RJ. Lipsitz LA. Rockwood K. Avorn J. Measuring frailty in Medicare data: Development and validation of a claims-based frailty index. Journals of Gerontology: Medical Sciences 2018;73(7):980-87.

Codes used for each component of the frailty score

| Condition | ICD9 Dx | ICD10 Dx | Coefficient |
|---|---|---|---|
| Intercept | | | 0.10288 |
| ntestinal infectious diseases | 001-009 | A00-A09 (exclude A02.1) | 0.00582 |
| Other and unspecified effects of external causes | 990-995 | A02.1, A22.7, A26.7, A32.7, A40, A41, A42.7, A45.8, B37.7, R65, T33, T34, T36-T50, T66-T78, T88 | 0.0085 |
| Other bacterial diseases | 030-041 | A30-A39; A42-A49 (exclude A32.7,A42.7,A45) | 0.01188 |
| Mycoses | 110-118 | B35-B49 (exclude B37.7) | 0.00831 |
| Malignant neoplasm of other and unspecified sites | 190-199 | C69-C80 | 0.00797 |
| Organic psychotic conditions | 290-294 | D01, D03, F02, F04, F05, F06, F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.991, F19.994, F19.950, F19.951, F19.96, F19.97, F19.99 | 0.04745 |
| Benign neoplasms | 210-229 | D10-D36 | -0.00513 |
| Neoplasms of uncertain behavior | 235-238 | D37-D48 | -0.00061 |
| Other and unspecified anemias | 285 | D62, D64 | 0.0085 |
| Purpura and other hemorrhagic conditions | 287 | D69 | -0.00804 |
| Diseases of white blood cells | 288 | D70, D71, D72, D76 | -0.0068 |
| Other metabolic and immunity disorders | 270-279 | D80-D84, D89, E65-E68, E70-E88, M10 (exclude E75.02, E75.19, E75.23, E75.25, E75.29, E75.4) | -0.00564 |
| Disorders of thyroid gland | 240-246 | E00-E07 | 0.00439 |
| Diseases of other endocrine glands | 250-259 | E08-E16,E20-E35 | 0.01078 |
| Hereditary and degenerative diseases of the central nervous system | 330-337 | E75.02, E75.19, E75.23, E75.25, E75.29, E75.4, F84.2, G10, G11, G12, G20, G21.0, G23, G24, G25, G30.9, G31, G80.3, G90, G91, G93.7, G93.89, G93.9, G94, G95, G99.2 | 0.01078 |

| Neurotic Disorders, Personality<br>Disorders, And Other Nonpsychotic<br>Mental Disorders | 300-316 | F07, F09, F32.9, F40-F44, F48, F54, F60, F64-F66, F68, F10-F19, F45.8, F45.9, F50, F51, F63.3, F80-F82, F88-F91, F93-F95, F98, R45.1, R48.0 (exclude F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F14.982, F14.988, F15.122, F15.159, F15.180, F15.181, F15.182, F15.188, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.959, F18.980, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.921, F19.982, F19.939, F19.94, F19.950, F19.951, F19.96, | 0.01353 |
|---|---|---|---|
| Other psychoses | 295-299 | F20, F22-F25, F28-F34, F39, F44.89, F84 (exclude F84.2, F32.9) | 0.02112 |
| Other disorders of the central nervous system | 340-349 | G35, G37, G40, G43, G47.4, G80-G83, G92, G93.0-G93.2, G93.4-G93.6, G96-G97, G98.8 (exclusion G80.3 ) | 0.04031 |
| Disorders of the peripheral nervous system | 350-359 | G60-G65 | 0.00338 |
| Disorders of the eye and adnexa | 360-379 | H00-H59 (exclude H54.7) | -0.00061 |
| Hypertensive disease | 401-405 | 110-116 | 0.0174 |
| Ischemic heart disease | 410-414 | 120-125 | 0.0192 |
| Other forms of heart disease | 420-429 | 130-152 | 0.01989 |
| Cerebrovascular disease | 430-438 | 160-169 | -0.00046 |
| Diseases of arteries, arterioles, and capillaries | 440-448 | 170-179 | 0.00106 |
| Diseases of veins and lymphatics, and other diseases of circulatory system | 451-459 | 180-189;195-199 | 0.01234 |
| Pneumonia and influenza | 480-487 | J09-J18 | 0.01185 |
| Other diseases of the upper respiratory tract | 470-478 | 130-139 | -0.0052 |
| Chronic obstructive pulmonary disease and allied conditions | 490-496 | J40-J45,J47,J67 | 0.01295 |
| Diseases of oral cavity, salivary glands, and jaws | 520-529 | K00-K14 | 0.00261 |
| Diseases of esophagus, stomach, and duodenum | 530-537 | K20-K31 | 0.0005 |
| Hernia of abdominal cavity | 550-553 | K40-K46 | 0.00388 |
| Infections of skin and subcutaneous tissue | 680-686 | L00-L08 | 0.00561 |
| Other inflammatory conditions | 690-698 | L10-L49, L51-L59 | -0.00053 |
| Arthropathies and related disorders | 710-719 | M00-M02, M04, M05-M09 M11-M14, M15-M19, M20-M25, M30-M36 (excluded M35.3) | 0.01408 |
| Rheumatism, excluding the back | 725-729 | M35.3, M60-M79,R25.2,R29.8x | 0.00021 |
| Dorsopathies | 720-724 | M40-M54 | 0.00984 |

## Appendix A Frailty markers

| Osteopathies, chondropathies, and acquired musculoskeletal deformities | 730-739 | M80-M85, M86-M90, M91-M95, M99 | 0.00389 |
|---|---|---|---|
| Nephritis, nephrotic syndrome, and nephrosis | 580-589 | N00-N05, N08,N17,N18, N25, N26,N27 | 0.01047 |
| Other diseases of urinary system | 590-599 | N30-N39 | 0.01062 |
| Diseases of male genital organs | 600-608 | N40-N53 | -0.02131 |
| Congenital anomalies in urinary system | 753 | Q60-Q64 | -0.00836 |
| Congenital anomalies in musculoskeletal system | 754-756 | Q65-Q79 | 0.00073 |
| Symptoms | 780-789 | R00-R39, R50-R63 (exclude R09.1, R09.2,R13,R25.2,R29.8,R51, R52) | 0.00593 |
| III-defined and unknown causes of morbidity and mortality | 797-799 | R09.1, R09.2,R41.8x,R68.13,R68.82, R64,R69,R99 | 0.01119 |
| Nonspecific abnormal findings | 790-796 | R70-R97 | -0.00231 |
| Contusion with intact skin surface | 920-924 | \$00.93, \$10.93, \$00.10-\$00.12, \$05.10-\$05.12, \$05.90-\$05.92, \$20.00-\$20.02, \$20.20-\$20.22, \$30.0-\$30.3, T14.8-T14.9, \$40.01-\$40.02, \$50.0-\$50.1, \$60.0-\$60.2, \$70.0-\$70.1, \$80.0-\$80.1, \$90.0-\$90.3 | 0.01074 |
| Open wound of lower limb | 890-897 | \$81 | 0.02042 |
| Persons with a condition influencing their health status | V40-V49 | F48.9, F52.9, F69, F81.9, H54.7, H93.9x, J95.850, M96.0, R13.10, R43.9, R46.8x, R47.89, R68.89, Z48.22-Z48.298, Z66, Z73.82, Z74.0x, Z76.82, Z78.x, Z86.59, Z87.898, Z89.0x (excluding 789.52x), 790.x (excluding (Z90.41x. Z90.71x), 791.15, 791.83, 792.82, 793.x-795.x, 796.3x-Z96.9, 797.x-799.x (excluding 798.5x, 795.87x) | 0.00191 |
| Persons without reported diagnosis encountered during examination and investigation of individuals and populations | V70-V82 | Z00-Z13 | -0.01208 |
| Persons with potential health hazards related to communicable diseases | V01-V09 | Z20-Z29 | -0.00189 |
| Persons encountering health services for specific procedures and aftercare | V50-V59 | Z40-Z53, Z79 (exclude Z48.280, Z48.23, Z48.24, Z48.288, Z48.298 , Z48.22, Z48.290) | 0.00118 |

| Condition | CPT Code | Coefficient |
|---|---|---|
| Office/other outpatient visit – established patient | 99214 | 0.00149 |
| Hospital care – initial | 99222 | 0.0017 |
| Office consultation | 99242 | -0.00094 |
| Office consultation | 99245 | 0.00169 |
| Nursing facility care – subsequent | 99308 | 0.01389 |
| Preventive medicine services | 99381-99429 | -0.00712 |
| Anesthesia – head | 00100-00222 | -0.00049 |
| Anesthesia – neck | 00300-00352 | 0.00614 |
| Anesthesia – intrathoracic | 00500-00580 | -0.01568 |
| Anesthesia – lower abdomen | 00800-00882 | -0.01053 |
| Anesthesia – knee and popliteal area | 01320-01444 | -0.01215 |
| Surgery – respiratory system | 30000-32999 | -0.00129 |
| Surgery – female genital system | 56405-58999 | 0.00327 |
| Surgery – nervous system | 61000-64999 | 0.00843 |
| Radiology – nuclear medicine | 78000-79999 | -0.00301 |
| Therapeutic drug assays | 80150-80299 | 0.00789 |
| Cytopathology | 88104-88199 | -0.01082 |
| Surgical pathology | 88300-88399 | -0.00427 |

## Appendix A Frailty markers

| Medicine – Ophthalmology | 92002-92499 | -0.00295 |
|----------------------------------------------------|-------------|----------|
| Medicine – Cardiovascular | 92950-93799 | -0.00046 |
| Medicine – Noninvasive vascular diagnostic studies | 93875-93990 | -0.00828 |
| Allergy and clinical immunology | 95004-95199 | -0.0084 |
| Physical medicine and rehabilitation | 97001-97799 | -0.00012 |
| Chiropractic manipulative treatment | 98940-98943 | -0.01426 |
| Special services, procedures and reports | 99000-99091 | 0.00127 |

| Condition | HCPCS Code | Coefficient |
|---|---|---|
| Transportation services including ambulance | A0021-A0999 | 0.01022 |
| Other supplies including diabetes supplies and contraceptives | A4244-A4290 | 0.0236 |
| Diabetic footwear | A5500-A5513 | 0.02375 |
| Breathing aids | A7000-A7046 | 0.00947 |
| Administrative, miscellaneous and experimental | A9150-A9999 | -0.00167 |
| Walking aids and attachments | E0100-E0159 | 0.02821 |
| Hospital beds and associated supplies | E0250-E0373 | 0.08649 |
| Oxygen delivery systems and related supplies | E0424-E0486 | 0.00665 |
| Humidifiers and nebulizers with related equipment | E0550-E0601 | 0.00385 |
| Wheelchair or transport chair and related accessories | E0950-E1298,<br>E2201-E2294,<br>E2300-E2399,<br>E2601-E2621 | 0.00805 |
| Accessories for oxygen delivery devices | E1353-E1406 | 0.02702 |
| Vaccine administration | G0008-G0010 | -0.00158 |
| Screening examinations and disease management training | G0101-G0124 | -0.01136 |
| Drugs, administered by injection | J0120-J7130 | 0.00664 |
| Inhalation solutions | J7608-J7684 | 0.00412 |
| Wheelchairs, components, and accessories | K0001-K0462,<br>K0669 | 0.07802 |

## Appendix A Frailty markers

Osteoporosis

| ICD10 Dx | ICD9 Dx | LongDesICD10 | LongDeslCD9 |
|---|---|---|---|
| M810 | 73300 | Age-related osteoporosis without current pathological | Osteoporosis, unspecified |
| | | fracture | |
| M810 | 73301 | Age-related osteoporosis without current pathological | Senile osteoporosis |
| | | fracture | |
| M818 | 73302 | Other osteoporosis without current pathological fracture | Idiopathic osteoporosis |
| M818 | 73303 | Other osteoporosis without current pathological fracture | Disuse osteoporosis |
| M816 | 73309 | Localized osteoporosis [Lequesne] | Other osteoporosis |
| M818 | 73309 | Other osteoporosis without current pathological fracture | Other osteoporosis |


| | _ | _ |
|---|---|---|
| 8065 | Unspecified injury to L3 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Unspecified injury to L4 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Unspecified injury to L5 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Unspecified injury to unspecified level of lumbar spinal cord, | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L1 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L2 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L3 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L4 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | encounter Complete lesion of L5 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | encounter Complete lesion of unspecified level of lumbar spinal cord | Open fracture of lumbar spine with spinal cord injury |
| | initial encounter | |
| 8065 | Incomplete lesion of L1 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L2 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L3 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L4 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L5 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of unspecified level of lumbar spinal cord, | Open fracture of lumbar spine with spinal cord injury |
| 80660 | Unspecified fracture of sacrum, initial encounter for closed | Closed fracture of sacrum and coccyx with unspecified spinal cord injury |
| 80660 | Fracture of coccyx, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with unspecified spinal cord injury |
| 80660 | Unspecified injury to sacral spinal cord, initial encounter | Closed fracture of sacrum and coccyx with unspecified spinal cord injury |
| 80661 | Unspecified fracture of sacrum, initial encounter for closed | Closed fracture of sacrum and coccyx with complete cauda equina lesion |
| 80661 | Fracture of coccyx, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with complete cauda |
| 80661 | Injury of cauda equina, initial encounter | equina lesion Closed fracture of sacrum and coccyx with complete cauda |
| 80662 | Unspecified fracture of sacrum, initial encounter for closed | equina lesion Closed fracture of sacrum and coccyx with other cauda equina |
| 80662 | fracture Fracture of coccyy, initial encounter for closed fracture | injury Closed fracture of sacrum and coccyx with other cauda equina |
| | Tracture of coccys, mittal encounter for dosed fracture | injury |
| 80662 | Injury of cauda equina, initial encounter | Closed fracture of sacrum and coccyx with other cauda equina injury |
| 80669 | Unspecified fracture of sacrum, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with other spinal cord injury |
| 80669 | Fracture of coccyx, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with other spinal cord |
| 80669 | Complete lesion of sacral spinal cord, initial encounter | injury Closed fracture of sacrum and coccyx with other spinal cord |
| 80669 | Incomplete lesion of sacral spinal cord, initial encounter | injury Closed fracture of sacrum and coccyx with other spinal cord |
| 80670 | Unspecified fracture of sacrum, initial encounter for open | Open fracture of sacrum and coccyx with unspecified spinal |
| 90670 | fracture of coccyx initial encounter for open fracture | cord injury Open fracture of sacrum and coccyx with unspecified spinal |
| 30070 | Tracture of occys, finitial encounter for open fracture | cord injury |
| | 8065 | encounter Unspecified injury to L4 level of lumbar spinal cord, initial encounter Unspecified injury to unspecified level of lumbar spinal cord, initial encounter 8065 Unspecified injury to unspecified level of lumbar spinal cord, initial encounter 8065 Complete lesion of L1 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L2 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L3 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L4 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L5 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L5 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L5 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L1 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L2 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L5 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L5 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L5 level of lumbar spinal cord, initial encounter 8066 Incomplete lesion of L5 level of lumbar spinal cord, initial encounter 8066 Incomplete lesion of L6 level of lumbar spinal cord, initial encounter 8066 Unspecified fracture of sacrum, initial encounter for closed fracture 80660 Unspecified fracture of sacrum, initial encounter for closed fracture 80661 Unspecified fracture of sacrum, initial encounter for closed fracture 80661 Fracture of coccyx, initial encounter for closed fracture 80662 Injury of cauda equina, initial encounter 80663 Unspecified fracture of sacrum, initial encounter for closed fracture 80664 Injury of cauda equina, initial encounter for closed fracture 80667 Incomplete lesion of sacral spinal cord, initial encounter for closed fracture 80669 Incomplete lesion of sacral spinal cord, initial encounter |


| end of humerus |
|----------------|
| end of humerus |
| end of numerus |
| erus |
| erus |
| erus |
| rus |
| erus |
| rus<br>rus |
| rus |
| rus<br>rus |


| fibula, initial encounter for closed fracture S82491A 82321 Other fracture of shaft of right fibula, initial encounter for closed fracture closed fracture | re of shaft of fibula alone re of shaft of fibula alone |
|---|---|
| S82491A 82321 Other fracture of shaft of right fibula, initial encounter for closed fracture | re of shaft of fibula alone |
| closed fracture | re of Shart of libura alone |
| JOETJEN DEJET TOUTHER HACKING OF SHARK OF TELL HIDDING, HILLIAN CHOOGHILLER FOR THE TOUTHER HACKING | re of shaft of fibula alone |
| closed fracture | ite of shall of libula alone |
| | re of shaft of fibula alone |
| for closed fracture | Te of shart of fibula alone |
| | re of shaft of fibula alone |
| encounter for closed fracture | Te of share of fibula atome |
| | re of shaft of fibula alone |
| encounter for closed fracture | |
| | re of shaft of fibula alone |
| encounter for closed fracture | |
| | re of shaft of fibula alone |
| encounter for closed fracture | |
| S82865A 82321 Nondisplaced Maisonneuve's fracture of left leg, initial Closed fracture | re of shaft of fibula alone |
| encounter for closed fracture | |
| S82866A 82321 Nondisplaced Maisonneuve's fracture of unspecified leg, Closed fracture | re of shaft of fibula alone |
| initial encounter for closed fracture | |
| S82201A 82322 Unspecified fracture of shaft of right tibia, initial encounter Closed fracture | re of shaft of fibula with tibia |
| for closed fracture | |
| S82202A 82322 Unspecified fracture of shaft of left tibia, initial encounter for Closed fracture | re of shaft of fibula with tibia |
| closed fracture | |
| | re of shaft of fibula with tibia |
| for closed fracture | |
| | re of shaft of fibula with tibia |
| for closed fracture | 6.1.6.6.111.1 |
| | e of shaft of tibia alone |
| for open fracture type I or II | f-h-ft -f+:h:l |
| | e of shaft of tibia alone |
| for open fracture type IIIA, IIIB, or IIIC S82202B 82330 Unspecified fracture of shaft of left tibia, initial encounter for Open fracture | e of shaft of tibia alone |
| open fracture type I or II | e of shall of tibia alone |
| | e of shaft of tibia alone |
| open fracture type IIIA, IIIB, or IIIC | |
| | e of shaft of tibia alone |
| encounter for open fracture type I or II | |
| S82221C 82330 Displaced transverse fracture of shaft of right tibia, initial Open fracture | e of shaft of tibia alone |
| encounter for open fracture type IIIA, IIIB, or IIIC | |
| S82222B 82330 Displaced transverse fracture of shaft of left tibia, initial Open fracture | e of shaft of tibia alone |
| encounter for open fracture type I or II | |
| | e of shaft of tibia alone |
| encounter for open fracture type IIIA, IIIB, or IIIC | |
| | e of shaft of tibia alone |
| initial encounter for open fracture type I or II | 6.1.6.6.00 |
| | e of shaft of tibia alone |
| initial encounter for open fracture type IIIA, IIIB, or IIIC | f -hft -f+:h:l |
| S82224B 82330 Nondisplaced transverse fracture of shaft of right tibia, initial Open fracture | e ot snatt of tibia alone |
| encounter for open fracture type I or II | a of shaft of tibia along |
| | e of shaft of tibia alone |
| encounter for open fracture type IIIA, IIIB, or IIIC S82225B 82330 Nondisplaced transverse fracture of shaft of left tibia, initial Open fracture | e of shaft of tibia alone |
| encounter for open fracture type I or II | C 5. Share of tibia alone |
| | e of shaft of tibia alone |
| encounter for open fracture type IIIA, IIIB, or IIIC | |
| | e of shaft of tibia alone |
| initial encounter for open fracture type I or II | |
| | e of shaft of tibia alone |
| initial encounter for open fracture type IIIA, IIIB, or IIIC | |


| | _ | |
|---|---|---|
| 82535 | Nondisplaced fracture of fourth metatarsal bone, unspecified | Open fracture of metatarsal bone(s) |
| 82535 | Displaced fracture of fifth metatarsal bone, right foot, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Displaced fracture of fifth metatarsal bone, left foot, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Displaced fracture of fifth metatarsal bone, unspecified foot, | Open fracture of metatarsal bone(s) |
| 82535 | Nondisplaced fracture of fifth metatarsal bone, right foot, | Open fracture of metatarsal bone(s) |
| | initial encounter for open fracture | · |
| 82535 | Nondisplaced fracture of fifth metatarsal bone, left foot, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Nondisplaced fracture of fifth metatarsal bone, unspecified foot, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Unspecified physeal fracture of right metatarsal, initial | Open fracture of metatarsal bone(s) |
| 82535 | Unspecified physeal fracture of left metatarsal, initial | Open fracture of metatarsal bone(s) |
| 82535 | Salter-Harris Type I physeal fracture of right metatarsal, | Open fracture of metatarsal bone(s) |
| 82535 | initial encounter for open fracture Salter-Harris Type I physeal fracture of left metatarsal, | Open fracture of metatarsal bone(s) |
| | initial encounter for open fracture | |
| 82535 | Salter-Harris Type II physeal fracture of right metatarsal, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Salter-Harris Type II physeal fracture of left metatarsal, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Salter-Harris Type III physeal fracture of right metatarsal, | Open fracture of metatarsal bone(s) |
| 82535 | Salter-Harris Type III physeal fracture of left metatarsal, | Open fracture of metatarsal bone(s) |
| 82535 | | Open fracture of metatarsal bone(s) |
| | initial encounter for open fracture | .,, |
| 82535 | Salter-Harris Type IV physeal fracture of left metatarsal, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Other physeal fracture of right metatarsal, initial encounter for open fracture | Open fracture of metatarsal bone(s) |
| 82535 | Other physeal fracture of left metatarsal, initial encounter | Open fracture of metatarsal bone(s) |
| 82539 | Fracture of unspecified metatarsal bone(s), right foot, initial | Other open fracture of tarsal and metatarsal bones |
| 82539 | Fracture of unspecified metatarsal bone(s), left foot, initial | Other open fracture of tarsal and metatarsal bones |
| 8260 | encounter for open fracture Displaced unspecified fracture of right great toe, initial | Closed fracture of one or more phalanges of foot |
| 0260 | encounter for closed fracture | Classifications of any angular photographs |
| 8200 | encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Nondisplaced unspecified fracture of right great toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Nondisplaced unspecified fracture of left great toe, initial | Closed fracture of one or more phalanges of foot |
| 8260 | Displaced fracture of proximal phalanx of right great toe, | Closed fracture of one or more phalanges of foot |
| 8260 | Displaced fracture of proximal phalanx of left great toe, | Closed fracture of one or more phalanges of foot |
| 8260 | initial encounter for closed fracture Displaced fracture of proximal phalanx of unspecified great | Closed fracture of one or more phalanges of foot |
| 0260 | toe, initial encounter for closed fracture | Closed fronting of any an array whelever a fifty |
| | initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Nondisplaced fracture of proximal phalanx of left great toe, initial encounter for closed fracture | Closed fracture of one or more phalanges of foot |
| 8260 | Nondisplaced fracture of proximal phalanx of unspecified | Closed fracture of one or more phalanges of foot |
| | 82535<br>82536<br>82536<br>82536<br>82536<br>82537<br>82539<br>8260 | foot, initial encounter for open fracture Displaced fracture of fifth metatarsal bone, right foot, initial encounter for open fracture Displaced fracture of fifth metatarsal bone, left foot, initial encounter for open fracture Displaced fracture of fifth metatarsal bone, unspecified foot, initial encounter for open fracture Nondisplaced fracture of fifth metatarsal bone, right foot, initial encounter for open fracture Nondisplaced fracture of fifth metatarsal bone, left foot, initial encounter for open fracture Nondisplaced fracture of fifth metatarsal bone, unspecified foot, initial encounter for open fracture Nondisplaced fracture of fifth metatarsal bone, unspecified foot, initial encounter for open fracture Unspecified physeal fracture of right metatarsal, initial encounter for open fracture Septimental fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type I physeal fracture of right metatarsal, initial encounter for open fracture Salter-Harris Type II physeal fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type II physeal fracture of right metatarsal, initial encounter for open fracture Salter-Harris Type II physeal fracture of right metatarsal, initial encounter for open fracture Salter-Harris Type III physeal fracture of right metatarsal, initial encounter for open fracture Salter-Harris Type III physeal fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type IV physeal fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type IV physeal fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type IV physeal fracture of left metatarsal, initial encounter for open fracture Salter-Harris Type IV physeal fracture of left metatarsal, initial encounter for open fracture Displaced unspecified fracture of left great toe, initial encounter for open fracture Salter-Harris Type IV physeal fracture of left great toe, initial encounter for dosed fracture Disp |


## Appendix A Frailty markers


#### Falls


## Appendix A Frailty markers

#### Combined Comorbidity Score for Claims Data

Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. Journal of Clinical Epidemiology 2011:64(7):749-59.

Sun JW. Rogers JR. Her O. Welch EC. Panozzo CA. Toh S. Gagne JJ. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. Medical Care. 2017 Dec 1:55(12):1046-51.

Codes used for each ICD-10-CM and ICD-9-CM version of the combined comorbidity score


## Appendix A Frailty markers


BM, backward mapping; GEMs, General Equivalence Mappings; FBM, forward-backward mapping; ICD-9-CM, International Classification of Diseases, 9<sup>th</sup> Revision, Clinical Modification; ICD-10-CM, International Classification of Diseases, 10<sup>th</sup> Revision, Clinical Modification

#### Lithium

| NDC Generic Name | |
|-------------------|------------------------------|
| LITHIUM ASPARTATE | LITHIUM CITRATE |
| LITHIUM CARBONATE | LITHIUM CITRATE TETRAHYDRATE |

#### Anti-epileptic mood stabilizers

| NDC Generic Name | |
|-------------------|---------------------------------------------------|
| CARBAMAZEPINE | OXCARBAZEPINE |
| DIVALPROEX SODIUM | VALPROIC ACID |
| LAMOTRIGINE | VALPROIC ACID (AS SODIUM SALT) (VALPROATE SODIUM) |

#### Anti-epileptic non-mood stabilizers

| Anti epileptie non mood stabilizers | |
|-------------------------------------|---------------|
| NDC Generic Name | |
| RUFINAMIDE | LACOSAMIDE |
| VIGABATRIN | ETHOSUXIMIDE |
| EZOGABINE | FELBAMATE |
| TIAGABINE HCL | LEVETIRACETAM |
| PHENYTOIN | TOPIRAMATE |
| ZONISAMIDE | PHENOBARBITAL |
| PRIMIDONE | GABAPENTIN |
| PREGABALIN | |

#### Atypical antipsychotics

| NDC Generic Name | |
|----------------------|---------------------|
| ZIPRASIDONE MESYLATE | ARIPIPRAZOLE |
| PALIPERIDONE | OLANZAPINE |
| ZIPRASIDONE HCL | RISPERIDONE |
| CLOZAPINE | QUETIAPINE FUMARATE |

#### Benzodiazepines

| 201120414120 | |
|-------------------------|----------------|
| NDC Generic Name | |
| ALPRAZOLAM | FLURAZEPAM HCL |
| CHLORDIAZEPOXIDE | LORAZEPAM |
| CLOBAZAM | MIDAZOLAM |
| CLONAZEPAM | OXAZEPAM |
| CLORAZEPATE DIPOTASSIUM | QUAZEPAM |
| DIAZEPAM | TEMAZEPAM |
| ESTAZOLAM | TRIAZOLAM |

#### Serotonin-norepinephrine reuptake inhibitor

| NDC Generic Name | |
|--------------------------|---------------------|
| DESVENLAFAXINE | DULOXETINE HCL |
| DESVENLAFAXINE FUMARATE | VENLAFAXINE HCL |
| DESVENLAFAXINE SUCCINATE | LEVOMILNACIPRAN HCL |

#### Selective serotonin reuptake inhibitor

| NDC Generic Name | |
|---------------------------|-----------------------------------------|
| PAROXETINE MESYLATE | CITALOPRAM HYDROBROMIDE |
| FLUOXETINE | FLUOXETINE HCL |
| OLANZAPINE/FLUOXETINE HCL | SERTRALINE HCL |
| FLUVOXAMINE MALEATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.17 |
| ESCITALOPRAM OXALATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.8 |
| PAROXETINE HCL | VILAZODONE HCL |

#### Tricyclic antidepressants

| NDC Generic Name | | |
|------------------------------------|--------------------------------|---|
| PROTRIPTYLINE HCL | DESIPRAMINE HCL | • |
| IMIPRAMINE PAMOATE | PERPHENAZINE/AMITRIPTYLINE HCL | |
| TRIMIPRAMINE MALEATE | NORTRIPTYLINE HCL | |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE HCL | |
| AMOXAPINE | DOXEPIN HCL | |
| CLOMIPRAMINE HCL | AMITRIPTYLINE HCL | • |

#### Typical antipsychotics

| NDC Generic Name | |
|------------------------|--------------------------------|
| FLUPHENAZINE ENANTHATE | THIOTHIXENE |
| LOXAPINE | FLUPHENAZINE HCL |
| PIMOZIDE | PERPHENAZINE/AMITRIPTYLINE HCL |

| MESORIDAZINE BESYLATE | TRIFLUOPERAZINE HCL |
|------------------------|---------------------|
| MOLINDONE HCL | CHLORPROMAZINE HCL |
| THIOTHIXENE HCL | HALOPERIDOL |
| FLUPHENAZINE DECANOATE | THIORIDAZINE HCL |
| PERPHENAZINE | |

#### Anticoagulants

| NDC Generic Name | |
|---|---|
| APIXABAN | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE |
| DABIGATRAN ETEXILATE MESYLATE | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE/PF |
| DALTEPARIN SODIUM,PORCINE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER |
| EDOXABAN TOSYLATE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER/PF |
| ENOXAPARIN SODIUM | HEPARIN SODIUM, PORCINE/PF |
| FONDAPARINUX SODIUM | RIVAROXABAN |
| HEPARIN SODIUM,BEEF | TINZAPARIN SODIUM,PORCINE |
| HEPARIN SODIUM, PORCINE | WARFARIN SODIUM |
| HEPARIN SODIUM, PORCINE IN 0.45 % SODIUM CHLORIDE | |

#### Antiplatelet agents

| ASPIRIN/CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN CIOPIDOGREL BISULFATE ASPIRIN/ACETAMINOPHEN ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE CODEINE PHOSPHATE/CARISOPODOU/ASPIRIN ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE/ASPIRIN/CAFFEINE ASPIRIN/CALCIUM CARBONATE DIHYDROCODEINE/ASPIRIN/CAFFEINE ASPIRIN/CALCIUM CARBONATE HYDROCODO BITARTRATE/ASPIRIN/CAFFEINE BEPLOINE/ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN BYRIN/CALCIUM CARBONATE/MAGNESIUM METHOCABBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CODEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLEROPANOLAMINE BITARTRATE/ASPIRIN/CHIORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHIORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHIORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHIORPHENIRAMINE ASPIRIN/SALICYAMIDE/CAETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHIORPHENIRAMINE ASPIRIN/SALICYAMIDE/CAETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHIORPHENIRAMINE CHIORPHENIRAMINE M | Antiplatelet agents | |
|---|---|---|
| ASPIRIN (CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN CLOPIDOGREL ISULIFATE ASPIRIN/ACETAMINOPHEN ASPIRIN/ACETAMINOPHEN ASPIRIN/ACETAMINOPHEN/CAFFEINE CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN ASPIRIN/ACETAMINOPHEN/CAFFEINE CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CARGUM CARBONATE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/CAFFEINE ASPIRIN/CACETAMINOPHEN/CARGUM CARBONATE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE DIPYRIDAMOLE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN DIPYRIDAMOLE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ORPHENADRINE CITRATE/ASPIRIN ASPIRIN/COLEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/COLEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BITTARTATE/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE JO-METHORPHAN HB/ASPIRIN CARGONATE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE JO-METHORPHAN HB/ASPIRIN CHARGEMENTAMINE A | NDC Generic Name | |
| ASPIRIN (CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM DIHYDROCODEINE/BASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE/BASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE DIHYDROCODEINE/BASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN DIHYDROCODEINE/BASPIRIN/CAFFEINE ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE HYDROCODONE BITARTATE/ASPIRIN ASPIRIN/CALCIUM CARBONATE HYDROCODONE BITARTATE/ASPIRIN ASPIRIN/CALCIUM CARBONATE HYDROCODONE BITARTATE/ASPIRIN ASPIRIN/CALCIUM CARBONATE HYDROCODONE BITARTATE/ASPIRIN ASPIRIN/CALCIUM CARBONATE HYDROCODONE BITARTATE/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE OXYCODONE HCI/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCI/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCI/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCI/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCI/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/CAPFEINE DIPHONEPHRINE HCI/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/CAPFEINE PHENYLEPORANOLAMINE BITARTATE/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/CITRIC ACID PENTAZOCINE HCI/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE HCI/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE HCI/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCI/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCI/ASPIRIN/CHLORPHENIRAMINE CARISOPRODOL/ASPIRIN PHENYLPROPANOLAMINE HCI/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAI/PHENYLEPHRINE | ABCIXIMAB | CILOSTAZOL |
| ASPIRIN/ACETAMINOPHEN ASPIRIN/ACETAMINOPHEN/CAFFEINE CODEINE PHOSPHATE/BUTALBTAL/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE/CALCIUM CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFEINE/POTASSIUM DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN DIPYRIDAMOLE ASPIRIN/CAFFEINE BPHEDRINE/ASPIRIN/CAFFEINE EPHEDRINE/ASPIRIN/CAFFEINE ASPIRIN/CALCIUM CARBONATE HYDROCODONE BITARTRATE/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/DIPHENHOPRAMINE CITRATE OXYCODONE HICARSPIRIN/CAFFEINE ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HICARSPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HICARSPIRIN ASPIRIN/DIPHENHYDRAMINE HICL OXYCODONE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HICL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HICL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE MICROPAUMINUM AMINOACETATI PHENYLEPHRINE HICL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLEPHRINE HICL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE HICL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE HICL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE HICL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE HICL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SOLIUM BICARBONATE/CITRIC ACID PHENYLPROPANOLAMINE HICL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SOLIUM BICARBONATE/CITRIC ACID PHENYLPROPANOLAMINE HICL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE BITARTRATE/ASPIRIN PRESUDOEPHEDRINE HICL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE BITARTRATE/ASPIRIN PROBAMATE | ASPIRIN | CINNAMEDRINE HCL/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE/CALCIUM CODEINE/ASPIRIN/SALICYLAMIDOPHEN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFFEINE/CASSIUM DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CAFEINE ASPIRIN/ACETAMINOPHEN/CAFEINE DIHYDROCODEINE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEINE DIHYDROCODEINE/ASPIRIN/CAFFEINE ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN BIPRIN/CALCIUM CARBONATE ASPIRIN/CAFEINE ASPIRIN/CALCIUM CARBONATE HYDROCODONE BITARTRATE/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCABBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE ASPIRIN/CODEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPRENHYDRAMINE CITRATE ASPIRIN/DIPRENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID ASPIRIN/DIPRENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPRIDAMOLE ASPIRIN/DIPRIDAMOLE ASPIRIN/DIPRIDAMOLE ASPIRIN/DIPRIDAMOLE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLEPRIPINE HCL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLEPRIPINE HCL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE CARISORODOL/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN TICAGEALOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGEALOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGEALOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TOGAGEALOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TOGAGEALOR TORMEN TO THE TARTATE ASPIRIN TOGAGEALOR TORMEN TORMEN TO THE TARTATE ASPIRIN TOG | ASPIRIN (CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN | CLOPIDOGREL BISULFATE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN DIHYDROCODEINE/ASPIRIN/CAFFEINE ASPIRIN/CAFEINE EPHEDRINE/ASPIRIN/ACETAMILDE/CAFFEINE ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/COLIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE GITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PHENTAZOCINE HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALIC | ASPIRIN/ACETAMINOPHEN | CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFERIN DIPYRIDAMOLE ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM ASPIRIN/CALCIUM CARBONATE/MAGNESIUM ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CODEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCIUE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCIUE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCIUE HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN TOTAGERICA CARISORODOLASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN TOTAGERICA TOTAGE TOTAGE TOTAGE TOTAGE | ASPIRIN/ACETAMINOPHEN/CAFFEINE | CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN |
| ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN DIPYRIDAMOLE ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN DIPYRIDAMOLE ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE HYDROCODONE BITARTRATE/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ORPHENADRINE CITRATE/ASPIRIN ASPIRIN/CODEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCIAL HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLEPPRINE HCL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MALL/PHENYLEPHRINE BITARTRATE/ASPIRIN PROPOXYPHENE HCL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MALL/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARAPA ARTHRITIS PAIN | ASPIRIN/ACETAMINOPHEN/CAFFEINE/CALCIUM | CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZCINE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZCINE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZCINE HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGRELOR ARTHRITIS PAIN FORMULA A-F ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN FORMULA A-F ECOTRIN MAYAP ARTHRITIS PAIN | ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM | DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM ASPIRIN/CALCIUM CARBONATE/MAGNESIUM ASPIRIN/CALCIUM CARBONATE/MAGNESIUM ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CODEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPYRIDAMOLE PHENYLEPHRINE HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLEPHRINE HCL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SAUCYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE ASPIRIN/SAUCYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE CARISOPRODOL/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE BAYER ASPIRIN ARTHRITIS PAIN FORMULA A-F ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN FORMULA A-F ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN MAPAP ARTHRITIS PAIN | ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE | DIHYDROCODEINE/ASPIRIN/CAFFEINE |
| ASPIRIN/CALCIUM CARBONATE ASPIRIN/CALCIUM CARBONATE/MAGNESIUM ASPIRIN/CALCIUM CARBONATE/MAGNESIUM ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE OXYCODODIE HCL/ASPIRIN ASPIRIN/CODEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPYRIDAMOLE PHENYLEPHRINE HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SAULCYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SAULCYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SAULCYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SOULUM BICARBONATE/CITRIC ACID PRASUGREL HCL PRASUGREL HCL ASPIRIN/SOULUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE /BITARTRATE/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MAL/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MAL/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MAL/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA A-F ARTHRITIS PAIN FORMULA A-F ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARAPA ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH | ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN | DIPYRIDAMOLE |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM METHOCARBAMOL/ASPIRIN ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE ASPIRIN/CODEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMOLE PHENYLEPHRINE HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE BITARTRATE/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN FORMULA ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER | ASPIRIN/CAFFEINE | EPHEDRINE/ASPIRIN/ACETANILIDE/CAFFEINE |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE ASPIRIN/CODEINE PHOSPHATE OXYCODONE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL OXYCODONE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CACFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN MAPAP ARTHRITIS PAIN PARTHRITIS PAIN RELIEVER | ASPIRIN/CALCIUM CARBONATE | HYDROCODONE BITARTRATE/ASPIRIN |
| ASPIRIN/CODEINE PHOSPHATE ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN ASPIRIN/DIPHENHYDRAMINE CITRATE OXYCODONE ASPIRIN ASPIRIN/DIPHENHYDRAMINE HCL ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/MIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID PHENYLEPHRINE HCL/ASPIRIN ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALFENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NOC BRANCH MAME ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN RELIEF ECOTRIN MAPAP ARTHRITIS PAIN MAPAP ARTHRITIS PAIN MAPAP ARTHRITIS PAIN | ASPIRIN/CALCIUM CARBONATE/MAGNESIUM | METHOCARBAMOL/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE CITRATE ASPIRIN/DIPHENHYDRAMINE HCL ASPIRIN/DIPHENHYDRAMINE HCL ASPIRIN/DIPHENHYDRAMINE HCL ASPIRIN/DIPHENHYDRAMINE SODIUM BICARBONATE/CITRIC ACID PENTAZOCINE HCL/ASPIRIN ASPIRIN/DIPYRIDAMOLE ASPIRIN/DIPYRIDAMOLE ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN DOC Brand Name ARTHRITIS PAIN ARTHRITIS PAIN BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF | ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE | ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/DIPHENHYDRAMINE HCL ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID ASPIRIN/DIPYRIDAMOLE ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLEPHRINE HCL/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN CARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN ARTHRITIS PAIN RELIEVER | ASPIRIN/CODEINE PHOSPHATE | OXYCODONE HCL/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID ASPIRIN/DIPYRIDAMOLE ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MEPROBAMATE ASPIRIN/MEPROBAMATE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE ARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN WORAPAXAR SULFATE BAYER ASPIRIN BAYER ASPIRIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH MAPAP ARTHRITIS PAIN BAPA ARTHRITIS PAIN BAPA ARTHRITIS PAIN MAPAP ARTHRITIS PAIN MAPAP ARTHRITIS PAIN | ASPIRIN/DIPHENHYDRAMINE CITRATE | OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| ASPIRIN/DIPYRIDAMOLE ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CAFFEINE ARISOPRODOL/ASPIRIN PRESUDGEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN BAYER ASPIRIN ARTHRITIS PAIN BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA AFFIRITIS PAIN FORMULA AFFIRITIS PAIN RELIEF ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN | ASPIRIN/DIPHENHYDRAMINE HCL | OXYCODONE/ASPIRIN |
| ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/MEPROBAMATE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MALL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE MDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF | ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID | PENTAZOCINE HCL/ASPIRIN |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE ASPIRIN/MEPROBAMATE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN BAPAP ARTHRITIS PAIN | ASPIRIN/DIPYRIDAMOLE | PHENYLEPHRINE HCL/ASPIRIN |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN ASPIRIN/MEPROBAMATE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA A-F ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN MAPAP ARTHRITIS PAIN MAPAP ARTHRITIS PAIN | ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN |
| ASPIRIN/MEPROBAMATE ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN BAYER ASPIRIN ARTHRITIS PAIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN | ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE ASPIRIN/SALICYLAMIDE/CAFFEINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN BAYER ASPIRIN ARTHRITIS PAIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA A-F ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN | ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN |
| ASPIRIN/SALICYLAMIDE/CAFFEINE PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE ASPIRIN/SODIUM BICARBONATE/CITRIC ACID PRASUGREL HCL BUTALBITAL/ASPIRIN/CAFFEINE PROPOXYPHENE HCL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN TICAGRELOR CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN MAPAP ARTHRITIS PAIN | ASPIRIN/MEPROBAMATE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/SODIUM BICARBONATE/CITRIC ACID BUTALBITAL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN | ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE |
| BUTALBITAL/ASPIRIN/CAFFEINE CARISOPRODOL/ASPIRIN CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN | ASPIRIN/SALICYLAMIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE |
| CARISOPRODOL/ASPIRIN PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN | ASPIRIN/SODIUM BICARBONATE/CITRIC ACID | PRASUGREL HCL |
| CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN VORAPAXAR SULFATE NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN | BUTALBITAL/ASPIRIN/CAFFEINE | PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN NDC Brand Name ARTHRITIS PAIN ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA -F ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEF MAPAP ARTHRITIS PAIN | CARISOPRODOL/ASPIRIN | PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| NDC Brand Name ARTHRITIS PAIN BAYER ASPIRIN ARTHRITIS PAIN FORMULA BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN | CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN | TICAGRELOR |
| ARTHRITIS PAIN ARTHRITIS PAIN FORMULA BAYER ASPIRIN MAXIMUM ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN | CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN | VORAPAXAR SULFATE |
| ARTHRITIS PAIN FORMULA ARTHRITIS PAIN FORMULA A-F ECOTRIN ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN | NDC Brand Name | |
| ARTHRITIS PAIN FORMULA A-F ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN | ARTHRITIS PAIN | BAYER ASPIRIN |
| ARTHRITIS PAIN RELIEF ECOTRIN MAXIMUM STRENGTH ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN | ARTHRITIS PAIN FORMULA | BAYER ASPIRIN MAXIMUM |
| ARTHRITIS PAIN RELIEVER MAPAP ARTHRITIS PAIN | ARTHRITIS PAIN FORMULA A-F | ECOTRIN |
| | ARTHRITIS PAIN RELIEF | ECOTRIN MAXIMUM STRENGTH |
| BAYER ARTHRITIS PAIN REGIMEN PLAVIX | ARTHRITIS PAIN RELIEVER | MAPAP ARTHRITIS PAIN |
| THE PARTY OF THE P | BAYER ARTHRITIS PAIN REGIMEN | PLAVIX |

#### Angiotensin II Receptor Blockers

| NDC Generic Name | |
|---|---|
| ALISKIREN/VALSARTAN | LOSARTAN POTASSIUM |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | LOSARTAN POTASSIUM/HYDROCHLOROTHIAZIDE |
| AMLODIPINE BESYLATE/VALSARTAN | OLMESARTAN MEDOXOMIL |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZID |
| AZILSARTAN MEDOXOMIL | OLMESARTAN MEDOXOMIL/HYDROCHLOROTHIAZIDE |
| AZILSARTAN MEDOXOMIL/CHLORTHALIDONE | TELMISARTAN |
| CANDESARTAN CILEXETIL | TELMISARTAN/AMLODIPINE BESYLATE |
| CANDESARTAN CILEXETIL/HYDROCHLOROTHIAZIDE | TELMISARTAN/HYDROCHLOROTHIAZIDE |
| IRBESARTAN | VALSARTAN |

| IRBESARTAN/HYDROCHLOROTHIAZIDE | VALSARTAN/HYDROCHLOROTHIAZIDE |
|--------------------------------|--------------------------------|
| NDC Brand Name | · |
| AMLODIPINE-VALSARTAN | EXFORGE HCT |
| ATACAND | HYZAAR |
| ATACAND HCT | IRBESARTAN |
| AVALIDE | IRBESARTAN-HYDROCHLOROTHIAZIDE |
| AVAPRO | LOSARTAN POTASSIUM |
| AZOR | LOSARTAN-HYDROCHLOROTHIAZIDE |
| BENICAR | MICARDIS |
| BENICAR HCT | MICARDIS HCT |
| CANDESARTAN CILEXETIL | TELMISARTAN |
| CANDESARTAN-HYDROCHLOROTHIAZID | TELMISARTAN-AMLODIPINE |
| COZAAR | TELMISARTAN-HYDROCHLOROTHIAZID |
| DIOVAN | TRIBENZOR |
| DIOVAN HCT | TWYNSTA |
| EDARBI | VALSARTAN |
| EDARBYCLOR | VALSARTAN-HYDROCHLOROTHIAZIDE |
| EXFORGE | VALTURNA |

| Angiotensin Converting Enzyme inhibitors | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | LISINOPRIL |
| BENAZEPRIL HCL | LISINOPRIL/HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL/HYDROCHLOROTHIAZIDE | MOEXIPRIL HCL |
| CAPTOPRIL | MOEXIPRIL HCL/HYDROCHLOROTHIAZIDE |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | PERINDOPRIL ERBUMINE |
| ENALAPRIL MALEATE | QUINAPRIL HCL |
| ENALAPRIL MALEATE/FELODIPINE | QUINAPRIL HCL/HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE/HYDROCHLOROTHIAZIDE | RAMIPRIL |
| ENALAPRILAT DIHYDRATE | TRANDOLAPRIL |
| FOSINOPRIL SODIUM | TRANDOLAPRIL/VERAPAMIL HCL |
| FOSINOPRIL SODIUM/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ACCUPRIL | LOTREL |
| ACCURETIC | LYTENSOPRIL |
| ACEON | LYTENSOPRIL-90 |
| ALTACE | MAVIK |
| AMLODIPINE BESYLATE-BENAZEPRIL | MOEXIPRIL HCL |
| BENAZEPRIL HCL | MOEXIPRIL-HYDROCHLOROTHIAZIDE |
| BENAZEPRIL HCL-HCTZ | MONOPRIL |
| BENAZEPRIL-HYDROCHLOROTHIAZIDE | MONOPRIL HCT |
| CAPOTEN | PERINDOPRIL ERBUMINE |
| CAPOZIDE | PRINIVIL |
| CAPTOPRIL | PRINZIDE |
| CAPTOPRIL-HYDROCHLOROTHIAZIDE | QUINAPRIL |
| CAPTOPRIL/HYDROCHLOROTHIAZIDE | QUINAPRIL HCL |
| ENALAPRIL MALEATE | QUINAPRIL-HYDROCHLOROTHIAZIDE |
| ENALAPRIL MALEATE-HCTZ | QUINARETIC |
| ENALAPRIL MALEATE/HCTZ | RAMIPRIL |
| ENALAPRIL-HYDROCHLOROTHIAZIDE | TARKA |
| ENALAPRILAT | TRANDOLAPRIL |
| EPANED | TRANDOLAPRIL-VERAPAMIL |
| FOSINOPRIL SODIUM | UNIRETIC |
| FOSINOPRIL-HYDROCHLOROTHIAZIDE | UNIVASC |
| LEXXEL | VASERETIC |
| LISINOPRIL | VASOTEC |
| LISINOPRIL-HCTZ | VASOTEC I.V. |
| LISINOPRIL-HYDROCHLOROTHIAZIDE | ZESTORETIC |
| LOTENSIN | ZESTRIL |
| LOTENSIN HCT | |

#### Beta blockers

| 2014 210411010 | |
|-------------------------|------------------------------------------|
| NDC Generic Name | |
| ACEBUTOLOL HCL | ESMOLOL HCL |
| ATENOLOL | LABETALOL HCL |
| ATENOLOL/CHLORTHALIDONE | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL SUCCINATE/HYDROCHLOROTHIAZIDE |
| BISOPROLOL FUMARATE | METOPROLOL TARTRATE |

| BISOPROLOL FUMARATE/HYDROCHLOROTHIAZIDE | METOPROLOL TARTRATE/HYDROCHLOROTHIAZIDE |
|---|---|
| BRIMONIDINE TARTRATE/TIMOLOL MALEATE | NEBIVOLOL HCL |
| CARTEOLOL HCL | SOTALOL HCL |
| CARVEDILOL | TIMOLOL |
| CARVEDILOL PHOSPHATE | TIMOLOL MALEATE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE | TIMOLOL MALEATE/HYDROCHLOROTHIAZIDE |
| DORZOLAMIDE HCL/TIMOLOL MALEATE/PF | TIMOLOL MALEATE/PF |
| NDC Brand Name | |
| ACEBUTOLOL HCL | ISTALOL |
| ATENOLOL | KERLONE |
| ATENOLOL W/CHLORTHALIDONE | LABETALOL HCL |
| ATENOLOL-CHLORTHALIDONE | LOPRESSOR |
| BETAPACE | LOPRESSOR HCT |
| BETAPACE AF | METOPROLOL SUCCINATE |
| BETAXOLOL HCL | METOPROLOL TARTRATE |
| BETIMOL | METOPROLOL-HYDROCHLOROTHIAZIDE |
| BETOPTIC | NORMODYNE |
| BETOPTIC S | OCUPRESS |
| BISOPROLOL FUMARATE | SECTRAL |
| BISOPROLOL FUMARATE-HCTZ | SENORMIN |
| BISOPROLOL FUMARATE/HCTZ | SORINE |
| BISOPROLOL-HYDROCHLOROTHIAZIDE | SOTALOL |
| BLOCADREN | SOTALOL AF |
| BREVIBLOC | SOTALOL HCL |
| BYSTOLIC | TENORETIC 100 |
| CARTEOLOL HCL | TENORETIC 50 |
| CARTROL | TENORMIN |
| CARVEDILOL | TENORMIN CALENDAR PAK |
| COMBIGAN | TIMOLIDE |
| COREG | TIMOLOL MALEATE |
| COREG CR | TIMOPTIC |
| COSOPT | TIMOPTIC OCUDOSE |
| COSOPT PF | TIMOPTIC-XE |
| DORZOLAMIDE-TIMOLOL | TOPROL XL |
| DUTOPROL | TRANDATE |
| ESMOLOL HCL | ZEBETA |
| HYPERTENSOLOL | ZIAC |

#### Calcium channel blockers

| Calcium channel blockers | |
|---|---|
| HCPCS | |
| C9248 | |
| NDC Generic Name | |
| ALISKIREN HEMIFUMARATE/AMLODIPINE BESYLATE | BEPRIDIL HCL |
| ALISKIREN HEMIFUMARATE/AMLODIPINE/HYDROCHLOROTHIAZIDE | CLEVIDIPINE BUTYRATE |
| AMLODIPINE BESYLATE | DILTIAZEM HCL |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | DILTIAZEM HCL IN 0.9 % SODIUM CHLORIDE |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | DILTIAZEM HCL/DEXTROSE 5 % IN WATER |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | DILTIAZEM MALATE |
| AMLODIPINE BESYLATE/VALSARTAN | ENALAPRIL MALEATE/FELODIPINE |
| AMLODIPINE BESYLATE/VALSARTAN/HYDROCHLOROTHIAZIDE | |
| NDC Brand Name | |
| ADALAT | ISOPTIN |
| ADALAT CC | ISOPTIN SR |
| AFEDITAB CR | ISRADIPINE |
| AMLODIPINE BESILATE | LEXXEL |
| AMLODIPINE BESYLATE | LOTREL |
| AMLODIPINE BESYLATE-BENAZEPRIL | MATZIM LA |
| AMLODIPINE-ATORVASTATIN | NICARDIPINE HCL |
| AMLODIPINE-VALSARTAN | NICARDIPINE HCL-D5W |
| AMTURNIDE | NIFEDIAC CC |
| AZOR | NIFEDICAL XL |
| CADUET | NIFEDIPINE |
| CALAN | NIFEDIPINE ER |
| CALAN SR | NIFEDIPINE XL |
| CARDENE | NIMODIPINE |
| CARDENE I.V. | NIMOTOP |
| CARDENE SR | NISOLDIPINE |
| CARDIZEM | NORVASC |

| NYMALIZE |
|------------------------|
| PLENDIL |
| POSICOR |
| PROCARDIA |
| PROCARDIA XL |
| SULAR |
| TARKA |
| TAZTIA XT |
| TEKAMLO |
| TELMISARTAN-AMLODIPINE |
| TIAMATE |
| TIAZAC |
| TRANDOLAPRIL-VERAPAMIL |
| TRIBENZOR |
| TWYNSTA |
| VASCOR |
| VERAPAMIL ER |
| VERAPAMIL ER PM |
| VERAPAMIL HCL |
| VERAPAMIL SR |
| VERELAN |
| VERELAN PM |

#### Diuretics

| NDC Generic Name | |
|-----------------------------------|---------------------|
| AMILORIDE HCL | HYDROCHLOROTHIAZIDE |
| AMILORIDE HCL/HYDROCHLOROTHIAZIDE | HYDROFLUMETHIAZIDE |
| BENDROFLUMETHIAZIDE | INDAPAMIDE |
| BUMETANIDE | METHYCLOTHIAZIDE |
| CHLOROTHIAZIDE | METOLAZONE |
| CHLORTHALIDONE | POLYTHIAZIDE |
| EPLERENONE | SPIRONOLACTONE |
| ETHACRYNATE SODIUM | TORSEMIDE |
| ETHACRYNIC ACID | TRIAMTERENE |
| FUROSEMIDE | TRICHLORMETHIAZIDE |

#### Nitrates

| Nitrates | |
|---|---|
| NDC Generic Name | |
| ISOSORBIDE DINITRATE | NITROGLYCERIN |
| ISOSORBIDE DINITRATE/HYDRALAZINE HCL | NITROGLYCERIN/DEXTROSE 5 % IN WATER |
| ISOSORBIDE MONONITRATE | RANOLAZINE |
| NDC Brand Name | |
| ANG-O-SPAN | NITRO-TRANS SYSTEM |
| ANGINABID | NITRO-TRANSDERMAL |
| BIDIL | NITRO-TRANSDERMAL SYSTEM |
| CARDABID | NITROBART |
| DEPONIT | NITROCAP |
| DILATRATE-SR | NITROCINE |
| IMDUR | NITROCOT |
| ISD | NITRODISC |
| ISMO | NITROGARD |
| ISO-BID | NITROGLYCERIN |
| ISO-D | NITROGLYCERIN IN D5W |
| ISOCHRON | NITROGLYCERIN PATCH |
| ISODITRATE | NITROGLYCERIN T/R |
| ISONATE | NITROGLYN |
| ISONATE TR | NITROGYLCERIN |
| ISOR-BID | NITROL |
| ISORDIL | NITROLINGUAL |
| ISORDIL TITRADOSE | NITROMED |
| ISOREX-10 | NITROMIST |
| ISOREX-2.5 | NITRONAL |
| ISOREX-5 | NITRONG |
| ISOSORBIDE DINITRATE | NITROQUICK |
| ISOSORBIDE MONONITRATE | NITROREX |
| ISOSORBIDE MONONITRATE ER | NITROSPAN |
| ISOTRATE | NITROSTAT |

| ISOTRATE ER | NITROSTAT IV |
|--------------------------|-----------------|
| KENSORBIDE | NITROSTAT SR |
| LEMOTRATE | NITROTAB |
| MI-TRATES 2.5 | NITROTYM |
| MI-TRATES 6.5 | NTG |
| MINITRAN | NTS |
| MONOKET | ONSET-10 |
| N-G-C | ONSET-5 |
| N.T.S. | RANEXA |
| NITREK | RECTIV |
| NITRO | SORATE-2.5 |
| NITRO MAST TIMED RELEASE | SORATE-40 |
| NITRO S.A. | SORATE-5 |
| NITRO T.D. | SORBATE-10 |
| NITRO TRANSDERM | SORBATE-5 |
| NITRO TRANSDERMAL | SORBIDE |
| NITRO-BID | SORBITRATE |
| NITRO-BID IV | SORBITRATE SA |
| NITRO-CAPS TIME DOSE | TRANSDERM-NITRO |
| NITRO-DUR | TRATES |
| NITRO-PAR | TRIDIL |
| NITRO-TD-ACA | WF-NITRO |
| NITRO-TIME | |

Lipid lowering drugs

| Lipid lowering drugs | |
|---|---|
| NDC Generic Name | |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | METHYLTETRAHYDROFOLATE GLUCOSAMINE/NIACINAMIDE/CUPRIC &ZN OX |
| ARGININE/NIACIN/YOHIMBE BARK/GINSENG/GNK/DAMIANA/SCHISANDRA | NIACIN |
| ATORVASTATIN CALCIUM | NIACIN (INOSITOL NIACINATE) |
| BETA-CAROTENE(A) W-C & E/NIACINAMIDE/VIT B2/LUT/MIN/GLU-ONE | NIACIN/CAPSAICIN/YOHIMBE BARK/GINSENG/GNK BI EX/DAMIANA/OATS |
| CERAMIDES 1,3,6-11/NIACINAMIDE | NIACIN/LOVASTATIN |
| CERAMIDES 1,3,6-11/NIACINAMIDE/HYALURONIC ACID | NIACIN/SIMVASTATIN |
| CHOLESTYRAMINE | NIACINAMIDE |
| CHOLESTYRAMINE (WITH SUGAR) | NIACINAMIDE ASCORBATE |
| CHOLESTYRAMINE/ASPARTAME | NIACINAMIDE/AZELAIC ACID/ZINC OXIDE/VIT B6/COPPER/FA |
| COLESEVELAM HCL | NIACINAMIDE/RIBOFLAVIN/BETA-CAROTENE(A) W-C & E/MINERALS |
| COLESTIPOL HCL | NIACINAMIDE/VIT B6/VIT C/FA/COPPER/MG CIT/ZN GLUC/ALIP ACID |
| EZETIMIBE | PECTIN/INOSITOL/BIOFLAVONOIDS/NIACIN/SOYBEAN |
| EZETIMIBE/ATORVASTATIN CALCIUM | PITAVASTATIN CALCIUM |
| EZETIMIBE/SIMVASTATIN | POLICOSANOL/INOSITOL NIACINATE/GARLIC |
| FENOFIBRATE | PRAVASTATIN SODIUM |
| FENOFIBRATE NANOCRYSTALLIZED | ROSUVASTATIN CALCIUM |
| FENOFIBRATE,MICRONIZED | SIMVASTATIN |
| FLUVASTATIN SODIUM | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| FOLIC ACID/NIACINAMIDE/CUPRIC OXIDE/ZINC OXIDE | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/CYANOCOBALAMIN/PROTEASE |
| FOLIC ACID/NIACINAMIDE/ZINC | THIAMINE HCL/RIBOFLAVIN/NIACINAMIDE/DEXPANTHENOL/PYRIDOXINE |
| GEMFIBROZIL | THIAMINE M.NIT/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/C/FA |
| INOSITOL NIACINATE | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/B6/B12/VIT C/FA |
| IRON FUMARATE & POLYSAC COMP/FOLIC ACID/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/VIT B6/B12/IRON |
| IRON FUMARATE & POLYSAC COMP/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/PANT ACID/B6/IRON/METHION/CHOLINE |
| IRON PYROPHOSPHATE/CYANOCOBALAMIN/FA/NIACIN/PYRIDOXINE HCL | VIT B2/NIACINAMIDE/PYRIDOXINE HCL/CYANOCOBALAMIN/D-PANTHENOL |
| LECITHIN/SITOSTEROLS/NIACIN/BETAINE/CHITOSAN | VIT C/PYRIDOXINE HCL/NIACIN/FA/VIT B12/HERBAL COMPLEX NO.192 |
| LOVASTATIN | VITAMIN B COMPLEX NO.12/NIACINAMIDE |
| LYSINE HCL/NIACINAMIDE/THIAMINE | VITAMIN B COMPLEX/NIACINAMIDE/PANTOTHENIC ACID/HERBAL DRUGS |
| MELATONIN/TRYPTOPHAN/VALERIAN/CHAMOMILE/NIACIN/INOSITOL/B6 | |

#### Non-insulin diabetes medications

| Non-insulin diabetes inedications | |
|--------------------------------------|-------------------------------------|
| NDC Generic Name | |
| ACARBOSE | MIGLITOL |
| ACETOHEXAMIDE | NATEGLINIDE |
| ALOGLIPTIN BENZOATE | PIOGLITAZONE HCL |
| ALOGLIPTIN BENZOATE/METFORMIN HCL | PIOGLITAZONE HCL/GLIMEPIRIDE |
| ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL | PIOGLITAZONE HCL/METFORMIN HCL |
| CANAGLIFLOZIN/METFORMIN HCL | REPAGLINIDE |
| CHLORPROPAMIDE | REPAGLINIDE/METFORMIN HCL |
| GLIMEPIRIDE | ROSIGLITAZONE MALEATE |
| GLIPIZIDE | ROSIGLITAZONE MALEATE/GLIMEPIRIDE |
| GLIPIZIDE/METFORMIN HCL | ROSIGLITAZONE MALEATE/METFORMIN HCL |

| GLYBURDE/METFORMIN HCL UNAGUPTIN METFORNININ ACARDOSE LCN-TOLAM ACACTOHLUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTOPILUS MET ACTORIUS MET INVOKAMET AVANDAMET AV | GLYBURIDE | SAXAGLIPTIN HCL |
|---|---|---|
| INAGIPTIN/METFORMIN HCI. METFORMIN HCI. METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOUNE METFORMIN/CAFFEIRE/AMINO ACIDS #7/HERBAL COMB.#125/CHOUNE BIT TOLBUTAMIDE METFORMIN/CAFFEIRE/AMINO ACIDS #7/HERBAL COMB.#125/CHOUNE BIT TOLBUTAMIDE MOD Brand Name ACARBOSE ACATOPLUS MET ACTOPLUS MET ACTOPLUS MET ACTOPLUS MET INVOKAMET ACTOPLUS MET INVOKAMET ACTOPLUS MET INVOKAMET ACTOPLUS MET INVOKAMET ACTOPLUS MET INVOKAMET ACTORIUS MET INVOKAMET A | GLYBURIDE/METFORMIN HCL | SAXAGLIPTIN HCL/METFORMIN HCL |
| METFORMIN HCL METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOLINE METFORMIN/CAFFEINE/AMINO ACIDS.#7/HERBAL COMB.#125/CHOLINE METFORMIN/CAFFEINE/AMINO ACIDS.#7/HERBAL COMB.#125/CHOLINE BIT MDC Brand Name ACARBOSE ICN-TOLAM ACACROSE ICN-TOLAM ACTOPLUS MET ACTOPLUS MET ACTOPLUS MET INVOKAMET ACTOS JANUMET INVOKAMET APPFORNIND JUVISYNC AVANDAMET AVANDAMET AVANDAMET AVANDAWI AVANDAWI AVANDAWI CHLORABETIC 250 METFORMIN HCL CHLORABETIC 250 METFORMIN HCL ER DIABIESE DIABIESE DIABIESE DIABIESE DIABIESE NATEGLINDE DIBABTAO DUSTACT ONGLYZA DYMELOR FORTAMET ORINASE GLIMEPRIDE GLIPZIDE KL GLIPZIDE KL GLIPZIDE KL GLIPZIDE KL GLIPZIDE KL GLIPZIDE KL GLIPZIDE KR GLIUCOPHAGE PRECOSE GLIUCOPHAGE | LINAGLIPTIN | SITAGLIPTIN PHOSPHATE |
| METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB#125/CHOUNE BIT NDC Brand Name ACARBOSE ICN-TOLBUT MET ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTORIUS MET NI ANUMET NI ACTORIUS MET NI ANUMET NI ANUMET NI ACTORIUS MET NI APPEORMIN IENTADUETO IPUTISTNC AVANDARY AVANDARY AVANDARY AVANDIA CHURRABETIC 250 METFORMIN HCL CHURRABETIC 250 METFORMIN HCL CHURRABETIC 250 METFORMIN HCL CHURRABETIC 250 ACTORIUS METFORMIN HCL CHURRABETIC 250 CHURLABETIC MICRONASE DIBBITIC ONGLYZA | LINAGLIPTIN/METFORMIN HCL | SITAGLIPTIN PHOSPHATE/METFORMIN HCL |
| MDC Brand Name ACARBOSE ACETOHEXAMIDE ACAROSE ICN-TOLAM ACETOHEXAMIDE INSULASE ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTORIUS MET NA AMARYL APPEORMIN IENTADUETO JANUMET NA APPEORMIN-D JUVIS'NTC AVANDAMET AVANDAMET AVANDAMET AVANDAMET AVANDAMET AVANDARYL AVANDARY AVANDARYL AVANDARY AVANDARYL AVANDA | METFORMIN HCL | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| MDC Brand Name ACARBOSE ACETOHEXAMIDE ACAROSE ICN-TOLAM ACETOHEXAMIDE INSULASE ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTOPIUS MET ACTORIUS MET NA AMARYL APPEORMIN IENTADUETO JANUMET NA APPEORMIN-D JUVIS'NTC AVANDAMET AVANDAMET AVANDAMET AVANDAMET AVANDAMET AVANDARYL AVANDARY AVANDARYL AVANDARY AVANDARYL AVANDA | METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOLINE | TOLAZAMIDE |
| ACARBOSE ACTOPLUS MET INSULASE INSULASE ACTOPLUS MET XR ACTOPLUS MET XR JANUMET XR ACTOPLUS MET XR JANUMET XR ACTOPLUS MET XR JANUMET XR AMARYL APPEORMIN JENITADUETO JUVISYNC AVANDAMET KAZANO AVANDAMET KAZANO AVANDAMET KAZANO AVANDAMET KAZANO AVANDAMET KAZANO AVANDARYL AVANDIA CHLORABETIC 250 METFORMIN HCL METFORMIN HCL METFORMIN | | TOLBUTAMIDE |
| ACTOPLUS MET INVOKAMET ACTOPUS MET XR ACTOPUS MET XR JANUMET ACTOS JANUMET ACTOS JANUMET XR ACTOPUS MET XR ACTOPUS MET XR ACTOS JANUMET XR AMARYL APPFORMIN JENTADUETO APPFORMINO JUVISYNC APANDAMET KAZANO AVANDAMET KAZANO AVANDAMET ACTOR AVANDAMET AVANDAMET AVANDAMET ACTOR AVANDAMET AVANDAMET AVA | NDC Brand Name | |
| ACTOPLUS MET XR JANUMET ACTOPUS MET XR JANUMET R ACTOS JANUMET XR AMARYL JANUVIA APPFORMIN JANUVIA APPFORMIND JUVISYNC AVANDAMET KAZANO AVANDAMET KAZANO AVANDAMYL KOMBIGLYZE XR AVANDIA METFORMIN HCL CHLORABETIC 250 M | ACARBOSE | ICN-TOLAM |
| ACTOPLUS MET XR ACTOS JANUMET ACTOS JANUMET XR AMARYL APPFORMIN APPFORMIN JENTADUETO APPFORMIN-D JUVISYNC KAZANO AVANDAMET KAZANO AVANDAMET AVANDARYL AVANDARYL KOMBIGLYZE XR AVANDIA METAGLIP CHLORABETIC 250 METFORMIN HCL CHLORAPROPAMIDE MICRONASE DIABITESE NATEGLINDE JIBAITROL DIBAITROL DIBATROL DIBATROL DIBATROL DIBATROL DIBATROL ORNETIC GUNPZIDE GUIPZIDE GUIPZIDE GUIPZIDE GUIPZIDE GUIPZIDE GUIPZIDE RR GUIPZIDE XL GUIPZIDE KR GUIPZIDE METFORMIN GUIPZIDE-METFORMIN GUILAZONBETIC GUIPZIDE METFORMIN GUILAZONBETIC GUIPZIDE METFORMIN GUILAZONBETIC GUIPZIDE RR GUIPZIDE RE GUIPZIDE RR GUIPZIDE RE GUIP | ACETOHEXAMIDE | INSULASE |
| ACTOS JANUMET XR AMARYL JANUVIA APPEORMIN APPEORMIN APPEORMIND APPEORMIND APPEORMIND AVANDAMET KAZANO AVANDAMET KAZANO AVANDARYL KOMBIGIYZE XR AVANDIA CHLORABETIC 250 METFORMIN HCL CHLORRPROPAMIDE METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABITASE NATEGUNIDE DIBABTA NESINA DIABITACI NESINA DUETACT ONGIYZA DYMELOR FORTAMET ORINASE GUMEPIRIDE OSENI GUIPZIDE GUIPZIDE X GUIPZIDE R GUIPZIDE AMETFORMIN GULCAMIDE GUIPZIDE METFORMIN GULCAMIDE GUIPZIDE METFORMIN GULCAMIDE GUICAMIDE GUICOPHAGE R GUICOPHAGE R GUICOTROL XI RONASE GUIVENDE GUINATIA GUIVANIC GUIVATIA GUIVANIC GUIVANIC GUIVANIC GUIVANIC GUIVANIC GUIVANIC GUIVANIC GUICAMIDE GUICOTROL GUICOTROL GUIVANIC GUIV | ACTOPLUS MET | INVOKAMET |
| AMARYL APPFORMIN JENTADUETO APPFORMIN-D JUVISYNC AVANDAMET KAZANO AVANDARYT KOMBIGLYZE XR AVANDIA WETAGUP CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE MICROMASE DIABITA DIBATROL DIBATROL DIBATROL DIBATROL ONGIYZA DYMELOR FORTAMET GUILPIZIDE GUIPZIDE ER GUIPZIDE ER PIOGLITAZONE-GUIMEPIRIDE GUIPZIDE XL GUIPZIDE XL GUIPZIDE METFORMIN GULCOPHAGE GLUCOPHAGE GLUCOPHAGE GLUCOPHAGE GLUCOTROL KL GUINETA STARIK GLUCOTROL KL GUINETA GLUCOTROL KL GUINETA GLUCOTROL GLUCOTROL GLUCOTROL GLUCOTROL GLUCOPHAGE GLUCOPHA | ACTOPLUS MET XR | JANUMET |
| APPFORMIND APPFORMIND APPFORMIND APPFORMIND AVANDAMET KAZANO AVANDAMET KAZANO AVANDARYL KOMBIGLYZE XR AVANDIA METAGLIP CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABITA MICRONASE DIABITA MICRONASE DIBAITAOL NESINA DUETACT ONGLYZA DYMELOR ORIBETIC FORTAMET GUIMEPIRIDE GUIPZIDE PIOGUITAZONE HCL GUIPZIDE ER GUIPZIDE RT GUIPZIDE AUTOMAGE BUILOCHAGE GUIVENDEMETFORMIN GUIVENDEMET GUIVE | ACTOS | JANUMET XR |
| APPFORMIN-D AVANDAMET KAZANO AVANDAMET KAZANO AVANDAYL KOMBIGIVZE XR AVANDIA CHIORABETIC 250 METFORMIN HCL CHIORABETIC 250 METFORMIN HCL ER DIABETA MICRONASE DIABIRSE MATEGINIDE DIBATROL DUETACT ONGLYZA DYMELOR OFFICE GUIPZIDE GUIPZIDE GUIPZIDE XL GUIPZIDE XL GUIPZIDE XL GUIPZIDE XL GUIPZIDE METFORMIN GUICOTROL GUIPZIDE MICRONIZED GUIPZIDE MICRONIZED GUIVANDE GUIPZIDE MICRONIZED GUIPZIDE MICRONIZED GUIVANDE GUIPZIDE MICRONIZED GUIPZIAMIDE GUIP | AMARYL | JANUVIA |
| AVANDAMET AVANDARYL KAZANO KAZANO KAYANDIA METAGUP CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABIESA MICRONASE DIABINESE NATEGUNIDE DIBATROL DUFFACT ONGLYZA DYMELOR FORTAMET GUMEPRIDE GUPZIDE ER GUPZIDE ER GUPZIDE ER GUIPZIDE-METFORMIN GULCOPHAGE GLUCOPHAGE GLUCOTROL GLUCOTROL GLUCOTROL GLUCOTROL GLUCOTROL GLUCOMACE GLUCOTROL GLUCOMACE GLUCOTROL GLUCOMACE GLUCOTROL GLUCOMACE GLU | APPFORMIN | JENTADUETO |
| AVANDIAYL AVANDIA AVANDIA METAGLIP CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABINESE MATEGLINIDE DIBATROL DUETACT ONGLYZA DYMELOR ORINASE GLIPIZIDE GLIPIZIDE GLIPIZIDE GLIPIZIDE R GLIPIZIDE XL GLIPIZ | APPFORMIN-D | JUVISYNC |
| AVANDIA METAGLIP CHLORABETIC 250 METFORMIN HCL CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABINESE MATEGLINIDE DIBATROL NESINA DUFTACT ONGLYZA DYMELOR ORIBETIC GUIMEPRIDE GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE PIOGLITAZONE-GLIMEPRIDE GLIPIZIDE NETFORMIN PRANDIMET GLUCOPHAGE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPORTED GLUCOTROL RICHARD GLUCOTROL RICHARD GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE SK-TOLBUTAMIDE GLYNASE TOLAMIDE GLYNASE TRADJETNAMI GLYNASE GLYNASE TRADJETNAMI GLYNASE GLYNASE TRADJETNAMI GLYCONICA METAGLIPIC M | AVANDAMET | KAZANO |
| CHLORABETIC 250 METFORMIN HCL CHLORPROPAMIDE METFORMIN HCL ER DIABETA MICRONASE DIABINESE MATEGLINIDE DIBATROL NESINA DUETACT ONGLYZA DYMELOR FORTAMET ORINASE GLIMEPIRIDE GLIPIZIDE GLIPIZIDE R GLIPIZIDE R GLIPIZIDE XL GLIPIZIDE XL GLIPIZIDE METFORMIN GLICAMIDE GLUCOPHAGE GLUCOPHAGE GLUCOPHAGE GLUCOPHAGE GLUCOTROL GLUCOTROL GLICOTROL G | AVANDARYL | KOMBIGLYZE XR |
| CHLORPROPAMIDE DIABETA DIABINESE DIABINESE DIBATROL DIBATROL DUETACT DYMELOR ORIBETIC GUIPIZIDE GLIPIZIDE ER GLIPIZIDE ARRADIME GLUCOPHAGE GLUCOPHAGE GLUCOTROL GLUCOTROL GLUCOTROL GLUCOTROL GLUCOTROL GLIPIZIDE GLYBURDE GLYBURD GLYBURD GLYBURD GRAND GLYBURD GLYBURD GRAND | AVANDIA | METAGLIP |
| DIABETA MICRONASE DIABINESE NATEGLINIDE DIBATROL NESINA DUETACT ONGLYZA DYMELOR ORIBETIC FORTAMET ORINASE GLIMEPIRIDE OSENI GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE RIPIZIDE PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIME GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOVANCE SK-TOLBUTAMIDE GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAMIDE GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYCON TOLBUTAMISE GLYCON GLYCON GLYCON GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON GLYCON GLYCON GLYCON GLYCON TOLBUTAMIDE GLYCON TOLBUTAMIDE GLYCON GRACH | CHLORABETIC 250 | METFORMIN HCL |
| DIABINESE DIBATROL DIBATROL NESINA DUETACT ONGLYZA DYMELOR ORIBETIC FORTAMET ORINASE GLIMEPIRIDE OSENI GLIPIZIDE GIPIZIDE R GIPIZIDE R GIPIZIDE R GUIPIZIDE R GUICONAGE GUIPIZIDE R GRANDIN GRANDIMET GLUCAMIDE FRANDIME GLUCOPHAGE PRANDIN GLUCOPHAGE REPAGLINIDE GLUCOPHAGE R GUCOPHAGE R GUCOPHAGE R GUCOYNOL RIOMET GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLYBURIDE GLYBURIDE MICRONIZED TOLAMIDE GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYCON TOLINASE GLYCON GLYNASE TRADJENTA | CHLORPROPAMIDE | METFORMIN HCL ER |
| DIBATROL DUETACT DUETACT DOMGLYZA DYMELOR ORIBETIC FORTAMET ORINASE GIMEPIRIDE OSENI GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE R PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCOPHAGE PRANDIN GLUCOPHAGE RUCOPHAGE RUCOPHAGE RUCOTROL RUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL ROMASE GLUCOTROL ROMASE GLUCOTROL GLUCOTROL GLUCOTROL SCHOOL GLUCOTROL GLUCOTRO | DIABETA | MICRONASE |
| DUETACT ONGLYZA DYMELOR ORIBETIC FORTAMET ORINASE GLIMEPIRIDE OSENI GUPIZIDE PIOGLITAZONE HCL GUPIZIDE ER PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE MICRONIZED TOLAMIDE GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYCON TOLBUTAMIDE GLYCON TOLINASE GLYCON TOLINASE GLYCON | DIABINESE | NATEGLINIDE |
| DYMELOR ORIBETIC FORTAMET ORINASE GLIMEPIRIDE OSENI GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE RIPIGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN GLIPIZIDE-METFORMIN GLICOPHAGE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL GLUCOTROL GLUCOTROL RIOMET GLUCOVANCE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYCRON TOLINASE | DIBATROL | NESINA |
| FORTAMET ORINASE GLIMEPIRIDE OSENI GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE ER PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIME GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE GLUMETZA STARLIX GLYBURIDE GLYBURIDE GLYBURIDE MICRONIZED GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYCRON TOLBUTAMIDE GLYCRON TOLBUTAMIDE GLYCRON TOLBUTAMIDE GLYCRON TOLINASE GLYCRON TOLINASE GLYCRON TOLINASE | DUETACT | ONGLYZA |
| GLIMEPIRIDE GLIPIZIDE GLIPIZIDE GLIPIZIDE ER GLIPIZIDE ER GLIPIZIDE XL PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE GLYBURIDE GLY | DYMELOR | ORIBETIC |
| GLIPIZIDE PIOGLITAZONE HCL GLIPIZIDE ER PIOGLITAZONE-GLIMEPIRIDE GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE SK-TOLBUTAMIDE GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | FORTAMET | ORINASE |
| GLIPIZIDE ER GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE GLUCOVANCE GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYCRON TOLBUTAMIDE GLYBURIDE GLYBURI | GLIMEPIRIDE | OSENI |
| GLIPIZIDE XL PIOGLITAZONE-METFORMIN GLIPIZIDE-METFORMIN PRANDIMET GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUCOVANCE SK-TOLBUTAMIDE GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDES GLYBURID | GLIPIZIDE | PIOGLITAZONE HCL |
| GLIPIZIDE-METFORMIN GLUCAMIDE GLUCOPHAGE GLUCOPHAGE GLUCOPHAGE PRECOSE GLUCOPHAGE XR GLUCOTROL GLUCOTROL GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE GLUCOVANCE GLUCOVANCE GLUMETZA GLYBURIDE GLYBURIDE GLYBURIDE GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE G | GLIPIZIDE ER | PIOGLITAZONE-GLIMEPIRIDE |
| GLUCAMIDE PRANDIN GLUCOPHAGE PRECOSE GLUCOPHAGE REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL ROMASE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDES GLYBURIDE TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDES GLYBURIDES GLYNASE TRADJENTA | GLIPIZIDE XL | PIOGLITAZONE-METFORMIN |
| GLUCOPHAGE PRECOSE GLUCOPHAGE XR REPAGLINIDE GLUCOTROL RIOMET GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYRON TOLINASE GLYNASE TRADJENTA | GLIPIZIDE-METFORMIN | PRANDIMET |
| GLUCOPHAGE XR GLUCOTROL GLUCOTROL XL GLUCOTROL XL RONASE GLUCOVANCE GLUCOVANCE GLUMETZA GLYBURIDE GLYBURIDE GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCAMIDE | PRANDIN |
| GLUCOTROL GLUCOTROL XL RONASE GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE GLYBURIDE GLYBURIDE TOLAMIDE GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOPHAGE | PRECOSE |
| GLUCOTROL XL GLUCOVANCE GLUCOVANCE GLUMETZA GLYBURIDE GLYBURIDE GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYBURIDE-METFORMIN HCL GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOPHAGE XR | REPAGLINIDE |
| GLUCOVANCE SK-TOLBUTAMIDE GLUMETZA STARLIX GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOTROL | RIOMET |
| GLUMETZA STARLIX GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOTROL XL | RONASE |
| GLYBURIDE TOLAMIDE GLYBURIDE MICRONIZED TOLAZAMIDE GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLUCOVANCE | SK-TOLBUTAMIDE |
| GLYBURIDE MICRONIZED GLYBURIDE-METFORMIN HCL GLYCRON TOLINASE GLYNASE TRADJENTA | GLUMETZA | STARLIX |
| GLYBURIDE-METFORMIN HCL TOLBUTAMIDE GLYCRON TOLINASE GLYNASE TRADJENTA | GLYBURIDE | TOLAMIDE |
| GLYCRON TOLINASE GLYNASE TRADJENTA | GLYBURIDE MICRONIZED | TOLAZAMIDE |
| GLYCRON TOLINASE GLYNASE TRADJENTA | GLYBURIDE-METFORMIN HCL | TOLBUTAMIDE |
| | GLYCRON | TOLINASE |
| GLYSFT | GLYNASE | TRADJENTA |
| OLIGET | GLYSET | |

### Insulin


| EXUBERA COMBINATION PACK 12 | INSULIN NPH BEEF |
|-----------------------------|--------------------------------|
| EXUBERA COMBINATION PACK 15 | INSULIN NPH PURIFIED PORK |
| EXUBERA KIT | INSULIN R PORK PURIFIED |
| EXUBERA PATIENT PACK | INSULIN R PURIFIED PORK |
| HUMALOG | INSULIN REGULAR PORK |
| HUMALOG MIX 50-50 | INSULIN REGULAR PURIFIED PORK |
| HUMALOG MIX 50/50 | ISOPHANE INSULIN BEEF |
| HUMALOG MIX 75-25 | ISOPHANE PURIFIED BEEF INSULIN |
| HUMULIN 50-50 | LANTUS |
| HUMULIN 70-30 | LANTUS SOLOSTAR |
| HUMULIN 70/30 | LENTE INSULIN BEEF |
| HUMULIN 70/30 KWIKPEN | LEVEMIR |
| HUMULIN BR | LEVEMIR FLEXPEN |
| HUMULIN L | LEVEMIR FLEXTOUCH |
| HUMULIN N | MONOTARD HUMAN LENTE |
| HUMULIN N KWIKPEN | NOVOLIN 70-30 |
| HUMULIN R | NOVOLIN 70-30 INNOLET |
| HUMULIN U | NOVOLIN 70/30 |
| ILETIN I LENTE | NOVOLIN L |
| ILETIN I NPH | NOVOLIN N |
| ILETIN I REGULAR | NOVOLIN N INNOLET |
| ILETIN I SEMILENTE | NOVOLIN R |
| ILETIN I ULTRALENTE | NOVOLOG |
| ILETIN II LENTE(BEEF) | NOVOLOG FLEXPEN |
| ILETIN II LENTE(PORK) | NOVOLOG MIX 70-30 |
| ILETIN II NPH(BEEF) | NOVOLOG MIX 70-30 FLEXPEN |
| ILETIN II NPH(PORK) | PROTAMINE ZINC INSULIN BEEF |
| ILETIN II REGULAR(BEEF) | PURIFIED BEEF INSULIN ZINC |
| ILETIN II REGULAR(PORK) | PURIFIED PORK INSULIN |
| ILETIN II REGULAR(PORK)CONC | VELOSULIN HUMAN |
| INSULATARD HUMAN N | VELOSULIN HUMAN BR |
| INSULATARD N | VELOSULIN HUMAN R |
| INSULATARD NPH HUMAN | VELOSULIN R |
| INSULIN L PURIFIED PORK | ZINC |
| INSULIN LENTE BEEF | |

#### Antidepressants

| HCPCS | |
|---|---|
| | T |
| J1320 NDC Generic Name | |
| | IN ALIDDA NAUNIS LLCI |
| AMITRIPTYLINE HCL | IMIPRAMINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE PAMOATE |
| AMOXAPINE | ISOCARBOXAZID |
| BUPROPION HBR | LEVOMILNACIPRAN HYDROCHLORIDE |
| BUPROPION HCL | MAPROTILINE HCL |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB15 | MIRTAZAPINE |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB16 | NEFAZODONE HCL |
| CITALOPRAM HYDROBROMIDE | NORTRIPTYLINE HCL |
| CLOMIPRAMINE HCL | OLANZAPINE/FLUOXETINE HCL |
| DESIPRAMINE HCL | PAROXETINE HCL |
| DESVENLAFAXINE | PAROXETINE MESYLATE |
| DESVENLAFAXINE FUMARATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| DESVENLAFAXINE SUCCINATE | PHENELZINE SULFATE |
| DOXEPIN HCL | PROTRIPTYLINE HCL |
| DULOXETINE HCL | SERTRALINE HCL |
| ESCITALOPRAM OXALATE | TRAZODONE HCL |
| FLUOXETINE | TRAZODONE HCL/DIETARY SUPPLEMENT,MISC.COMBO8 |
| FLUOXETINE HCL | TRIMIPRAMINE MALEATE |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC COMB17 | VENLAFAXINE HCL |
| FLUOXETINE HCL/DIETARY SUPPLEMENT, MISC. COMBO8 | VILAZODONE HYDROCHLORIDE |
| FLUVOXAMINE MALEATE | VORTIOXETINE HYDROBROMIDE |
| NDC Brand Name | |
| ADAPIN | LIMBITROL DS |
| AMITID | LUDIOMIL |
| AMITRIPTYLINE HCL | LUVOX |
| AMITRIPTYLINE W/PERPHENAZINE | LUVOX CR |
| AMITRIPTYLINE-CHLORDIAZEPOXIDE | MAPROTILINE HCL |
| AMITRIPTYLINE-PERPHENAZINE | MARPLAN |

| AMITRIPTYLINE/CHLORDIAZEPOXIDE | MIRTAZAPINE |
|---|---|
| AMOXAPINE | MIRTAZAPINE ANHYDROUS |
| ANAFRANIL | NARDIL |
| APLENZIN | NEFAZODONE HCL |
| APPBUTAMONE | NORFRANIL |
| APPBUTAMONE-D | NORPRAMIN |
| ASENDIN | NORTRIPTYLINE HCL |
| AVENTYL HCL | OLANZAPINE-FLUOXETINE HCL |
| BRINTELLIX | OLEPTRO ER |
| BRISDELLE | PAMELOR |
| BUDEPRION SR | PAROXETINE HCL |
| BUDEPRION XL | PAXIL |
| BUPROBAN | PAXIL CR |
| BUPROPION HCL | PER-TRIP |
| BUPROPION HCL ER | PERPHENAZINE-AMITRIPTYLINE |
| BUPROPION HCL SR | PEXEVA |
| BUPROPION XL | PHENELZINE SULFATE |
| CELEXA | PRISTIQ ER |
| CHLORDIAZEPOXIDE-AMITRIPTYLINE | PROTRIPTYLINE HCL |
| CITALOPRAM | PROZAC |
| CITALOPRAM HBR | PROZAC WEEKLY |
| CLOMIPRAMINE HCL | PRUDOXIN |
| CYMBALTA | Q.E.L |
| DECONIL | RAPIFLUX |
| DESIPRAMINE HCL | RE-LIVE |
| DESVENLAFAXINE ER | REMERON |
| DESVENDATAXINE EIX DESVENDATAXINE FUMARATE ER | SARAFEM |
| DESYREL | SELFEMRA |
| DOXEPIN HCL | SENTROXATINE |
| DULOXETINE HCL | SERTRALINE HCL |
| E-VILL 10 | SERZONE |
| L VILL 10 | SEINZOINE |
| E-VIII 100 | SILENOR |
| E-VILL 100 | SILENOR<br>SINFOLIAN |
| E-VILL 25 | SINEQUAN |
| E-VILL 25<br>E-VILL 50 | SINEQUAN<br>SK-AMITRIPTYLINE |
| E-VILL 25 E-VILL 50 E-VILL 75 | SINEQUAN<br>SK-AMITRIPTYLINE<br>SK-PRAMINE |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-4 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE HCL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-25 TRIAVIL 4-50 |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE FLUVOXAMINE MALEATE ER | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VIIBRYD |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VIBRYD VIVACTIL |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VELBUTRIN |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5-2 TRIAVIL 25-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL VENLAFAXINE HCL WELLBUTRIN WELLBUTRIN |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5 TRIAVIL 2-5-4 TRIAVIL 2-5-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXAMINE MALEATE FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL KHEDEZLA | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 25-2 TRIAVIL 25-2 TRIAVIL 25-6 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN SR WELLBUTRIN XL ZOLOFT |
| E-VILL 25 E-VILL 50 E-VILL 75 EFFEXOR EFFEXOR XR ELAVIL EMITRIP ENDEP ENOVIL ESCITALOPRAM OXALATE ETNOFRIL ETRAFON 2-10 ETRAFON 2-25 ETRAFON A 4-10 ETRAFON FORTE 4-25 FETZIMA FLUOXETINE DR FLUOXETINE DR FLUOXETINE HCL FLUVOXAMINE MALEATE ER FORFIVO XL GABOXETINE IMAVATE IMIPRAMINE HCL IMIPRAMINE PAMOATE JANIMINE KENVIL | SINEQUAN SK-AMITRIPTYLINE SK-PRAMINE STABANIL SURMONTIL SYMBYAX TOFRANIL TOFRANIL-PM TRAZAMINE TRAZODONE HCL TRIAVIL 10-2 TRIAVIL 2-10 TRIAVIL 2-25 TRIAVIL 2-5 TRIAVIL 2-5-4 TRIAVIL 2-5-4 TRIAVIL 4-10 TRIAVIL 4-10 TRIAVIL 4-25 TRIAVIL 4-50 TRIMIPRAMINE MALEATE VANATRIP VENLAFAXINE HCL VENLAFAXINE HCL ER VIIBRYD VIVACTIL WELLBUTRIN WELLBUTRIN SR |

## Appendix A Comorbid conditions

**Atrial Fibrillation** 

125110

125111

125118

125119

41070

41071

4108

41080


Coronary Artery Disease ICD10 Dx ICD9 Dx LongDesICD10 LongDesICD9 1200 ACUTE MYOCARDIAL INFARCTION 410 Unstable angina 1201 4100 ACUTE MYOCARDIAL INFARCTION OF ANTEROLATERAL WALL Angina pectoris with documented spasm 1208 41000 ACUTE MYOCARDIAL INFARCTION OF ANTEROLATERAL WALL Other forms of angina pectoris EPISODE OF CARE UNSPECIFIED 1209 41001 Angina pectoris, unspecified ACUTE MYOCARDIAL INFARCTION OF ANTEROLATERAL WALL INITIAL EPISODE OF CARE 12101 4101 ST elevation (STEMI) myocardial infarction involving left ACUTE MYOCARDIAL INFARCTION OF OTHER ANTERIOR main coronary artery WALL 12102 41010 ST elevation (STEMI) myocardial infarction involving left ACUTE MYOCARDIAL INFARCTION OF OTHER ANTERIOR WALL EPISODE OF CARE UNSPECIFIED anterior descending coronary artery 12109 41011 ST elevation (STEMI) myocardial infarction involving other ACUTE MYOCARDIAL INFARCTION OF OTHER ANTERIOR WALL INITIAL EPISODE OF CARE coronary artery of anterior wall 12111 4102 ST elevation (STEMI) myocardial infarction involving right ACUTE MYOCARDIAL INFARCTION OF INFEROLATERAL WALL coronary artery 12119 41020 ST elevation (STEMI) myocardial infarction involving other ACUTE MYOCARDIAL INFARCTION OF INFEROLATERAL WALL coronary artery of inferior wall EPISODE OF CARE UNSPECIFIED 12121 41021 ST elevation (STEMI) myocardial infarction involving left ACUTE MYOCARDIAL INFARCTION OF INFEROLATERAL WALL NITIAL EPISODE OF CARE circumflex coronary artery 12129 4103 ST elevation (STEMI) myocardial infarction involving other ACUTE MYOCARDIAL INFARCTION OF INFEROPOSTERIOR sites ACUTE MYOCARDIAL INFARCTION OF INFEROPOSTERIOR 41030 1213 ST elevation (STEMI) myocardial infarction of unspecified WALL EPISODE OF CARE UNSPECIFIED 1214 41031 Non-ST elevation (NSTEMI) myocardial infarction ACUTE MYOCARDIAL INFARCTION OF INFEROPOSTERIOR WALL INITIAL EPISODE OF CARE 1220 4104 Subsequent ST elevation (STEMI) myocardial infarction of ACUTE MYOCARDIAL INFARCTION OF OTHER INFERIOR WALL anterior wall 1221 41040 ACUTE MYOCARDIAL INFARCTION OF OTHER INFERIOR WALL Subsequent ST elevation (STEMI) myocardial infarction of EPISODE OF CARE UNSPECIFIED inferior wall 1222 41041 Subsequent non-ST elevation (NSTEMI) myocardial infarction ACUTE MYOCARDIAL INFARCTION OF OTHER INFERIOR WALL NITIAL EPISODE OF CARE 1228 4105 ACUTE MYOCARDIAL INFARCTION OF OTHER LATERAL WALL Subsequent ST elevation (STEMI) myocardial infarction of other sites 1229 41050 Subsequent ST elevation (STEMI) myocardial infarction of ACUTE MYOCARDIAL INFARCTION OF OTHER LATERAL WALL unspecified site EPISODE OF CARE UNSPECIFIED 1240 41051 Acute coronary thrombosis not resulting in myocardial ACUTE MYOCARDIAL INFARCTION OF OTHER LATERAL WALL infarction INITIAL EPISODE OF CARE 1241 4106 TRUE POSTERIOR WALL INFARCTION Dressler's syndrome Other forms of acute ischemic heart disease TRUE POSTERIOR WALL INFARCTION EPISODE OF CARE 1248 41060 UNSPECIFIED 41061 1249 TRUE POSTERIOR WALL INFARCTION INITIAL EPISODE OF Acute ischemic heart disease, unspecified 12510 4107 Atherosclerotic heart disease of native coronary artery SUBENDOCARDIAL INFARCTION without angina pectoris

Atherosclerotic heart disease of native coronary artery with

unstable angina pectoris

other forms of angina pectoris

unspecified angina pectoris

angina pectoris with documented spasm

SUBENDOCARDIAL INFARCTION EPISODE OF CARE

SUBENDOCARDIAL INFARCTION INITIAL EPISODE OF CARE

ACUTE MYOCARDIAL INFARCTION OF OTHER SPECIFIED

ACUTE MYOCARDIAL INFARCTION OF OTHER SPECIFIED

SITES EPISODE OF CARE UNSPECIFIED

JNSPECIFIED


## Appendix A Comorbid conditions


**Heart Failure** 


| Dilation of Loft Internal Corptial Autory, Differentian with | T |
|---|---|
| •• | |
| , , | |
| , | |
| · · | |
| , | |
| · | |
| 1 1 11 | |
| • | |
| • | |
| · | |
| •• | |
| • | |
| Dilation of Left Internal Carotid Artery with Three | |
| Intraluminal Devices, Open Approach- | |
| Dilation of Left Internal Carotid Artery, Bifurcation, with | |
| Four or More Intraluminal Devices, Open Approach— | |
| Dilation of Left Internal Carotid Artery with Four or More | |
| Intraluminal Devices, Open Approach– | |
| Dilation of Left Internal Carotid Artery, Bifurcation, Open | |
| 2: | |
| , , , | |
| · | |
| _ · | |
| Dilation of Right External Carotid Artery, Biflircation, with | |
| Dilation of Right External Carotid Artery, Bifurcation, with<br>Three Drug-eluting Intraluminal Devices, Open Approach- | |
| | Intraluminal Devices, Open Approach— Dilation of Left Internal Carotid Artery, Bifurcation, with Four or More Intraluminal Devices, Open Approach— Dilation of Left Internal Carotid Artery with Four or More Intraluminal Devices, Open Approach— Dilation of Left Internal Carotid Artery, Bifurcation, Open Approach— Dilation of Left Internal Carotid Artery, Bifurcation, Open Approach— Dilation of Right External Carotid Artery, Bifurcation, with Drug-eluting Intraluminal Device, Open Approach— Dilation of Right External Carotid Artery with Drug-eluting Intraluminal Device, Open Approach Dilation of Right External Carotid Artery with Drug-eluting Intraluminal Device, Open Approach— Dilation of Right External Carotid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Open Approach— Dilation of Right External Carotid Artery with Two Drug-eluting Intraluminal Devices, Open Approach— Dilation of Right External Carotid Artery with Two Drug-eluting Intraluminal Devices, Open Approach—eluting Intraluminal Devices, Open Approach— |


| Dilation of Left Vertebral Artery with Drug-eluting | |
|---|---|
| - | |
| - | |
| , | |
| 1 11 | |
| · | |
| , | |
| · | |
| , | |
| 1 11 | |
| · | |
| i ii | |
| · | |
| • | |
| i ii | |
| ** | |
| Approach- | |
| Dilation of Left Vertebral Artery, Open Approach- | |
| Dilation of Face Artery, Bifurcation, with Drug-eluting | |
| Intraluminal Device, Open Approach-eluting Intraluminal | |
| Device, Open Approach | |
| Dilation of Face Artery with Drug-eluting Intraluminal | |
| Device, Open Approach-eluting Intraluminal Device, Open | |
| Approach | |
| Dilation of Face Artery, Bifurcation, with Two Drug-eluting | |
| Intraluminal Devices, Open Approach-eluting Intraluminal | |
| Devices, Open Approach | |
| Dilation of Face Artery with Two Drug-eluting Intraluminal | |
| Devices, Open Approach-eluting Intraluminal Devices, Open | |
| Approach | |
| Dilation of Face Artery, Bifurcation, with Three Drug-eluting | |
| Intraluminal Devices, Open Approach-eluting Intraluminal | |
| Devices, Open Approach | |
| Dilation of Face Artery with Three Drug-eluting Intraluminal | |
| Devices, Open Approach-eluting Intraluminal Devices, Open | |
| · | |
| | Intraluminal Device, Open Approach-eluting Intraluminal Device, Open Approach Dilation of Left Vertebral Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Open Approach-eluting Intraluminal Devices, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, with Intraluminal Device, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, with Intraluminal Device, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, with Two Intraluminal Devices, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, with Tree Intraluminal Devices, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, with Tree Intraluminal Devices, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, with Four or More Intraluminal Devices, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, with Four or More Intraluminal Devices, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, Open Approach-Dilation of Left Vertebral Artery, Bifurcation, With Four or More Intraluminal Devices, Open Approach-Dilation of Face Artery, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach-Dilation of Face Artery, Bifurcation, with Drug-eluting Intraluminal Devices, Open Approach-Dilation of Face |


| Dilation of Calcula Autom. Differentian with Introduction | |
|---|---|
| • | |
| , | |
| , | |
| Dilation of Splenic Artery, Bifurcation, with Three | |
| Intraluminal Devices, Open Approach | |
| Dilation of Splenic Artery with Three Intraluminal Devices, | |
| Open Approach | |
| Dilation of Splenic Artery, Bifurcation, with Four or More | |
| Intraluminal Devices, Open Approach- | |
| Dilation of Splenic Artery with Four or More Intraluminal | |
| Devices, Open Approach | |
| Dilation of Splenic Artery, Bifurcation, Open Approach— | |
| Dilation of Splenic Artery, Open Approach- | |
| Dilation of Splenic Artery with Drug-eluting Intraluminal | |
| , , , , | |
| , | |
| . , | |
| - | |
| , , | |
| , | |
| * | |
| · | |
| • | |
| ·· | |
| · | |
| • • • | |
| • | |
| ··· | |
| * | |
| , | |
| ** | |
| Approach- | |
| Dilation of Splenic Artery, Percutaneous Approach- | |
| Dilation of Splenic Artery with Drug-eluting Intraluminal | |
| Device, Percutaneous Endoscopic Approach-eluting | |
| Intraluminal Device, Percutaneous Endoscopic Approach | |
| Dilation of Splenic Artery with Two Drug-eluting | |
| Intraluminal Devices, Percutaneous Endoscopic Approach- | |
| eluting Intraluminal Devices, Percutaneous Endoscopic | |
| Approach | |
| Dilation of Splenic Artery with Three Drug-eluting | |
| Intraluminal Devices, Percutaneous Endoscopic Approach- | |
| eluting Intraluminal Devices, Percutaneous Endoscopic | |
| | Dilation of Splenic Artery with Three Intraluminal Devices, Open Approach— Dilation of Splenic Artery, Bifurcation, with Four or More Intraluminal Devices, Open Approach— Dilation of Splenic Artery with Four or More Intraluminal Devices, Open Approach— Dilation of Splenic Artery, Bifurcation, Open Approach— Dilation of Splenic Artery, Open Approach— Dilation of Splenic Artery with Drug-eluting Intraluminal Device, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach— Dilation of Splenic Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Splenic Artery with Intraluminal Device, Percutaneous Approach— Dilation of Splenic Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery, Bifurcation, Percutaneous Approach— Dilation of Splenic Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Splenic Artery with Four or More Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Splenic Artery with Torug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Splenic Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Splenic |


| Dilation of Left Femoral Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach-oated Balloon, Percutaneous Approach-Oated Balloon, Percutaneous Approach-Oated Balloon, Percutaneous Approach-Oated Balloon, Percutaneous Approach-Obliation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach-Obliation of Left Femoral Artery, Bifurcation, with Two Intraluminal Device, Percutaneous Approach-Obliation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach-Obliation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach-Obliation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach-Obliation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach-Obliation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach-Obliation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach-Obliation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach-Obliation of Left Femoral Artery, Bifurcation, With Drug-eluting Intraluminal Device, Using Drug-Coated Balloon, Percutaneous Approach-Obliation of Left Femoral Art |
|---|
| Approach-eluting intraluminal Devices, Percutaneous Approach Dilation of teft Femoral Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of teft Femoral Artery with Intraluminal Device, using Drug-Coated Balloon, Percutaneous Approach Dilation of teft Femoral Artery, Bifurcation, with Intraluminal Device, using Drug-Coated Balloon, Percutaneous Approach Dilation of teft Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, With Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, With Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Bifurc |
| O471376 Approach Dilation of Left Femoral Artery with Four or More Drug- eluting Intraluminal Devices, Percutaneous Approach-eluting intraluminal Devices, Percutaneous Approach-eluting intraluminal Devices, Percutaneous Approach-Osated Balloon, Percutaneous Approach O4713D1 Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, with intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Two intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Two intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or Dilation of Left Femoral Artery, Bifurcation, with Four or Dilation of Left Femoral Artery, Bifurcation, with Four or Dilation of Left Femoral Artery, Bifurcation, with Four or Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, With Drug- eluting intraluminal Device, Legal Legal Legal Legal Dilation of Left Femoral Artery, Bifurcation, With Drug- eluting intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Bifurcat |
| Dilation of Left Femoral Artery with Four or More Drug- eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Femoral Artery with intraluminal Device, using Drug-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Left Percutaneous Endoscopic Approach-Left Left Percutaneous Endoscopic Approach-Left Left Percutane |
| eluting Intraluminal Devices, Percutaneous Approache-luting Intraluminal Devices, Percutaneous Approach Dilation of Left Femoral Artery with Intraluminal Device, using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach- Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, With Drug- eluting Intraluminal Device, Using Drug-Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Using Drug-Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Per |
| 0471372 Intraluminal Devices, Percutaneous Approach Dilation of Left Femoral Artery with Intraluminal Device, using Drug-Coaded Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach-Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Device, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach-Dilation of Left Femoral Artery usin Four or More Intraluminal Devices, Percutaneous Approach-Dilation of Left Femoral Artery, Bifurcation, Percutaneous Endoscopic Approach-Di |
| Dilation of Left Femoral Artery with Intraluminal Device, using Drug-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery using Drug Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approac |
| using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or O4713F2 Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or O4713G2 Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Dilation of Left Femoral Artery, Bifurcation, Percutaneous Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Using Drug-Coated Billoon, Percutaneous Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Bifurcation, wi |
| Balloon, Percutaneous Approach |
| Dilation of Left Femoral Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Endoscopic Approacheluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, with Drug-eluting |
| Intraluminal Device, Percutaneous Approach— |
| Dilation of Left Femoral Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous DA71321 Dilation of Left Femoral Artery, Bifurcation, Percutaneous DA71322 Dilation of Left Femoral Artery, Bifurcation, Percutaneous DA71323 Dilation of Left Femoral Artery, Bifurcation, Percutaneous DA71324 Dilation of Left Femoral Artery, Bifurcation, Percutaneous DA71325 Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Device, Percutaneous Endoscopic DA71446 Dilation of Left Femoral Artery with Drug-eluting Device, Percutaneous Endoscopic DA71446 Dilation of Left Femoral Artery with Drug-eluting |
| 04713DZ Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting |
| Dilation of Left Femoral Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, using Drug eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous |
| O47L3E6 Intraluminal Devices, Percutaneous Approach— |
| Dilation of Left Femoral Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, lusing Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery Bifurcation, with Drug-eluting Intraluminal Device, Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-Bitalian Device, Percutaneous Endoscopic Approach—Bitalian Device, Percutaneous App |
| Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery, Bifurcation, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Endoscopic Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery, Bifurcation, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery with Drug-eluting |
| Intraluminal Devices, Percutaneous Approach— |
| Dilation of Left Femoral Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| Devices, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug Puting Intraluminal Device, using Drug Puting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach— Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| 047L3G6 More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— O47L3Z6 Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— O47L3Z6 Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| Intraluminal Devices, Percutaneous Approach— Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— O47L3Z6 Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery using Drug-Coated Balloon, Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— O47L3Z6 Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| Percutaneous Approach-Coated Balloon, Percutaneous Approach Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— O47L3Z6 Approach— Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting Dilation of Left Femoral Artery with Drug-eluting |
| 047L3Z1 Approach 047L3Z6 Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— 047L3ZZ Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery, Bifurcation, Percutaneous Approach— O47L3ZZ Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| 047L3ZE Approach— 047L3ZZ Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery, Percutaneous Approach— Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery with Drug-eluting Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| Intraluminal Device, using Drug-eluting Intraluminal Device, using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| 047L441 using Drug Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous 047L446 Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous 047L446 Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| Approach-eluting Intraluminal Device, Percutaneous 047L446 Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| 047L446 Endoscopic Approach Dilation of Left Femoral Artery with Drug-eluting |
| Dilation of Left Femoral Artery with Drug-eluting |
| , |
| Intraluminal Device, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Device, Percutaneous Endoscopic |
| 047L44Z Approach |
| Dilation of Left Femoral Artery, Bifurcation, with Two Drug- |
| eluting Intraluminal Devices, Percutaneous Endoscopic |
| Approach-eluting Intraluminal Devices, Percutaneous |
| 047L456 Endoscopic Approach |
| Dilation of Left Femoral Artery with Two Drug-eluting |
| Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic 047L45Z Approach |
| Dilation of Left Femoral Artery, Bifurcation, with Three Drug- |
| eluting Intraluminal Devices, Percutaneous Endoscopic |
| Approach-eluting Intraluminal Devices, Percutaneous |
| 047L466 Endoscopic Approach |
| Dilation of Left Femoral Artery with Three Drug-eluting |
| Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic |
| 047L46Z Approach |


| Supplement Hemiazygos Vein with Autologous Tissue Substitute, Open Approach Supplement Hemiazygos Vein with Synthetic Substitute, | |
|---|---|
| Supplement Hemiazygos Vein with Synthetic Substitute, | |
| Open Approach | |
| Supplement Hemiazygos Vein with Nonautologous Tissue | |
| Substitute, Open Approach— | |
| Supplement Hemiazygos Vein with Autologous Tissue | |
| • | |
| 1. | |
| _ · · | |
| · | |
| 1 11 | |
| Substitute, Percutaneous Approach– | |
| Supplement Right Innominate Vein with Synthetic | |
| Substitute, Percutaneous Approach– | |
| Supplement Right Innominate Vein with Nonautologous | |
| Tissue Substitute, Percutaneous Approach— | |
| Supplement Right Innominate Vein with Autologous Tissue | |
| Substitute, Percutaneous Endoscopic Approach | |
| Supplement Right Innominate Vein with Synthetic | |
| Substitute, Percutaneous Endoscopic Approach | |
| Supplement Right Innominate Vein with Nonautologous | |
| Tissue Substitute, Percutaneous Endoscopic Approach— | |
| Supplement Left Innominate Vein with Autologous Tissue | |
| Substitute, Open Approach- | |
| Supplement Left Innominate Vein with Synthetic Substitute, | |
| Open Approach | |
| Supplement Left Innominate Vein with Nonautologous | |
| Tissue Substitute, Open Approach- | |
| Supplement Left Innominate Vein with Autologous Tissue | |
| Substitute, Percutaneous Approach– | |
| Supplement Left Innominate Vein with Synthetic Substitute, | |
| Percutaneous Approach | |
| Supplement Left Innominate Vein with Nonautologous | |
| Tissue Substitute, Percutaneous Approach | |
| Supplement Left Innominate Vein with Autologous Tissue | |
| Substitute, Percutaneous Endoscopic Approach | |
| Supplement Left Innominate Vein with Synthetic Substitute, | |
| Percutaneous Endoscopic Approach- | |
| Supplement Left Innominate Vein with Nonautologous | |
| Tissue Substitute, Percutaneous Endoscopic Approach— | |
| Supplement Right Subclavian Vein with Autologous Tissue | |
| Substitute, Open Approach- | |
| Supplement Right Subclavian Vein with Synthetic | |
| Substitute, Open Approach- | |
| | Substitute, Percutaneous Approach— Supplement Hemiazygos Vein with Synthetic Substitute, Percutaneous Approach— Supplement Hemiazygos Vein with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Hemiazygos Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Hemiazygos Vein with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Hemiazygos Vein with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Innominate Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Innominate Vein with Synthetic Substitute, Open Approach— Supplement Right Innominate Vein with Nonautologous Tissue Substitute, Open Approach— Supplement Right Innominate Vein with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Innominate Vein with Synthetic Substitute, Percutaneous Approach— Supplement Right Innominate Vein with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Right Innominate Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Innominate Vein with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Innominate Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Open Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Open Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Open Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Innominate Vein with Nonautologous Tissue Substitute, Percutane |


| _ |
|---|


| Dilation of Inferior Vana Court Department Annually | |
|---|---|
| · | |
| Approach- | |
| Dilation of Splenic Vein, Open Approach | |
| Dilation of Splenic Vein with Intraluminal Device, | |
| Percutaneous Approach | |
| Dilation of Splenic Vein, Percutaneous Approach- | |
| Dilation of Splenic Vein with Intraluminal Device, | |
| Percutaneous Endoscopic Approach | |
| Dilation of Splenic Vein, Percutaneous Endoscopic Approach— | |
| Dilation of Gastric Vein with Intraluminal Device, Open | |
| Approach | |
| Dilation of Gastric Vein, Open Approach | |
| Dilation of Gastric Vein with Intraluminal Device, | |
| Percutaneous Approach | |
| Dilation of Gastric Vein, Percutaneous Approach— | |
| Dilation of Gastric Vein with Intraluminal Device, | |
| Percutaneous Endoscopic Approach- | |
| Dilation of Contrie Vain Department of Endoardin Assessed | |
| 1 11 | |
| Approach- | |
| Dilation of Hepatic Vein with Intraluminal Device, Open | |
| Approach- | |
| Dilation of Hepatic Vein, Open Approach— | |
| Dilation of Hepatic Vein with Intraluminal Device, | |
| Percutaneous Approach | |
| Dilation of Hepatic Vein, Percutaneous Approach | |
| Dilation of Hepatic Vein with Intraluminal Device, | |
| Percutaneous Endoscopic Approach | |
| · · | |
| 7 1 11 | |
| · | |
| * * | |
| · | |
| • • | |
| Device, Percutaneous Endoscopic Approach— | |
| Dilation of Superior Mesenteric Vein, Percutaneous | |
| | 1 |
| | Dilation of Splenic Vein, Open Approach— Dilation of Splenic Vein with Intraluminal Device, Percutaneous Approach— Dilation of Splenic Vein, Percutaneous Approach— Dilation of Splenic Vein, Percutaneous Approach— Dilation of Splenic Vein, Percutaneous Endoscopic Approach— Dilation of Gastric Vein with Intraluminal Device, Open Approach— Dilation of Gastric Vein with Intraluminal Device, Open Approach— Dilation of Gastric Vein with Intraluminal Device, Percutaneous Approach— Dilation of Gastric Vein, Open Approach— Dilation of Gastric Vein, Percutaneous Approach— Dilation of Gastric Vein, Percutaneous Approach— Dilation of Gastric Vein, Percutaneous Endoscopic Approach— Dilation of Esophageal Vein with Intraluminal Device, Open Approach— Dilation of Esophageal Vein, Open Approach— Dilation of Esophageal Vein with Intraluminal Device, Percutaneous Approach— Dilation of Esophageal Vein, Percutaneous Approach— Dilation of Esophageal Vein, Percutaneous Approach— Dilation of Esophageal Vein, Percutaneous Endoscopic Approach— Dilation of Esophageal Vein, Percutaneous Endoscopic Approach— Dilation of Hepatic Vein with Intraluminal Device, Open Approach— Dilation of Hepatic Vein with Intraluminal Device, Open Approach— Dilation of Hepatic Vein with Intraluminal Device, Open Approach— Dilation of Hepatic Vein with Intraluminal Device, Percutaneous Approach— Dilation of Hepatic Vein with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Hepatic Vein with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Superior Mesenteric Vein with Intraluminal Device, Open Approach— Dilation of Superior Mesenteric Vein with Intraluminal Device, Percutaneous Approach— Dilation of Superior Mesenteric Vein with Intraluminal Device, Percutaneous Approach— Dilation of Superior Mesenteric Vein with Intraluminal Device, Percutaneous Approach— Dilation of Superior Mesenteric Vein with Intraluminal Device, Percutaneous Approach— Dilation of Superior Mesenteric Vein with Intraluminal Device, Percutaneous Endoscop |


| Insertion of Intraluminal Device into Left Femoral Vein, | |
|---|---|
| Percutaneous Approach- | |
| Insertion of Intraluminal Device into Left Femoral Vein, | |
| Percutaneous Endoscopic Approach— | |
| Insertion of Intraluminal Device into Right Greater | |
| Saphenous Vein, Open Approach– | |
| Insertion of Intraluminal Device into Right Greater | |
| Saphenous Vein, Percutaneous Approach– | |
| Insertion of Intraluminal Device into Right Greater | |
| Saphenous Vein, Percutaneous Endoscopic Approach | |
| Insertion of Intraluminal Device into Left Greater Saphenous | |
| Vein, Open Approach- | |
| Insertion of Intraluminal Device into Left Greater Saphenous | |
| · · | |
| Vein, Open Approach- | |
| · · · | |
| · • | |
| 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
| · | |
| · | |
| · · · | |
| Percutaneous Approach | |
| Insertion of Intraluminal Device into Left Foot Vein, | |
| Percutaneous Endoscopic Approach— | |
| Insertion of Monitoring Device into Lower Vein, Open | |
| Approach- | |
| Insertion of Intraluminal Device into Lower Vein, Open | |
| Approach- | |
| Insertion of Intraluminal Device into Lower Vein, | |
| Percutaneous Approach | |
| Insertion of Monitoring Device into Lower Vein, | |
| Percutaneous Endoscopic Approach— | |
| Insertion of Intraluminal Device into Lower Vein, | |
| Percutaneous Endoscopic Approach— | |
| Release Inferior Vena Cava, Open Approach— | |
| Release Inferior Vena Cava, Percutaneous Approach- | |
| Release Inferior Vena Cava, Percutaneous Endoscopic | |
| Approach– | |
| Approach— Release Splenic Vein, Open Approach— | |
| | Open Approach— Insertion of Intraluminal Device into Left Femoral Vein, Percutaneous Approach— Insertion of Intraluminal Device into Left Femoral Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Right Greater Saphenous Vein, Open Approach— Insertion of Intraluminal Device into Right Greater Saphenous Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Right Greater Saphenous Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Left Greater Saphenous Vein, Open Approach— Insertion of Intraluminal Device into Left Greater Saphenous Vein, Open Approach— Insertion of Intraluminal Device into Left Greater Saphenous Vein, Percutaneous Approach— Insertion of Intraluminal Device into Right Lesser Saphenous Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Right Lesser Saphenous Vein, Open Approach— Insertion of Intraluminal Device into Right Lesser Saphenous Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Left Lesser Saphenous Vein, Percutaneous Approach— Insertion of Intraluminal Device into Left Lesser Saphenous Vein, Open Approach— Insertion of Intraluminal Device into Left Lesser Saphenous Vein, Percutaneous Approach— Insertion of Intraluminal Device into Left Lesser Saphenous Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Right Foot Vein, Open Approach— Insertion of Intraluminal Device into Right Foot Vein, Open Approach— Insertion of Intraluminal Device into Right Foot Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Left Foot Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Left Foot Vein, Percutaneous Approach— Insertion of Intraluminal Device into Lower Vein, Open Approach— Insertion of Intraluminal Device into Lower Vein, Open Approach— Insertion of Intraluminal Device into Lower Vein, Percutaneous Endoscopic Approach— Insertion of Intraluminal Device into Lower Vein, Percutaneous Endos |


| Reposition Right Lesser Saphenous Vein, Percutaneous Approach— | |
|---|---|
| | 1 |
| · | |
| i i | |
| Reposition Right Foot Vein, Open Approach— | |
| Reposition Right Foot Vein, Percutaneous Approach- | |
| Reposition Right Foot Vein, Percutaneous Endoscopic | |
| Approach- | |
| Reposition Left Foot Vein, Open Approach— | |
| Reposition Left Foot Vein, Percutaneous Approach- | |
| Reposition Left Foot Vein, Percutaneous Endoscopic | |
| Approach- | |
| Reposition Lower Vein, Open Approach— | |
| neposition tower vein, rescutarieous Approach- | |
| Renosition Lower Vein Percutaneous Endoscopic Approach | |
| | <u> </u> |
| 1 1 | |
| Percutaneous Approach | |
| Supplement Inferior Vena Cava with Nonautologous Tissue | |
| Substitute, Percutaneous Approach | |
| Supplement Inferior Vena Cava with Autologous Tissue | |
| Substitute, Percutaneous Endoscopic Approach— | |
| Supplement Inferior Vena Cava with Synthetic Substitute, | |
| Percutaneous Endoscopic Approach— | |
| Supplement Inferior Vena Cava with Nonautologous Tissue | |
| Substitute, Percutaneous Endoscopic Approach | |
| 1 1 | |
| Supplement Splenic Vein with Nonautologous Tissue | |
| | Reposition Right Foot Vein, Percutaneous Endoscopic Approach— Reposition Left Foot Vein, Open Approach— Reposition Left Foot Vein, Percutaneous Approach— Reposition Left Foot Vein, Percutaneous Endoscopic Approach— Reposition Lower Vein, Open Approach— Reposition Lower Vein, Percutaneous Approach— Reposition Lower Vein, Percutaneous Endoscopic Approach— Reposition Lower Vein, Percutaneous Endoscopic Approach— Supplement Inferior Vena Cava with Autologous Tissue Substitute, Open Approach— Supplement Inferior Vena Cava with Synthetic Substitute, Open Approach— Supplement Inferior Vena Cava with Nonautologous Tissue Substitute, Open Approach— Supplement Inferior Vena Cava with Synthetic Substitute, Percutaneous Approach— Supplement Inferior Vena Cava with Synthetic Substitute, Percutaneous Approach— Supplement Inferior Vena Cava with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Inferior Vena Cava with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Inferior Vena Cava with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Inferior Vena Cava with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Inferior Vena Cava with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Inferior Vena Cava with Nonautologous Tissue |


| | Revision of Extraluminal Device in Lower Vein, Percutaneous | |
|---|---|---|
| 06WY4CZ | Endoscopic Approach— | |
| | Revision of Intraluminal Device in Lower Vein, Percutaneous | |
| 06WY4DZ | Endoscopic Approach- | |
| HCPCS | | |
| 35256 | | |
| 35286 | | |
| 35351 | | |
| 35355 | | |
| 35361 | | |
| 35363 | | |
| 35371 | | |
| 35372 | | |
| 35381 | | |
| 35454 | | |
| 35456 | | |
| 35459<br>35470 | | |
| 35473 | | |
| 35474 | | |
| 35482 | | |
| 35483 | | |
| 35485 | | |
| 35492 | | |
| 35493 | | |
| 35495 | | |
| 35521 | | |
| 35533 | | |
| 35556 | | l. |
| 35558 | | |
| 35563 | | |
| 35565 | | |
| 35566 | | |
| 35571 | | |
| 35621 | | |
| 35623 | | |
| 35641 | | |
| 35646 | | |
| 35647 | | |
| 35650 | | |
| 35651 | | |
| 35654 | | |
| 35656 | | |
| 35661 | | |
| 35663 | | |
| 35666 | | |
| 35671 | | |
| Hypertension | | |
| Hypertension | ICD9 Dy LongDosICD10 | LongDesiCD0 |

| 110 | 4010 | Fescartial (nyimaya) bunaytansian | Malignant assential hypertension |
|---|---|---|---|
| I10<br>I10 | 4010<br>4011 | Essential (primary) hypertension | Malignant essential hypertension |
| 110 | 4011 | Essential (primary) hypertension Essential (primary) hypertension | Benign essential hypertension Unspecified essential hypertension |
| 1160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| 1161 | 4019 | Hypertensive digency Hypertensive emergency | Unspecified essential hypertension |
| 1169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| l119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| I110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| 1119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| 1110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart failure |
| 1110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| l129 | 40300 | Hypertensive chronic kidney disease with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive chronic kidney disease, malignant, with chroni kidney disease stage I through stage IV, or unspecified |
| 1120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, malignant, with chroni |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| 1129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney disease | kidney disease stage I through stage IV, or unspecified |
| I120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| 1129 | 40390 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, unspecified, with |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney | chronic kidney disease stage I through stage IV, or |
| | | disease | unspecified |
| l120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, unspecified, with |
| | | kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal disease |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | through stage IV, or unspecified |
| I130 | 40401 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| 1130 | 40401 | | 1 |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| 11211 | 40403 | or unspecified chronic kidney disease | through stage IV, or unspecified |
| I1311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| 1132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and with stage 5 chronic kidney disease, or end stage | with heart failure and with chronic kidney disease stage V o |
| | | renal disease | end stage renal disease |
| 11310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | through stage IV, or unspecified |
| 1130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I through |
| | | or unspecified chronic kidney disease | stage IV, or unspecified |
| 11311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| 1132 | 40415 | failure and with stage 5 chronic kidney disease, or end stage | heart failure and chronic kidney disease stage V or end stag |
| | | renal disease | renal disease |
| 11210 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| 11310 | 40430 | | |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | THE PROPERTY OF THE PROPERTY OF CULTURE KINDON GLCGGCG | through stage IV, or unspecified |
| 14.33 | 40.40: | disease, or unspecified chronic kidney disease | |
| I130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| 1130 | 40491 | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and with chronic kidney disease stage I |
| | | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| I130<br>I1311 | 40491 | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified Hypertensive heart and chronic kidney disease, unspecified, |
| | | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive heart and chronic kidney disease, unspecified, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |

| l132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
|---|---|---|---|
| | | failure and with stage 5 chronic kidney disease, or end stage | with heart failure and chronic kidney disease stage V or end |
| | | renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| I150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| I158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| I150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| I151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| I152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| I158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| I159 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |

Diabetes


Hyperlipidemia

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| E780 | 2720 | Pure hypercholesterolemia | PURE HYPERCHOLESTEROLEMIA |
| E7800 | 2722 | | MIXED HYPERLIPIDEMIA |
| E781 | 2724 | Pure hyperglyceridemia | OTHER AND UNSPECIFIED HYPERLIPIDEMIA |
| E782 | | Mixed hyperlipidemia | |
| E784 | | Other hyperlipidemia | |
| E785 | | Hyperlipidemia, unspecified | |

Renal dysfunction


| M10372 | 40410 | Gout due to renal impairment, left ankle and foot | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE<br>BENIGN WITHOUT HEART FAILURE WITH CHRONIC KIDNEY |
|---|---|---|---|
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| M10379 | 40411 | Gout due to renal impairment, unspecified ankle and foot | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE BENIGN WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| M1038 | 40412 | Gout due to renal impairment, vertebrae | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| 1411030 | 40412 | Godt dde to rendr impairment, vertebrae | BENIGN WITHOUT HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| N44020 | 40412 | Cout due to revel imperiment moultiple sites | |
| M1039 | 40413 | Gout due to renal impairment, multiple sites | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | BENIGN WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| M3214 | 4049 | Glomerular disease in systemic lupus erythematosus | UNSPECIFIED HYPERTENSIVE HEART AND KIDNEY DISEASE |
| M3215 | 40490 | Tubulo-interstitial nephropathy in systemic lupus | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | erythematosus | UNSPECIFIED WITHOUT HEART FAILURE WITH CHRONIC |
| | | | KIDNEY DISEASE STAGE I THROUGH STAGE IV OR |
| | | | UNSPECIFIED |
| M3504 | 40491 | Sicca syndrome with tubulo-interstitial nephropathy | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | | UNSPECIFIED WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE I THROUGH STAGE IV OR UNSPECIFIED |
| N000 | 40492 | Acute nephritic syndrome with minor glomerular | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| 11000 | 40432 | | |
| | | abnormality | UNSPECIFIED WITHOUT HEART FAILURE WITH CHRONIC |
| | | | KIDNEY DISEASE STAGE V OR END STAGE RENAL DISEASE |
| N001 | 40493 | Acute nephritic syndrome with focal and segmental | HYPERTENSIVE HEART AND CHRONIC KIDNEY DISEASE |
| | | glomerular lesions | UNSPECIFIED WITH HEART FAILURE WITH CHRONIC KIDNEY |
| | | | DISEASE STAGE V OR END STAGE RENAL DISEASE |
| N002 | 4533 | Acute nephritic syndrome with diffuse membranous glomerulonephritis | EMBOLISM AND THROMBOSIS OF RENAL VEIN |
| N003 | 5800 | Acute nephritic syndrome with diffuse mesangial | ACUTE GLOMERULONEPHRITIS WITH LESION OF |
| | | proliferative glomerulonephritis | PROLIFERATIVE GLOMERULONEPHRITIS |
| N004 | 5804 | Acute nephritic syndrome with diffuse endocapillary | ACUTE GLOMERULONEPHRITIS WITH LESION OF RAPIDLY |
| | | proliferative glomerulonephritis | PROGRESSIVE GLOMERULONEPHRITIS |
| N005 | 5808 | Acute nephritic syndrome with diffuse mesangiocapillary | ACUTE GLOMERULONEPHRITIS WITH OTHER SPECIFIED |
| | 5000 | glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N006 | 5809 | Acute nephritic syndrome with dense deposit disease | ACUTE GLOMERULONEPHRITIS WITH UNSPECIFIED |
| 11000 | 3003 | Acute hepimitie syndrome with dense deposit disease | PATHOLOGICAL LESION IN KIDNEY |
| N007 | 581 | Acute nephritic syndrome with diffuse crescentic | NEPHROTIC SYNDROME |
| | | glomerulonephritis | |
| N008 | 5810 | Acute nephritic syndrome with other morphologic changes | NEPHROTIC SYNDROME WITH LESION OF PROLIFERATIVE |
| | | | GLOMERULONEPHRITIS |
| N009 | 5811 | Acute nephritic syndrome with unspecified morphologic | NEPHROTIC SYNDROME WITH LESION OF MEMBRANOUS |
| .1005 | 5522 | changes | GLOMERULONEPHRITIS |
| N010 | 5812 | Rapidly progressive nephritic syndrome with minor | NEPHROTIC SYNDROME WITH LESION OF |
| NOIO | 3012 | glomerular abnormality | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| NO11 | Γ012 | | |
| N011 | 5813 | Rapidly progressive nephritic syndrome with focal and | NEPHROTIC SYNDROME WITH LESION OF MINIMAL CHANG |
| NOTO | F045 | segmental glomerular lesions | GLOMERULONEPHRITIS |
| N012 | 5818 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH OTHER SPECIFIED |
| | | membranous glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N013 | 58181 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME IN DISEASES CLASSIFIED |
| | | mesangial proliferative glomerulonephritis | ELSEWHERE |
| N014 | 58189 | Rapidly progressive nephritic syndrome with diffuse | OTHER NEPHROTIC SYNDROME WITH SPECIFIED |
| | | endocapillary proliferative glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N015 | 5819 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH UNSPECIFIED PATHOLOGICA |
| | | mesangiocapillary glomerulonephritis | LESION IN KIDNEY |
| N016 | 5820 | Rapidly progressive nephritic syndrome with dense deposit | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | 3020 | disease | PROLIFERATIVE GLOMERULONEPHRITIS |
| NO17 | F024 | | |
| N017 | 5821 | Rapidly progressive nephritic syndrome with diffuse | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | crescentic glomerulonephritis | MEMBRANOUS GLOMERULONEPHRITIS |
| N018 | 5822 | Rapidly progressive nephritic syndrome with other | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | morphologic changes | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N019 | 5824 | Rapidly progressive nephritic syndrome with unspecified | CHRONIC GLOMERULONEPHRITIS WITH LESION OF RAPIDL |
| INOIS | | | |

| N020 | 5828 | Recurrent and persistent hematuria with minor glomerular | CHRONIC GLOMERULONEPHRITIS WITH OTHER SPECIFIED |
|---|---|---|---|
| NUZU | 3828 | abnormality | PATHOLOGICAL LESION IN KIDNEY |
| N021 | 5829 | Recurrent and persistent hematuria with focal and | CHRONIC GLOMERULONEPHRITIS WITH UNSPECIFIED |
| 11021 | 3023 | segmental glomerular lesions | PATHOLOGICAL LESION IN KIDNEY |
| N022 | 5830 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | membranous glomerulonephritis | OR CHRONIC WITH LESION OF PROLIFERATIVE |
| | | | GLOMERULONEPHRITIS |
| N023 | 5831 | Recurrent and persistent hematuria with diffuse mesangial | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | proliferative glomerulonephritis | OR CHRONIC WITH LESION OF MEMBRANOUS |
| | | | GLOMERULONEPHRITIS |
| N024 | 5832 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | endocapillary proliferative glomerulonephritis | OR CHRONIC WITH LESION OF MEMBRANOPROLIFERATIVE |
| | | | GLOMERULONEPHRITIS |
| N025 | 5834 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | mesangiocapillary glomerulonephritis | OR CHRONIC WITH LESION OF RAPIDLY PROGRESSIVE |
| | | | GLOMERULONEPHRITIS |
| N026 | 5836 | Recurrent and persistent hematuria with dense deposit | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | disease | OR CHRONIC WITH LESION OF RENAL CORTICAL NECROSIS |
| N027 | 5837 | Recurrent and persistent hematuria with diffuse crescentic | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| | | glomerulonephritis | OR CHRONIC WITH LESION OF RENAL MEDULLARY NECROSIS |
| NOSE | F020 | Recurrent and persistent hematuria with other morphologic | NEDUDITIC AND MEDUDODATUV NOT CRECIFIED AS A SUTE |
| N028 | 5838 | changes | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH OTHER SPECIFIED PATHOLOGICAL LESION |
| | | Changes | IN KIDNEY |
| N029 | 5839 | Recurrent and persistent hematuria with unspecified | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE |
| 14023 | 3633 | morphologic changes | OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN |
| | | Thorphologic changes | KIDNEY |
| N030 | 5846 | Chronic nephritic syndrome with minor glomerular | ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL |
| | 30.0 | abnormality | NECROSIS |
| N031 | 5847 | Chronic nephritic syndrome with focal and segmental | ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLAR |
| | | glomerular lesions | (PAPILLARY) NECROSIS |
| N032 | 5848 | Chronic nephritic syndrome with diffuse membranous | ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED |
| | | glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N033 | 5849 | Chronic nephritic syndrome with diffuse mesangial | ACUTE KIDNEY FAILURE UNSPECIFIED |
| | | proliferative glomerulonephritis | |
| N034 | 5851 | Chronic nephritic syndrome with diffuse endocapillary | CHRONIC KIDNEY DISEASE STAGE I |
| | | proliferative glomerulonephritis | |
| N035 | 5852 | Chronic nephritic syndrome with diffuse mesangiocapillary | CHRONIC KIDNEY DISEASE STAGE II (MILD) |
| | | glomerulonephritis | |
| N036 | 5853 | Chronic nephritic syndrome with dense deposit disease | CHRONIC KIDNEY DISEASE STAGE III (MODERATE) |
| N037 | 5854 | Chronic nephritic syndrome with diffuse crescentic | CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) |
| NOSO | 5055 | glomerulonephritis | CURONIC VIRNEY DISEASE STACE V |
| N038 | 5855 | Chronic nephritic syndrome with other morphologic changes | CHRONIC KIDNEY DISEASE STAGE V |
| N039 | 5856 | Chronic nephritic syndrome with unspecified morphologic | END STAGE RENAL DISEASE |
| 14033 | 3030 | changes | END STAGE RENALDISEASE |
| N040 | 5859 | Nephrotic syndrome with minor glomerular abnormality | CHRONIC KIDNEY DISEASE UNSPECIFIED |
| N041 | 86600 | Nephrotic syndrome with focal and segmental glomerular | UNSPECIFIED INJURY TO KIDNEY WITHOUT OPEN WOUND |
| | | lesions | INTO CAVITY |
| N042 | 86601 | Nephrotic syndrome with diffuse membranous | HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE |
| | | glomerulonephritis | WITHOUT OPEN WOUND INTO CAVITY |
| N043 | 8661 | Nephrotic syndrome with diffuse mesangial proliferative | INJURY TO KIDNEY WITH OPEN WOUND INTO CAVITY |
| | | glomerulonephritis | |
| N044 | | Nephrotic syndrome with diffuse endocapillary proliferative | |
| | | glomerulonephritis | |
| N045 | | Nephrotic syndrome with diffuse mesangiocapillary | |
| | | glomerulonephritis | |
| N046 | | Nephrotic syndrome with dense deposit disease | |
| N047 | | Nephrotic syndrome with diffuse crescentic | |
| NO40 | | glomerulonephritis | |
| N048 | | Nephrotic syndrome with other morphologic changes | |
| N049 | <u> </u> | Nephrotic syndrome with unspecified morphologic changes | |

| | | T |
|---|---|---|
| N050 | Unspecified nephritic syndrome with minor glomerular | |
| NOE1 | abnormality | |
| N051 | Unspecified nephritic syndrome with focal and segmental glomerular lesions | |
| N052 | Unspecified nephritic syndrome with diffuse membranous | |
| | glomerulonephritis | |
| N053 | Unspecified nephritic syndrome with diffuse mesangial | |
| | proliferative glomerulonephritis | |
| N054 | Unspecified nephritic syndrome with diffuse endocapillary | |
| 11054 | proliferative glomerulonephritis | |
| N055 | Unspecified nephritic syndrome with diffuse | |
| 14055 | mesangiocapillary glomerulonephritis | |
| N056 | Unspecified nephritic syndrome with dense deposit disease | |
| N057 | Unspecified nephritic syndrome with diffuse crescentic | |
| INU57 | | |
| NOTO | glomerulonephritis | |
| N058 | Unspecified nephritic syndrome with other morphologic | |
| | changes | |
| N059 | Unspecified nephritic syndrome with unspecified | |
| | morphologic changes | |
| N060 | Isolated proteinuria with minor glomerular abnormality | |
| N061 | Isolated proteinuria with focal and segmental glomerular | |
| | lesions | |
| N062 | Isolated proteinuria with diffuse membranous | |
| | glomerulonephritis | |
| N063 | Isolated proteinuria with diffuse mesangial proliferative | |
| | glomerulonephritis | |
| N064 | Isolated proteinuria with diffuse endocapillary proliferative | |
| | glomerulonephritis | |
| N065 | Isolated proteinuria with diffuse mesangiocapillary | |
| | glomerulonephritis | |
| N066 | Isolated proteinuria with dense deposit disease | |
| N067 | Isolated proteinuria with diffuse crescentic | |
| | glomerulonephritis | |
| N068 | Isolated proteinuria with other morphologic lesion | |
| N069 | Isolated proteinuria with unspecified morphologic lesion | |
| N070 | Hereditary nephropathy, not elsewhere classified with | |
| | minor glomerular abnormality | |
| N071 | Hereditary nephropathy, not elsewhere classified with focal | |
| | and segmental glomerular lesions | |
| N072 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse membranous glomerulonephritis | |
| N073 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse mesangial proliferative glomerulonephritis | |
| N074 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse endocapillary proliferative glomerulonephritis | |
| N075 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse mesangiocapillary glomerulonephritis | |
| N076 | Hereditary nephropathy, not elsewhere classified with | |
| 1,0,0 | dense deposit disease | |
| N077 | Hereditary nephropathy, not elsewhere classified with | |
| , | diffuse crescentic glomerulonephritis | |
| N078 | Hereditary nephropathy, not elsewhere classified with | |
| 1,070 | other morphologic lesions | |
| N079 | Hereditary nephropathy, not elsewhere classified with | |
| 14075 | unspecified morphologic lesions | |
| N08 | Glomerular disorders in diseases classified elsewhere | |
| N140 | Analgesic nephropathy Nephropathy indused by other drugs medicaments and | |
| N141 | Nephropathy induced by other drugs, medicaments and | |
| N14.63 | biological substances | |
| N142 | Nephropathy induced by unspecified drug, medicament or | |
| N14.63 | biological substance | |
| N143 | Nephropathy induced by heavy metals | |


## Appendix A Comorbid conditions

| 964 |
|-----|
| 965 |
| 966 |
| 967 |
| 968 |
| 969 |
| 970 |
| 989 |
| 993 |
| 512 |
| 559 |


## Appendix A Comorbid conditions

| K7581 | Nonalcoholic steatohepatitis (NASH) |
|-------|---------------------------------------------------|
| K7589 | Other specified inflammatory liver diseases |
| K759 | Inflammatory liver disease, unspecified |
| K760 | Fatty (change of) liver, not elsewhere classified |
| K761 | Chronic passive congestion of liver |
| K763 | Infarction of liver |
| K764 | Peliosis hepatis |
| K765 | Hepatic veno-occlusive disease |
| K766 | Portal hypertension |
| K767 | Hepatorenal syndrome |
| K7681 | Hepatopulmonary syndrome |
| K7689 | Other specified diseases of liver |
| K769 | Liver disease, unspecified |
| K77 | Liver disorders in diseases classified elsewhere |

## **Asthma**


Ischemic heart disease


## Appendix A Comorbid conditions


COPD

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| J40 | 490 | Bronchitis, not specified as acute or chronic | BRONCHITIS NOT SPECIFIED AS ACUTE OR CHRONIC |
| J410 | 491 | Simple chronic bronchitis | CHRONIC BRONCHITIS |
| J411 | 4910 | Mucopurulent chronic bronchitis | SIMPLE CHRONIC BRONCHITIS |
| J418 | 4911 | Mixed simple and mucopurulent chronic bronchitis | MUCOPURULENT CHRONIC BRONCHITIS |
| J42 | 4912 | Unspecified chronic bronchitis | OBSTRUCTIVE CHRONIC BRONCHITIS |
| J430 | 49120 | Unilateral pulmonary emphysema [MacLeod's syndrome] | OBSTRUCTIVE CHRONIC BRONCHITIS WITHOUT |
| | | | EXACERBATION |
| J431 | 49121 | Panlobular emphysema | OBSTRUCTIVE CHRONIC BRONCHITIS WITH (ACUTE) |
| | | | EXACERBATION |
| J432 | 49122 | Centrilobular emphysema | OBSTRUCTIVE CHRONIC BRONCHITIS WITH ACUTE |
| | | | BRONCHITIS |
| J438 | 4918 | Other emphysema | OTHER CHRONIC BRONCHITIS |
| J439 | 4919 | Emphysema, unspecified | UNSPECIFIED CHRONIC BRONCHITIS |
| J440 | 492 | Chronic obstructive pulmonary disease with acute lower | EMPHYSEMA |
| | | respiratory infection | |
| J441 | 4920 | Chronic obstructive pulmonary disease with (acute) | EMPHYSEMATOUS BLEB |
| | | exacerbation | |
| J449 | 4928 | Chronic obstructive pulmonary disease, unspecified | OTHER EMPHYSEMA |
| J470 | 494 | Bronchiectasis with acute lower respiratory infection | BRONCHIECTASIS |
| J471 | 4940 | Bronchiectasis with (acute) exacerbation | BRONCHIECTASIS WITHOUT ACUTE EXACERBATION |
| J479 | 4941 | Bronchiectasis, uncomplicated | BRONCHIECTASIS WITH ACUTE EXACERBATION |
| | 496 | | CHRONIC AIRWAY OBSTRUCTION NOT ELSEWHERE |
| | | | CLASSIFIED |

Occurence of malignancy

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| C000 | 140 | Malignant neoplasm of external upper lip | MALIGNANT NEOPLASM OF LIP |
| C001 | 1400 | Malignant neoplasm of external lower lip | MALIGNANT NEOPLASM OF UPPER LIP VERMILION BORDER |
| C002 | 1401 | Malignant neoplasm of external lip, unspecified | MALIGNANT NEOPLASM OF LOWER LIP VERMILION BORDER |
| C003 | 1403 | Malignant neoplasm of upper lip, inner aspect | MALIGNANT NEOPLASM OF UPPER LIP INNER ASPECT |
| C004 | 1404 | Malignant neoplasm of lower lip, inner aspect | MALIGNANT NEOPLASM OF LOWER LIP INNER ASPECT |
| C005 | 1405 | Malignant neoplasm of lip, unspecified, inner aspect | MALIGNANT NEOPLASM OF LIP UNSPECIFIED INNER ASPECT |
| C006 | 1406 | Malignant neoplasm of commissure of lip, unspecified | MALIGNANT NEOPLASM OF COMMISSURE OF LIP |
| C008 | 1408 | Malignant neoplasm of overlapping sites of lip | MALIGNANT NEOPLASM OF OTHER SITES OF LIP |
| C009 | 1409 | Malignant neoplasm of lip, unspecified | MALIGNANT NEOPLASM OF LIP UNSPECIFIED VERMILION |
| | | | BORDER |
| C01 | 141 | Malignant neoplasm of base of tongue | MALIGNANT NEOPLASM OF TONGUE |
| C020 | 1410 | Malignant neoplasm of dorsal surface of tongue | MALIGNANT NEOPLASM OF BASE OF TONGUE |
| C021 | 1411 | Malignant neoplasm of border of tongue | MALIGNANT NEOPLASM OF DORSAL SURFACE OF TONGUE |
| C022 | 1412 | Malignant neoplasm of ventral surface of tongue | MALIGNANT NEOPLASM OF TIP AND LATERAL BORDER OF |
| | | | TONGUE |

| C023 | 1413 | Malignant neoplasm of anterior two-thirds of tongue, part unspecified | MALIGNANT NEOPLASM OF VENTRAL SURFACE OF TONGUE |
|---|---|---|---|
| C024 | 1414 | Malignant neoplasm of lingual tonsil | MALIGNANT NEOPLASM OF ANTERIOR TWO-THIRDS OF TONGUE PART UNSPECIFIED |
| C028 | 1415 | Malignant neoplasm of overlapping sites of tongue | MALIGNANT NEOPLASM OF JUNCTIONAL ZONE OF TONGUE |
| C029 | 1416 | Malignant neoplasm of tongue, unspecified | MALIGNANT NEOPLASM OF LINGUAL TONSIL |
| C030 | 1418 | Malignant neoplasm of upper gum | MALIGNANT NEOPLASM OF OTHER SITES OF TONGUE |
| C031 | 1419 | Malignant neoplasm of lower gum | MALIGNANT NEOPLASM OF TONGUE UNSPECIFIED |
| C039 | 142 | Malignant neoplasm of gum, unspecified | MALIGNANT NEOPLASM OF MAJOR SALIVARY GLANDS |
| C040 | 1420 | Malignant neoplasm of anterior floor of mouth | MALIGNANT NEOPLASM OF PAROTID GLAND |
| C041 | 1421 | Malignant neoplasm of lateral floor of mouth | MALIGNANT NEOPLASM OF SUBMANDIBULAR GLAND |
| C048 | 1422 | Malignant neoplasm of overlapping sites of floor of mouth | MALIGNANT NEOPLASM OF SUBLINGUAL GLAND |
| C049 | 1428 | Malignant neoplasm of floor of mouth, unspecified | MALIGNANT NEOPLASM OF OTHER MAJOR SALIVARY GLANDS |
| C050 | 1429 | Malignant neoplasm of hard palate | MALIGNANT NEOPLASM OF SALIVARY GLAND UNSPECIFIED |
| C051 | 143 | Malignant neoplasm of soft palate | MALIGNANT NEOPLASM OF GUM |
| C052 | 1430 | Malignant neoplasm of uvula | MALIGNANT NEOPLASM OF UPPER GUM |
| C058 | 1431 | Malignant neoplasm of overlapping sites of palate | MALIGNANT NEOPLASM OF LOWER GUM |
| C059 | 1438 | Malignant neoplasm of palate, unspecified | MALIGNANT NEOPLASM OF OTHER SITES OF GUM |
| C060 | 1439 | Malignant neoplasm of cheek mucosa | MALIGNANT NEOPLASM OF GUM UNSPECIFIED |
| C061 | 144 | Malignant neoplasm of vestibule of mouth | MALIGNANT NEOPLASM OF FLOOR OF MOUTH |
| C062 | 1440 | Malignant neoplasm of retromolar area | MALIGNANT NEOPLASM OF ANTERIOR PORTION OF FLOOR OF MOUTH |
| C0680 | 1441 | Malignant neoplasm of overlapping sites of unspecified parts of mouth | MALIGNANT NEOPLASM OF LATERAL PORTION OF FLOOR OF MOUTH |
| C0689 | 1448 | Malignant neoplasm of overlapping sites of other parts of mouth | MALIGNANT NEOPLASM OF OTHER SITES OF FLOOR OF MOUTH |
| C069 | 1449 | Malignant neoplasm of mouth, unspecified | MALIGNANT NEOPLASM OF FLOOR OF MOUTH PART UNSPECIFIED |
| C07 | 145 | Malignant neoplasm of parotid gland | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED PARTS OF MOUTH |
| C080 | 1450 | Malignant neoplasm of submandibular gland | MALIGNANT NEOPLASM OF CHEEK MUCOSA |
| C081 | 1451 | Malignant neoplasm of sublingual gland | MALIGNANT NEOPLASM OF VESTIBULE OF MOUTH |
| C089 | 1452 | Malignant neoplasm of major salivary gland, unspecified | MALIGNANT NEOPLASM OF HARD PALATE |
| C090 | 1453 | Malignant neoplasm of tonsillar fossa | MALIGNANT NEOPLASM OF SOFT PALATE |
| C091 | 1454 | Malignant neoplasm of tonsillar pillar (anterior) (posterior) | MALIGNANT NEOPLASM OF UVULA |
| C098 | 1455 | Malignant neoplasm of overlapping sites of tonsil | MALIGNANT NEOPLASM OF PALATE UNSPECIFIED |
| C099 | 1456 | Malignant neoplasm of tonsil, unspecified | MALIGNANT NEOPLASM OF RETROMOLAR AREA |
| C100 | 1458 | Malignant neoplasm of vallecula | MALIGNANT NEOPLASM OF OTHER SPECIFIED PARTS OF MOUTH |
| C101 | 1459 | Malignant neoplasm of anterior surface of epiglottis | MALIGNANT NEOPLASM OF MOUTH UNSPECIFIED |
| C102 | 146 | Malignant neoplasm of lateral wall of oropharynx | MALIGNANT NEOPLASM OF OROPHARYNX |
| C103 | 1460 | Malignant neoplasm of posterior wall of oropharynx | MALIGNANT NEOPLASM OF TONSIL |
| C104 | 1461 | Malignant neoplasm of branchial cleft | MALIGNANT NEOPLASM OF TONSILLAR FOSSA |
| C108 | 1462 | Malignant neoplasm of overlapping sites of oropharynx | MALIGNANT NEOPLASM OF TONSILLAR PILLARS (ANTERIOR) (POSTERIOR) |
| C109 | 1463 | Malignant neoplasm of oropharynx, unspecified | MALIGNANT NEOPLASM OF VALLECULA EPIGLOTTICA |
| C110 | 1464 | Malignant neoplasm of superior wall of nasopharynx | MALIGNANT NEOPLASM OF ANTERIOR ASPECT OF EPIGLOTTIS |
| C111 | 1465 | Malignant neoplasm of posterior wall of nasopharynx | MALIGNANT NEOPLASM OF JUNCTIONAL REGION OF OROPHARYNX |
| C112 | 1466 | Malignant neoplasm of lateral wall of nasopharynx | MALIGNANT NEOPLASM OF LATERAL WALL OF<br>OROPHARYNX |
| C113 | 1467 | Malignant neoplasm of anterior wall of nasopharynx | MALIGNANT NEOPLASM OF POSTERIOR WALL OF OROPHARYNX |
| C118 | 1468 | Malignant neoplasm of overlapping sites of nasopharynx | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF OROPHARYNX |
| C119 | 1469 | Malignant neoplasm of nasopharynx, unspecified | MALIGNANT NEOPLASM OF OROPHARYNX UNSPECIFIED SITE |
| C12 | 147 | Malignant neoplasm of pyriform sinus | MALIGNANT NEOPLASM OF NASOPHARYNX |

| C130 | 1470 | Malignant neoplasm of postcricoid region | MALIGNANT NEOPLASM OF SUPERIOR WALL OF |
|---|---|---|---|
| | | | NASOPHARYNX |
| C131 | 1471 | Malignant neoplasm of aryepiglottic fold, hypopharyngeal aspect | MALIGNANT NEOPLASM OF POSTERIOR WALL OF NASOPHARYNX |
| C132 | 1472 | Malignant neoplasm of posterior wall of hypopharynx | MALIGNANT NEOPLASM OF LATERAL WALL OF NASOPHARYNX |
| C138 | 1473 | Malignant neoplasm of overlapping sites of hypopharynx | MALIGNANT NEOPLASM OF ANTERIOR WALL OF |
| C136 | 14/3 | ivialignant neoplasm of overlapping sites of hypophalynx | NASOPHARYNX |
| C139 | 1478 | Malignant neoplasm of hypopharynx, unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| C139 | 1476 | | NASOPHARYNX |
| C140 | 1479 | Malignant neoplasm of pharynx, unspecified | MALIGNANT NEOPLASM OF NASOPHARYNX UNSPECIFIED SITE |
| C142 | 148 | Malignant neoplasm of Waldeyer's ring | MALIGNANT NEOPLASM OF HYPOPHARYNX |
| C148 | 1480 | Malignant neoplasm of overlapping sites of lip, oral cavity | MALIGNANT NEOPLASM OF POSTCRICOID REGION OF |
| | | and pharynx | HYPOPHARYNX |
| C153 | 1481 | Malignant neoplasm of upper third of esophagus | MALIGNANT NEOPLASM OF PYRIFORM SINUS |
| C154 | 1482 | Malignant neoplasm of middle third of esophagus | MALIGNANT NEOPLASM OF ARYEPIGLOTTIC FOLD |
| | | | HYPOPHARYNGEAL ASPECT |
| C155 | 1483 | Malignant neoplasm of lower third of esophagus | MALIGNANT NEOPLASM OF POSTERIOR HYPOPHARYNGEAL |
| | | | WALL |
| C158 | 1488 | Malignant neoplasm of overlapping sites of esophagus | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | | HYPOPHARYNX |
| C159 | 1489 | Malignant neoplasm of esophagus, unspecified | MALIGNANT NEOPLASM OF HYPOPHARYNX UNSPECIFIED |
| | | | SITE |
| C160 | 149 | Malignant neoplasm of cardia | MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITES |
| | | | WITHIN THE LIP ORAL CAVITY AND PHARYNX |
| C161 | 1490 | Malignant neoplasm of fundus of stomach | MALIGNANT NEOPLASM OF PHARYNX UNSPECIFIED |
| C162 | 1491 | Malignant neoplasm of body of stomach | MALIGNANT NEOPLASM OF WALDEYER'S RING |
| C163 | 1498 | Malignant neoplasm of pyloric antrum | MALIGNANT NEOPLASM OF OTHER SITES WITHIN THE LIP |
| | | | AND ORAL CAVITY |
| C164 | 1499 | Malignant neoplasm of pylorus | MALIGNANT NEOPLASM OF ILL-DEFINED SITES WITHIN THE |
| | | , | LIP AND ORAL CAVITY |
| C165 | 150 | Malignant neoplasm of lesser curvature of stomach, unspecified | MALIGNANT NEOPLASM OF ESOPHAGUS |
| C166 | 1500 | Malignant neoplasm of greater curvature of stomach, unspecified | MALIGNANT NEOPLASM OF CERVICAL ESOPHAGUS |
| C168 | 1501 | Malignant neoplasm of overlapping sites of stomach | MALIGNANT NEOPLASM OF THORACIC ESOPHAGUS |
| C169 | 1502 | Malignant neoplasm of stomach, unspecified | MALIGNANT NEOPLASM OF ABDOMINAL ESOPHAGUS |
| C170 | 1503 | Malignant neoplasm of duodenum | MALIGNANT NEOPLASM OF UPPER THIRD OF ESOPHAGUS |
| C171 | 1504 | Malignant neoplasm of jejunum | MALIGNANT NEOPLASM OF MIDDLE THIRD OF ESOPHAGUS |
| C172 | 1505 | Malianant nagalaga afilana | MANUCNANT NEODIACA OF LOWER THIRD OF ECODIACHE |
| C172<br>C173 | 1505<br>1508 | Malignant neoplasm of ileum | MALIGNANT NEOPLASM OF LOWER THIRD OF ESOPHAGUS MALIGNANT NEOPLASM OF OTHER SPECIFIED PART OF |
| C1/3 | 1508 | Meckel's diverticulum, malignant | ESOPHAGUS |
| C178 | 1509 | Malignant neoplasm of overlapping sites of small intestine | MALIGNANT NEOPLASM OF ESOPHAGUS UNSPECIFIED SITE |
| C179 | 151 | Malignant neoplasm of small intestine, unspecified | MALIGNANT NEOPLASM OF STOMACH |
| C180 | 1510 | Malignant neoplasm of small intestine, unspecified Malignant neoplasm of cecum | MALIGNANT NEOPLASM OF STOMACH MALIGNANT NEOPLASM OF CARDIA |
| C180 | 1510 | Malignant neoplasm of cecum Malignant neoplasm of appendix | MALIGNANT NEOPLASM OF PYLORUS |
| C182 | 1511 | Malignant neoplasm of ascending colon | MALIGNANT NEOPLASM OF PYLORUS MALIGNANT NEOPLASM OF PYLORIC ANTRUM |
| C183 | 1512 | Malignant neoplasm of ascending colon Malignant neoplasm of hepatic flexure | MALIGNANT NEOPLASM OF FYLORIC ANTROM MALIGNANT NEOPLASM OF FUNDUS OF STOMACH |
| C184 | 1513 | Malignant neoplasm of nepatic flexure Malignant neoplasm of transverse colon | MALIGNANT NEOPLASM OF FUNDOS OF STOMACH MALIGNANT NEOPLASM OF BODY OF STOMACH |
| C184 | 1514 | Malignant neoplasm of transverse colon Malignant neoplasm of splenic flexure | MALIGNANT NEOPLASM OF BODY OF STOMACH MALIGNANT NEOPLASM OF LESSER CURVATURE OF |
| C103 | 1313 | manghant neopiasin of spieriic flexule | STOMACH UNSPECIFIED |
| C186 | 1516 | Malignant neoplasm of descending colon | MALIGNANT NEOPLASM OF GREATER CURVATURE OF |
| | | | STOMACH UNSPECIFIED |
| C187 | 1518 | Malignant neoplasm of sigmoid colon | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF STOMACH |
| C188 | 1519 | Malignant neoplasm of overlapping sites of colon | MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED SITE |
| C188 | 1519 | Malignant neoplasm of colon, unspecified | MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED SITE MALIGNANT NEOPLASM OF SMALL INTESTINE INCLUDING |
| C103 | 132 | iviangnant neopiasin of colon, unspecified | DUODENUM |
| C19 | 1520 | Malignant neoplasm of rectosigmoid junction | MALIGNANT NEOPLASM OF DUODENUM |
| C19 | 1520 | I wangnant neopiasin of rectosignord junction | INIMININI INEOLIAZINI OL DOODENOINI |

| C20 | 1521 | Malignant neoplasm of rectum | MALIGNANT NEOPLASM OF JEJUNUM |
|---|---|---|---|
| C210 | 1522 | Malignant neoplasm of anus, unspecified | MALIGNANT NEOPLASM OF ILEUM |
| C211 | 1523 | Malignant neoplasm of anal canal | MALIGNANT NEOPLASM OF MECKEL'S DIVERTICULUM |
| C212 | 1528 | Malignant neoplasm of cloacogenic zone | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| CLIL | 1320 | Manghane neophasm of diodeogethic zone | SMALL INTESTINE |
| C218 | 1529 | Malignant neoplasm of overlapping sites of rectum, anus | MALIGNANT NEOPLASM OF SMALL INTESTINE UNSPECIFIED |
| CLIC | 1323 | and anal canal | ISITE |
| C220 | 153 | Liver cell carcinoma | MALIGNANT NEOPLASM OF COLON |
| C221 | 1530 | Intrahepatic bile duct carcinoma | MALIGNANT NEOPLASM OF HEPATIC FLEXURE |
| C222 | 1531 | Hepatoblastoma | MALIGNANT NEOPLASM OF TRANSVERSE COLON |
| C223 | 1532 | Angiosarcoma of liver | MALIGNANT NEOPLASM OF DESCENDING COLON |
| C224 | 1533 | Other sarcomas of liver | MALIGNANT NEOPLASM OF SIGMOID COLON |
| C227 | 1534 | Other specified carcinomas of liver | MALIGNANT NEOPLASM OF CECUM |
| C228 | 1535 | Malignant neoplasm of liver, primary, unspecified as to type | |
| CZZO | 1555 | wanghant heopiasin of liver, primary, anspealied as to type | WALIGNAM NEOFENSIN OF ATTEMPTA VERIMIN ORIVINS |
| C229 | 1536 | Malignant neoplasm of liver, not specified as primary or | MALIGNANT NEOPLASM OF ASCENDING COLON |
| CZZJ | 1550 | secondary | WALIGNANT NEOF EASIN OF ASCENDING COLON |
| C23 | 1537 | Malignant neoplasm of gallbladder | MALIGNANT NEOPLASM OF SPLENIC FLEXURE |
| C240 | 1538 | Malignant neoplasm of extrahepatic bile duct | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| C240 | 1556 | Walighant neoplasm of extranepatic bile duct | LARGE INTESTINE |
| C241 | 1539 | Malignant neoplasm of ampulla of Vater | MALIGNANT NEOPLASM OF COLON UNSPECIFIED SITE |
| C241<br>C248 | 1539 | Malignant neoplasm of overlapping sites of biliary tract | MALIGNANT NEOPLASM OF RECTUM RECTOSIGMOID |
| C246 | 154 | Manghant neoplasm of overlapping sites of billary tract | JUNCTION AND ANUS |
| C249 | 1540 | Malignant pooplasm of hillians tract, unspecified | MALIGNANT NEOPLASM OF RECTOSIGMOID JUNCTION |
| C249<br>C250 | 1540 | Malignant neoplasm of biliary tract, unspecified Malignant neoplasm of head of pancreas | MALIGNANT NEOPLASM OF RECTUM |
| | | Malignant neoplasm of body of pancreas | |
| C251 | 1542 | , , | MALIGNANT NEOPLASM OF ANAL CANAL |
| C252 | 1543 | Malignant neoplasm of tail of pancreas | MALIGNANT NEOPLASM OF ANUS UNSPECIFIED SITE |
| C253 | 1548 | Malignant neoplasm of pancreatic duct | MALIGNANT NEOPLASM OF OTHER SITES OF RECTUM |
| 625.4 | 455 | AA-P | RECTOSIGMOID JUNCTION AND ANUS |
| C254 | 155 | Malignant neoplasm of endocrine pancreas | MALIGNANT NEOPLASM OF LIVER AND INTRAHEPATIC BILE |
| 6257 | 4550 | Ad-Providence for the control of control | DUCTS |
| C257 | 1550 | Malignant neoplasm of other parts of pancreas | MALIGNANT NEOPLASM OF LIVER PRIMARY |
| C258 | 1551 | Malignant neoplasm of overlapping sites of pancreas | MALIGNANT NEOPLASM OF INTRAHEPATIC BILE DUCTS |
| C259 | 1552 | Malignant neoplasm of pancreas, unspecified | MALIGNANT NEOPLASM OF LIVER NOT SPECIFIED AS |
| 6260 | 456 | Malta and an effect of the start and an effect of | PRIMARY OR SECONDARY |
| C260 | 156 | Malignant neoplasm of intestinal tract, part unspecified | MALIGNANT NEOPLASM OF GALLBLADDER AND |
| 6264 | 4560 | AA-P | EXTRAHEPATIC BILE DUCTS |
| C261 | 1560 | Malignant neoplasm of spleen | MALIGNANT NEOPLASM OF GALLBLADDER |
| C269 | 1561 | Malignant neoplasm of ill-defined sites within the digestive | MALIGNANT NEOPLASM OF EXTRAHEPATIC BILE DUCTS |
| 6200 | 4562 | system | MANUCHANT NEODIACAA OF ANADIHLA OF WATER |
| C300 | 1562 | Malignant neoplasm of nasal cavity | MALIGNANT NEOPLASM OF AMPULLA OF VATER |
| C301 | 1568 | Malignant neoplasm of middle ear | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| 0040 | 4560 | AA II | GALLBLADDER AND EXTRAHEPATIC BILE DUCTS |
| C310 | 1569 | Malignant neoplasm of maxillary sinus | MALIGNANT NEOPLASM OF BILIARY TRACT PART |
| | | | UNSPECIFIED SITE |
| C311 | 157 | Malignant neoplasm of ethmoidal sinus | MALIGNANT NEOPLASM OF PANCREAS |
| C312 | 1570 | Malignant neoplasm of frontal sinus | MALIGNANT NEOPLASM OF HEAD OF PANCREAS |
| C313 | 1571 | Malignant neoplasm of sphenoid sinus | MALIGNANT NEOPLASM OF BODY OF PANCREAS |
| C318 | 1572 | Malignant neoplasm of overlapping sites of accessory | MALIGNANT NEOPLASM OF TAIL OF PANCREAS |
| | | sinuses | |
| C319 | 1573 | Malignant neoplasm of accessory sinus, unspecified | MALIGNANT NEOPLASM OF PANCREATIC DUCT |
| C320 | 1574 | Malignant neoplasm of glottis | MALIGNANT NEOPLASM OF ISLETS OF LANGERHANS |
| C321 | 1578 | Malignant neoplasm of supraglottis | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |
| | | | PANCREAS |
| C322 | 1579 | Malignant neoplasm of subglottis | MALIGNANT NEOPLASM OF PANCREAS PART UNSPECIFIED |
| C323 | 158 | Malignant neoplasm of laryngeal cartilage | MALIGNANT NEOPLASM OF RETROPERITONEUM AND |
| | | | PERITONEUM |
| C328 | 1580 | Malignant neoplasm of overlapping sites of larynx | MALIGNANT NEOPLASM OF RETROPERITONEUM |
| C329 | 1588 | Malignant neoplasm of larynx, unspecified | MALIGNANT NEOPLASM OF SPECIFIED PARTS OF |
| | | | PERITONEUM |
| C33 | 1589 | Malignant neoplasm of trachea | MALIGNANT NEOPLASM OF PERITONEUM UNSPECIFIED |


| | 1722 | Malignant melanoma of overlapping sites of skin | MALIGNANT MELANOMA OF SKIN OF EAR AND EXTERNAL AUDITORY CANAL |
|---|---|---|---|
| C439 | 1723 | Malignant melanoma of skin, unspecified | MALIGNANT MELANOMA OF SKIN OF OTHER AND UNSPECIFIED PARTS OF FACE |
| C450 | 1724 | Mesothelioma of pleura | MALIGNANT MELANOMA OF SKIN OF SCALP AND NECK |
| C451 | 1725 | Mesothelioma of peritoneum | MALIGNANT MELANOMA OF SKIN OF TRUNK EXCEPT |
| C452 | 1726 | Mesothelioma of pericardium | SCROTUM MALIGNANT MELANOMA OF SKIN OF UPPER LIMB |
| | | | INCLUDING SHOULDER |
| C457 | 1727 | Mesothelioma of other sites | MALIGNANT MELANOMA OF SKIN OF LOWER LIMB INCLUDING HIP |
| C459 | 1728 | Mesothelioma, unspecified | MALIGNANT MELANOMA OF OTHER SPECIFIED SITES OF |
| | | | SKIN |
| C460 | 1729 | Kaposi's sarcoma of skin | MELANOMA OF SKIN SITE UNSPECIFIED |
| C461 | 174 | Kaposi's sarcoma of soft tissue | MALIGNANT NEOPLASM OF FEMALE BREAST |
| C462 | 1740 | Kaposi's sarcoma of palate | MALIGNANT NEOPLASM OF NIPPLE AND AREOLA OF FEMALE BREAST |
| C463 | 1741 | Kaposi's sarcoma of lymph nodes | MALIGNANT NEOPLASM OF CENTRAL PORTION OF FEMALI<br>BREAST |
| C464 | 1742 | Kaposi's sarcoma of gastrointestinal sites | MALIGNANT NEOPLASM OF UPPER-INNER QUADRANT OF |
| | | | FEMALE BREAST |
| C4650 | 1743 | Kaposi's sarcoma of unspecified lung | MALIGNANT NEOPLASM OF LOWER-INNER QUADRANT OF FEMALE BREAST |
| C4651 | 1744 | Kaposi's sarcoma of right lung | MALIGNANT NEOPLASM OF UPPER-OUTER QUADRANT OF |
| C4652 | 1745 | Kaposi's sarcoma of left lung | FEMALE BREAST MALIGNANT NEOPLASM OF LOWER-OUTER QUADRANT OF |
| C4032 | 1745 | Raposi's sarcoma of left fung | FEMALE BREAST |
| C467 | 1746 | Kaposi's sarcoma of other sites | MALIGNANT NEOPLASM OF AXILLARY TAIL OF FEMALE |
| | | | BREAST |
| C469 | 1748 | Kaposi's sarcoma, unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF FEMALE BREAST |
| C470 | 1749 | Malignant neoplasm of peripheral nerves of head, face and neck | MALIGNANT NEOPLASM OF BREAST (FEMALE) UNSPECIFIE SITE |
| C4710 | 175 | Malignant neoplasm of peripheral nerves of unspecified upper limb, including shoulder | MALIGNANT NEOPLASM OF MALE BREAST |
| C4711 | 1750 | Malignant neoplasm of peripheral nerves of right upper limb, including shoulder | MALIGNANT NEOPLASM OF NIPPLE AND AREOLA OF MALE |
| C4712 | 1759 | Malignant neoplasm of peripheral nerves of left upper limb, | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED SITE |
| | | including shoulder | OF MALE BREAST |
| C4720 | 176 | Malignant neoplasm of peripheral nerves of unspecified lower limb, including hip | KAPOSI'S SARCOMA |
| C4721 | 1760 | Malignant neoplasm of peripheral nerves of right lower limb, including hip | KAPOSI'S SARCOMA SKIN |
| C4722 | 1761 | Malignant neoplasm of peripheral nerves of left lower limb, | KAPOSI'S SARCOMA SOFT TISSUE |
| C472 | 1763 | including hip Makingant populasm of peripheral perves of theray | VADOSI'S SADCOMA DALATE |
| C473<br>C474 | 1762<br>1763 | Malignant neoplasm of peripheral nerves of thorax Malignant neoplasm of peripheral nerves of abdomen | KAPOSI'S SARCOMA PALATE |
| | | | KAPOSI'S SARCOMA GASTROINTESTINAL SITES |
| C475<br>C476 | 1764<br>1765 | Malignant neoplasm of peripheral nerves of pelvis Malignant neoplasm of peripheral nerves of trunk, | KAPOSI'S SARCOMA LYMPH NODES |
| C478 | 1768 | unspecified Malignant neoplasm of overlapping sites of peripheral | KAPOSI'S SARCOMA OTHER SPECIFIED SITES |
| C470 | 1700 | nerves and autonomic nervous system | NAT OST S SAILCOMA OTHER STEED SITES |
| C479 | 1769 | Malignant neoplasm of peripheral nerves and autonomic nervous system, unspecified | KAPOSI'S SARCOMA UNSPECIFIED SITE |
| C480 | 179 | Malignant neoplasm of retroperitoneum | MALIGNANT NEOPLASM OF UTERUS-PART UNS |
| C481 | 180 | Malignant neoplasm of specified parts of peritoneum | MALIGNANT NEOPLASM OF CERVIX UTERI |
| C481 | 1800 | Malignant neoplasm of peritoneum, unspecified | MALIGNANT NEOPLASM OF ENDOCERVIX |
| C482 | 1801 | Malignant neoplasm of overlapping sites of retroperitoneum | |
| | | and peritoneum | |
| C490 | 1808 | Malignant neoplasm of connective and soft tissue of head, | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF |


| C50929 | 1909 | Malignant neoplasm of unspecified site of unspecified male breast | MALIGNANT NEOPLASM OF EYE PART UNSPECIFIED |
|---|---|---|---|
| C510 | 191 | Malignant neoplasm of labium majus | MALIGNANT NEOPLASM OF BRAIN |
| C511 | 1910 | Malignant neoplasm of labium minus | MALIGNANT NEOPLASM OF CEREBRUM EXCEPT LOBES AN VENTRICLES |
| C512 | 1911 | Malignant neoplasm of clitoris | MALIGNANT NEOPLASM OF FRONTAL LOBE |
| C518 | 1912 | Malignant neoplasm of overlapping sites of vulva | MALIGNANT NEOPLASM OF TEMPORAL LOBE |
| C519 | 1913 | Malignant neoplasm of vulva, unspecified | MALIGNANT NEOPLASM OF PARIETAL LOBE |
| C52 | 1914 | Malignant neoplasm of vagina | MALIGNANT NEOPLASM OF OCCIPITAL LOBE |
| C530 | 1915 | Malignant neoplasm of endocervix | MALIGNANT NEOPLASM OF VENTRICLES |
| C531 | 1916 | Malignant neoplasm of exocervix | MALIGNANT NEOPLASM OF CEREBELLUM NOT OTHERWIS |
| 0001 | 1510 | mang. and neephasm of electricity | SPECIFIED |
| C538 | 1917 | Malignant neoplasm of overlapping sites of cervix uteri | MALIGNANT NEOPLASM OF BRAIN STEM |
| C539 | 1918 | Malignant neoplasm of cervix uteri, unspecified | MALIGNANT NEOPLASM OF OTHER PARTS OF BRAIN |
| C540 | 1919 | Malignant neoplasm of isthmus uteri | MALIGNANT NEOPLASM OF BRAIN UNSPECIFIED SITE |
| C541 | 192 | Malignant neoplasm of endometrium | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED PARTS OF NERVOUS SYSTEM |
| C542 | 1920 | Malignant neoplasm of myometrium | MALIGNANT NEOPLASM OF CRANIAL NERVES |
| | | Malignant neoplasm of fundus uteri | MALIGNANT NEOPLASM OF CRANIAL NERVES MALIGNANT NEOPLASM OF CEREBRAL MENINGES |
| C543 | 1921 | · | |
| C548 | 1922 | Malignant neoplasm of overlapping sites of corpus uteri | MALIGNANT NEOPLASM OF SPINAL CORD |
| C549 | 1923 | Malignant neoplasm of corpus uteri, unspecified | MALIGNANT NEOPLASM OF SPINAL MENINGES |
| C55 | 1928 | Malignant neoplasm of uterus, part unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES OF NERVOUS SYSTEM |
| CEC1 | 1020 | Malignant needlasm of right overv | MALIGNANT NEOPLASM OF NERVOUS SYSTEM PART |
| C561 | 1929 | Malignant neoplasm of right ovary | UNSPECIFIED |
| CEGO | 102 | Malignant needless of left every | |
| C562 | 193 | Malignant neoplasm of left ovary | MALIGNANT NEOPLASM OF THYROID GLAND |
| C569 | 194 | Malignant neoplasm of unspecified ovary | MALIGNANT NEOPLASM OF OTHER ENDOCRINE GLANDS |
| 05700 | 1010 | | AND RELATED STRUCTURES |
| C5700 | 1940 | Malignant neoplasm of unspecified fallopian tube | MALIGNANT NEOPLASM OF ADRENAL GLAND |
| C5701 | 1941 | Malignant neoplasm of right fallopian tube | MALIGNANT NEOPLASM OF PARATHYROID GLAND |
| C5702 | 1943 | Malignant neoplasm of left fallopian tube | MALIGNANT NEOPLASM OF PITUITARY GLAND AND |
| | | | CRANIOPHARYNGEAL DUCT |
| C5710 | 1944 | Malignant neoplasm of unspecified broad ligament | MALIGNANT NEOPLASM OF PINEAL GLAND |
| C5711 | 1945 | Malignant neoplasm of right broad ligament | MALIGNANT NEOPLASM OF CAROTID BODY |
| C5712 | 1946 | Malignant neoplasm of left broad ligament | MALIGNANT NEOPLASM OF AORTIC BODY AND OTHER PARAGANGLIA |
| C5720 | 1948 | Malignant neoplasm of unspecified round ligament | MALIGNANT NEOPLASM OF OTHER ENDOCRINE GLANDS |
| 03720 | 25 .0 | manghant heopiasin of anopeanies rouns ngament | AND RELATED STRUCTURES |
| C5721 | 1949 | Malignant neoplasm of right round ligament | MALIGNANT NEOPLASM OF ENDOCRINE GLAND SITE |
| C3721 | 1343 | Wanghane neoplasm of right Found ngament | UNSPECIFIED |
| C5722 | 195 | Malignant neoplasm of left round ligament | MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED SITE |
| C573 | 1950 | Malignant neoplasm of parametrium | MALIGNANT NEOPLASM OF HEAD FACE AND NECK |
| C574 | 1951 | Malignant neoplasm of uterine adnexa, unspecified | MALIGNANT NEOPLASM OF THORAX |
| C577 | 1952 | Malignant neoplasm of other specified female genital organs | S MALIGNANT NEOPLASM OF ABDOMEN |
| C578 | 1953 | Malignant neoplasm of overlapping sites of female genital | MALIGNANT NEOPLASM OF PELVIS |
| C579 | 1954 | organs Malignant neoplasm of female genital organ, unspecified | MALIGNANT NEOPLASM OF UPPER LIMB |
| C579 | 1954 | Malignant neoplasm of lemale genital organ, unspecified Malignant neoplasm of placenta | MALIGNANT NEOPLASM OF LOWER LIMB |
| C600 | | Malignant neoplasm of prepuce | |
| | 1958 | Malignant neoplasm of prepuce Malignant neoplasm of glans penis | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES |
| C601 | 196 | Mangnant neoplasm of glans penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM LYMPH NODES |
| C602 | 1960 | Malignant neoplasm of body of penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| 0000 | | | LYMPH NODES OF HEAD FACE AND NECK |
| C608 | 1961 | Malignant neoplasm of overlapping sites of penis | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM INTRATHORACIC LYMPH NODES |
| C609 | 1962 | Malignant neoplasm of penis, unspecified | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| 2233 | 1332 | | INTRA-ABDOMINAL LYMPH NODES |
| C61 | 1963 | Malignant neoplasm of prostate | SECONDARY AND UNSPECIFIED MALIGNANT NEOPLASM |
| COI | 1,000 | manghant neoplasm of prostate | SESSIONIL AND ONSI EGI IED MALIGINAMI MEOFEASIM |


| | | _ |
|---|---|---|
| D409 | Neoplasm of uncertain behavior of male genital organ, | |
| | unspecified | |
| D4100 | Neoplasm of uncertain behavior of unspecified kidney | |
| D4101 | Neoplasm of uncertain behavior of right kidney | |
| D4102 | Neoplasm of uncertain behavior of left kidney | |
| D4110 | Neoplasm of uncertain behavior of unspecified renal pelvis | |
| D4111 | Neoplasm of uncertain behavior of right renal pelvis | |
| D4112 | Neoplasm of uncertain behavior of left renal pelvis | |
| D4120 | Neoplasm of uncertain behavior of unspecified ureter | |
| D4121 | Neoplasm of uncertain behavior of right ureter | |
| D4122 | Neoplasm of uncertain behavior of left ureter | |
| D413 | Neoplasm of uncertain behavior of urethra | |
| D414 | Neoplasm of uncertain behavior of bladder | |
| D418 | Neoplasm of uncertain behavior of other specified urinary organs | |
| D419 | Neoplasm of uncertain behavior of unspecified urinary organ | |
| D420 | Neoplasm of uncertain behavior of cerebral meninges | |
| D421 | Neoplasm of uncertain behavior of spinal meninges | |
| D429 | Neoplasm of uncertain behavior of spinal meninges Neoplasm of uncertain behavior of meninges, unspecified | |
| D430 | Neoplasm of uncertain behavior of brain, supratentorial | |
| D430 | Neoplasm of uncertain behavior of brain, suprateritorial | |
| D431 | Neoplasm of uncertain behavior of brain, unspecified | |
| D433 | Neoplasm of uncertain behavior of cranial nerves | |
| D434 | Neoplasm of uncertain behavior of spinal cord | |
| D438 | Neoplasm of uncertain behavior of other specified parts of | |
| D430 | | |
| D439 | central nervous system Neoplasm of uncertain behavior of central nervous system, | |
| D439 | unspecified | |
| D440 | Neoplasm of uncertain behavior of thyroid gland | |
| D4410 | Neoplasm of uncertain behavior of unspecified adrenal gland | |
| 04410 | Neopiasiii oi uncertaini benavior oi unspecineu aurenar gianu | |
| D4411 | Neoplasm of uncertain behavior of right adrenal gland | |
| D4411 | Neoplasm of uncertain behavior of left adrenal gland | |
| D4412 | Neoplasm of uncertain behavior of parathyroid gland | |
| D443 | Neoplasm of uncertain behavior of paratry rold grand | |
| D444 | Neoplasm of uncertain behavior of craniopharyngeal duct | |
| D445 | . , , | |
| | Neoplasm of uncertain behavior of pineal gland | |
| D446<br>D447 | Neoplasm of uncertain behavior of carotid body | |
| 0447 | Neoplasm of uncertain behavior of aortic body and other | |
| D440 | paraganglia | |
| D449 | Neoplasm of uncertain behavior of unspecified endocrine | |
| DAE | gland Polygythomia yara | <del> </del> |
| D45 | Polycythemia vera | <del> </del> |
| D460 | Refractory anemia without ring sideroblasts, so stated | |
| D461 | Refractory anemia with ring sideroblasts | |
| D4620 | Refractory anemia with excess of blasts, unspecified | |
| D4621 | Refractory anemia with excess of blasts 1 | |
| D4622 | Refractory anemia with excess of blasts 2 | |
| D464 | Refractory anemia, unspecified | |
| D469 | Myelodysplastic syndrome, unspecified | |
| D46A | Refractory cytopenia with multilineage dysplasia | <del> </del> |
| D46B | Refractory cytopenia with multilineage dysplasia and ring | |
| DAGG | sideroblasts | <del> </del> |
| D46C | Myelodysplastic syndrome with isolated del(5q) | |
| 5.105 | chromosomal abnormality | |
| D46Z | Other myelodysplastic syndromes | |
| D470 | Histiocytic and mast cell tumors of uncertain behavior | |
| D471 | Chronic myeloproliferative disease | |
| D473 | Essential (hemorrhagic) thrombocythemia | |
| D479 | Neoplasm of uncertain behavior of lymphoid, hematopoietic | |
| | and related tissue, unspecified | |


Drug abuse or dependence (includes alcohol)


Venous throm boem bolism


## Appendix A Comorbid conditions
